ClinicalTrials.gov Official Title: A Study of Rucaparib Versus Physician's Choice of Therapy in Patients With Metastatic Castration-resistant Prostate Cancer and Homologous Recombination Gene Deficiency (TRITON3)

ClinicalTrials.gov Identifier Number: NCT02975934

**Document Date:** 18 February 2022

**Document:** Clinical Study Protocol CO-338-063

**Study Title:** TRITON3: A Multicenter, Randomized, Open-label Phase 3 Study of Rucaparib versus Physician's Choice of Therapy for Patients with Metastatic Castration-resistant Prostate Cancer Associated with Homologous Recombination Deficiency

# Clinical Study Protocol: CO-338-063

Study Title: TRITON3: A Multicenter, Randomized, Open-label Phase 3 Study of

Rucaparib versus Physician's Choice of Therapy for Patients with Metastatic Castration-resistant Prostate Cancer Associated with

Homologous Recombination Deficiency

Study Number: CO-338-063

**Study Phase:** Phase 3

**Product Name:** Rucaparib (CO-338)

IND Number:

EUDRA CT

Number

Indication: Metastatic Castration-resistant Prostate Cancer

**Investigators:** Multicenter

Sponsor Name: Clovis Oncology, Inc.

**Sponsor Address:** 

Responsible Medical Officer:

| Protocol Version | <u>Date</u> |
|------------------|------------------|
| Amendment 4: | 18 February 2022 |

## Confidentiality Statement

This document contains confidential information belonging to Clovis Oncology, Inc. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Clovis Oncology, Inc., must be promptly notified

# COORDINATING INVESTIGATORS FOR THE STUDY



# PROTOCOL APPROVAL SIGNATURE PAGE

Protocol: CO-338-063

Title: TRITON3: A Multicenter, Randomized, Open-label Phase 3 Study of

Rucaparib versus Physician's Choice of Therapy for Patients with Metastatic Castration-resistant Prostate Cancer Associated with

Homologous Recombination Deficiency

Date: 18 February 2022

Version: Amendment 4



# PROTOCOL ACCEPTANCE FORM

| Protocol: | CO-338-063 | |
|---|---|---|
| Title: | TRITON3: A Multicenter, Randomized, Open-label Phase<br>Rucaparib versus Physician's Choice of Therapy for Patie<br>Castration-resistant Prostate Cancer Associated with Hom<br>Recombination Deficiency | ents with Metastatic |
| Date: | 18 February 2022 | |
| Version: | Amendment 4 | |
| required to conduc | ad this protocol and agree that it contains all of the necessa<br>t this study. I agree to conduct this study as described and<br>sinki, ICH Guidelines for GCP, and all applicable regulato | according to the |
| Investigator's Sign | aature | Date (dd month yyyy) |
| Name (printed) | | |

# 1 SYNOPSIS

# Sponsor

Clovis Oncology, Inc.

## **Name of Finished Product**

Rucaparib tablets

## Name of Active Ingredient

Rucaparib camsylate (CO-338)

# **Study Title**

TRITON3: A Multicenter, Randomized, Open-label Phase 3 Study of Rucaparib versus Physician's Choice of Therapy for Patients with Metastatic Castration-resistant Prostate Cancer Associated with Homologous Recombination Deficiency

## **Study Number**

CO-338-063

# **Study Phase**

Phase 3

#### Rationale

Deoxyribonucleic acid (DNA) is constantly damaged by both endogenous and exogenous (environmental) assaults. Normal cells repair single-strand breaks (SSBs) in DNA through a process known as base excision repair (BER). While there are several variations of BER, all pathways rely on the activity of poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) enzymes. SSBs that are not repaired result in stalled replication forks and the development of double-strand breaks (DSBs), which are in turn repaired by homologous recombination (HR) DNA repair, a complex process involving multiple proteins, including those encoded by breast cancer susceptibility gene 1 and 2 (BRCA1 and BRCA2), as well as ataxia telangiectasia mutated serine/threonine kinase (ATM), RAD51, Fanconi anemia core complex, and ataxia telangiectasia and RAD3-related (ATR) protein, among others. Homologous recombination defects or PARP inhibition on their own can be overcome by a cell, but the combination is fatal, a concept termed "synthetic lethality", and which forms the basis of the therapeutic approach of using PARP inhibition to kill cancer cells with a HR-deficient background. 1-3

Prostate cancer is the most common malignancy among men in the United States, and the second-most common cause of cancer-related mortality, with approximately 30,000 men dying of the disease each year. Based upon GLOBOCAN 2012 estimates, prostate cancer is the second leading malignancy diagnosis and fifth leading cause of death from cancer in men in worldwide, with 307,000 deaths estimated in 2012. The course of prostate cancer from diagnosis to death is often a series of clinical states progressing from localized disease to metastatic castration-resistant prostate cancer (mCRPC), a disease state characterized by resistance to standard androgen deprivation therapies (ADT) and that accounts for the majority of prostate cancer deaths.

Homologous recombination deficiency (HRD) has been observed in many carcinomas, including prostate cancer. Men with a germline mutation in BRCA2 are at increased risk for developing prostate cancer, estimated at 2.5 to 8.6-fold compared with non-carriers. Men with prostate cancer and a germline mutation in BRCA2 typically develop disease at a younger age, have more aggressive features and higher mortality rates. While less common in prostate cancer, germline mutations in BRCA1 are also associated with more aggressive disease. In addition to germline mutations in BRCA1/2, somatic mutations in BRCA1/2 and other homologous recombination repair (HRR) genes (eg, ATM, Fanconi anemia, complementation group A [FANCA]) have been shown to occur in advanced prostate cancer, suggesting that a significant percentage of patients with mCRPC may benefit from approaches exploiting a deficiency in HRR, such as treatment with a PARP inhibitor (PARPi).8 A recent clinical study reported that 16 of 49 evaluable patients with advanced heavily pre-treated mCRPC had a response to the PARPi olaparib. Among the 16 evaluable patients in this study with HRR gene mutations, 14 (88%) had a response. Consistent with previous findings, gene mutations were most commonly observed in BRCA2 and ATM. These findings provide compelling evidence for use of a PARPi in a selected population of mCRPC patients with predicted loss-of-function mutations in BRCA1/2 and ATM.

Androgen deprivation therapy is the standard first-line systemic treatment for metastatic prostate cancer. It is highly active with clinical, radiographic and prostate-specific antigen (PSA) responses for most patients – but almost all men will eventually progress to mCRPC. Over the last 10 years, multiple therapies have been shown to confer a survival benefit for patients with mCRPC and were approved on this basis, including docetaxel, cabazitaxel, Sipuleucel-T, radium Ra 223 dichloride, and two agents that target the androgen receptor (AR) pathway, abiraterone acetate and enzalutamide. 10-14 More recently, abiraterone has demonstrated a survival advantage for patients with metastatic high-risk castration-sensitive prostate cancer, 15 and in separate studies, both enzalutamide and apalutamide have demonstrated improvement in metastasis-free survival in patients with non-metastatic castration-resistant prostate cancer. 16, 17 Based on their tolerability and proven efficacy in the pre-chemotherapy setting, abiraterone acetate and enzalutamide are often used as first-line therapies for mCRPC; however, patients progress on these agents after a median duration of 16 to 18 months on treatment. Some patients receive a second regimen of AR-directed therapy; however, response rates are low in this setting. <sup>18-21</sup> For many patients who have progressed on AR-directed therapy, systemic chemotherapy is the next treatment option. Treatment options include docetaxel (75 mg/m<sup>2</sup> every 3 weeks) plus prednisone, cabazitaxel plus prednisone, radium Ra 223 dichloride, and sipuleucel-T. The two latter agents are generally well-tolerated and thus reasonable treatment options for patients prior to receiving treatment with chemotherapy or for patients with bone-only disease.

Despite clinical benefit from AR-directed therapy and chemotherapy, mCRPC patients eventually develop progressive disease. Novel therapies that provide robust clinical benefit and have a good safety profile are still needed for patients with advanced mCRPC, and a targeted therapy such as a PARPi for the subset of patients who exhibit features of HRD represents an attractive option.

# **Primary Objective:**

• To assess the efficacy of rucaparib versus physician's choice of treatment based on radiographic progression free survival (rPFS) in mCRPC patients with HRD who

progressed on prior AR-directed therapy and have not yet received chemotherapy in the castration-resistant setting.

# **Secondary Objectives:**

- To assess overall survival (OS)
- To assess objective response rate (ORR) using modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in patients with measurable (nodal or visceral) disease
- To assess duration of response (DOR) using modified RECIST Version 1.1 in patients with measurable (nodal or visceral) disease
- To assess time to PSA progression
- To assess PSA response  $\geq 50\%$  (all patients)
- To assess PSA response  $\geq 90\%$  (all patients)
- To evaluate Patient-reported Outcome (PRO) using the following instruments:
  - EuroQol 5 dimensions 5 level questionnaire (EQ-5D-5L),
  - Functional Assessment of Cancer Therapy–Prostate (FACT-P),
  - Analgesic drug score, and
  - Brief Pain Inventory–Short Form (BPI-SF) instruments
- To assess clinical benefit rate (CBR)
- To assess sparse pharmacokinetics (PK)
- To assess safety and tolerability

# **Exploratory Objectives:**

- To assess concordance in BRCA/ATM gene mutation status in matched Pre-Screening biopsy tissue, archival primary and metastatic tumor tissue, and plasma circulating cell-free tumor DNA (ctDNA)
- To assess changes in the molecular profile over time of matched pre and post-treatment tumor or plasma samples
- To evaluate loss of heterozygosity (LOH) in metastatic disease site biopsy and archival primary and metastatic tumor tissue samples
- To evaluate mechanisms of response and resistance in ctDNA and progression tumor tissue samples.

# **Study Design**

This is a Phase 3, multicenter, randomized, study of rucaparib versus physician's choice of second-line AR-directed therapy (abiraterone acetate or enzalutamide) or docetaxel as treatment for mCRPC patients who have progressed on one prior AR-directed therapy (abiraterone acetate, enzalutamide, apalutamide, or investigational AR-targeted agent) and have not yet received chemotherapy in the castration-resistant setting. Patients who received prior PARPi treatment will be excluded. This study will enroll mCRPC patients with

deleterious mutations in BRCA1/2 or ATM genes. The primary endpoint is rPFS by central independent radiology review (IRR; rPFSirr) using modified RECIST Version 1.1/ Prostate Cancer Working Group Guidelines Version 3 (PCWG3) criteria.

This study consists of a Pre-Screening Phase, Screening Phase, Randomization, Treatment Phase, Post-Treatment Phase, and Cross-over Phase (if applicable). Patients will receive rucaparib monotherapy or physician's choice of comparator therapy (pre-designated prior to randomization) in the Treatment Phase, and will undergo procedures and assessments including regular safety and efficacy evaluations during the entire conduct of the study. Patients randomized to the control arm in the Treatment Phase will have the opportunity to receive treatment with rucaparib in the Cross-over Phase.

# Pre-Screening Phase

The purpose of the Pre-Screening Phase is to perform central plasma and tumor tissue testing to identify patients with qualifying deleterious BRCA1/2 or ATM gene mutations. If a patient has a qualifying deleterious BRCA1/2 or ATM gene mutation identified from local testing, the Pre-Screening Phase is not required and the patient should proceed to the Screening Phase.

To enter the Pre-Screening Phase, patients should have evidence of radiographic or biochemical disease progression, and be eligible for this study as their immediate next therapy. Patient tissue and plasma samples should be submitted simultaneously during Pre-Screening. Tissue submitted for Pre-Screening testing should be from a newly obtained metastatic biopsy, if there is a lesion suitable for biopsy and the patient consents to this procedure. A biopsy or resection of a visceral or nodal site of metastasis is preferred; however, biopsy of primary tumor or of a site of bony metastasis is also acceptable. If a metastatic biopsy is not feasible, archival tissue samples should be submitted, if available. To reduce the chance of test failure, archival tissue should be < 3 years old.

# Screening Phase

The purpose of the Screening Phase is to perform study-specific screening assessments, other than testing for qualifying deleterious BRCA1/2 or ATM gene mutations. All patients must have a deleterious gene mutation in BRCA1/2 or ATM in order to enter the Screening Phase. Mutations may be identified by local testing, or through central testing provided by the sponsor during the Pre-Screening Phase. For local test results, the classification of the mutation as deleterious must be documented in the patient's medical record.

## Randomization

Eligible patients will be randomized 2:1 to receive rucaparib (600 mg twice a day [BID]) or physician's choice of either docetaxel or AR-directed therapy (abiraterone acetate or enzalutamide, whichever the patient has not yet received). The physician's choice of agent in the control arm must be prespecified prior to randomization.

## **Treatment Phase**

Rucaparib will be administered at a starting dose of 600 mg BID and comparator treatments according to labelling and local practice. Tumor assessments by computed tomography (CT)/magnetic resonance imaging (MRI) and bone scans will be performed during the Screening Phase, at the end of every 8 calendar weeks (± 7 days) from Study Day 1 (Week 1) up to 24 weeks and every 12 calendar weeks (± 7 days) thereafter, and at the Treatment Discontinuation Visit, if applicable. Modified RECIST Version 1.1 criteria will be used to document radiographic response in soft tissue (visceral and nodal) disease and PCWG3 criteria

will be used to document radiographic progression of bone lesions. Any drug modifications (interruption, dose reduction, or discontinuation) should be documented in the electronic case report form (eCRF) and source documents. If study treatment is interrupted, tumor assessments will not be delayed and will proceed on the regular study schedule. Copies of all radiographic scans will be submitted for central IRR until after the analysis of the primary endpoint has been performed, at which time IRR will be discontinued and all radiographic scans will be evaluated by the investigator for radiographic progression.

Patients will receive study drug until radiographic disease progression is confirmed by IRR until analysis of the primary endpoint has been performed, or by investigator assessment after analysis of the primary endpoint has been performed and IRR is discontinued, based on modified RECIST Version 1.1 (for nodal/visceral lesions only) and PCWG3 (for bone lesions only) criteria, unequivocal clinical disease progression, unacceptable toxicity or inability to tolerate further treatment, loss to follow-up, or withdrawal of consent. Patients in the docetaxel arm will receive study drug for a maximum of 10 cycles only and so may not be actively on treatment at the time of disease progression. PSA rise without evidence of confirmed radiographic progression is strongly discouraged as a criterion to start a new systemic antineoplastic therapy during the first 12 weeks of therapy and is discouraged as a criterion to start a new systemic antineoplastic therapy throughout the study. Radiographic assessments will continue until confirmation of radiographic disease progression, irrespective of whether the patient has discontinued study drug treatment or initiated subsequent anticancer therapy. Palliative radiation for treatment of painful bony metastases and initiation of bisphosphonates or other approved bone-targeting agents are allowed and should not result in discontinuation of study drug therapy.

If a patient demonstrates radiographic progression while receiving treatment with study drug, but continues to derive clinical benefit per investigator assessment, then continuation of treatment beyond progression is permitted. In such cases, the patient must consent prior to continuing treatment with study drug.

Safety and efficacy data will be periodically reviewed by an Independent Data Monitoring Committee (IDMC).

## Post-treatment Phase

Upon treatment discontinuation, patients will have a Treatment Discontinuation Visit, a 28-day Follow-up Visit, and then will proceed to long-term follow-up. An optional tumor biopsy will be collected prior to the start of subsequent anticancer therapy from patients who experience radiographic disease progression or unequivocal clinical disease progression and provide appropriate consent.

Radiographic tumor assessments (using the same methodology as was used at initial study screening [eg, CT scan and bone scan]) will continue until radiographic disease progression is confirmed by IRR, irrespective of whether the patient has initiated subsequent anticancer therapy. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR.

Ongoing serious adverse events (SAEs), adverse events of special interest (AESIs), and treatment-related Grade 3/4 adverse events (AEs) will be followed until either resolution or stabilization has been determined or until lost to follow-up. After the 28-day Follow-up Visit,

only SAEs assessed as potentially related to study drug should be reported per Clovis Oncology Pharmacovigilance (PV) requirements and captured in the Clovis Oncology PV database.

After the 28-day Follow-up Visit, **AESIs of myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML), irrespective of causality, should be reported** per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

AESIs of pneumonitis or similar events (ie, interstitial lung disease, pulmonary fibrosis, acute interstitial pneumonitis, alveolitis necrotizing, alveolitis, hypersensitivity pneumonitis, and organizing pneumonia) should be reported up to, but not beyond, the 28-Day Follow-up Visit (28-days after the last dose of rucaparib). After the 28-day Follow-up Visit, only pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements.

All patients will be followed for survival and subsequent treatments every 12 weeks ( $\pm$  14 days) relative to the last dose of study drug until death, loss to follow-up, withdrawal of consent, or study closure.

## Cross-over Phase

Patients randomized to comparator therapy will be given the opportunity to cross-over to receive rucaparib therapy after radiographic progression is confirmed by IRR until analysis of the primary endpoint has been performed, or by investigator assessment after analysis of the primary endpoint has been performed and IRR is discontinued. After providing consent, patients will be assessed to ensure criteria are met for the Cross-over Phase. If eligible, the patient will have protocol assessments per the rucaparib Treatment Phase, as well as including the Post-Treatment Phase.

## Blinding

This is an open-label study; the study drugs will not be blinded or masked to the investigator or patient, so each will know the treatment being administered. A Blinding Plan will be put in place to limit the knowledge of aggregate efficacy data by sponsor personnel.

## **Number of Patients**

The total enrollment planned for this study is approximately 400 patients. A total of approximately 300 patients with a deleterious BRCA1/2 gene mutation will be randomized and approximately 100 patients with a deleterious ATM gene mutation may be randomized. This is a multicenter, multinational study. Patients will be randomized across approximately 150 study sites worldwide.

#### **Inclusion Criteria:**

All patients enrolling into the study must meet all of the following inclusion criteria:

- 1. Have signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form prior to any study-specific evaluation
- 2. Male  $\geq$ 18 years of age at the time the informed consent form is signed

- 3. Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate (pure small-cell histologies or pure high-grade neuroendocrine histologies are excluded; neuroendocrine differentiation is allowed) that is metastatic
- 4. Surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL (1.73 nM). If currently being treated with luteinizing hormone–releasing hormone (LHRH) analogs (patients who have not undergone an orchiectomy), therapy must be continued throughout the study
- 5. Eligible for treatment with physician's choice of comparator treatment, selected prior to randomization, per the corresponding prescribing information
- 6. Evidence of disease progression after treatment with 1 prior next-generation AR-targeted therapy (abiraterone acetate, enzalutamide, apalutamide, or investigational AR-targeted agent); treatment with the older anti-androgen therapies such as bicalutamide, flutamide, and nilutamide are not counted toward this limit
- 7. Disease progression after initiation of most recent therapy is based on <u>any</u> of the following criteria:
  - a. Rise in PSA: a minimum of two consecutive rising levels, with an interval of  $\geq 1$  week between each determination. The most recent screening measurement must have been  $\geq 2$  ng/mL
  - b. Transaxial imaging: new or progressive soft tissue masses on CT or MRI scans as defined by modified RECIST Version 1.1
  - c. Radionuclide bone scan: at least 2 new metastatic lesions
- 8. All patients must have a deleterious gene mutation in BRCA1/2 or ATM. Mutations may be identified by local testing, or through central testing by the sponsor of plasma or tumor tissue. For local test results, the classification of the mutation as deleterious must be documented in the patient's medical record
- 9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
- 10. Have adequate organ function confirmed by the following clinical laboratory values obtained within 14 days prior to the first dose of study drug:
  - a. Bone Marrow Function
    - i. Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^9/L$
    - ii. Platelets  $> 100 \times 10^9/L$
    - iii. Hemoglobin  $\geq 10$  g/dL independent of transfusion within 14 days
  - b. Hepatic Function
    - i. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)  $\leq$  3  $\times$  the upper limit of normal (ULN)
    - ii. Bilirubin  $\leq 1.5 \times \text{ULN}$  ( $< 2 \times \text{ULN}$  if hyperbilirubinemia is due to Gilbert's syndrome)
  - c. Renal Function
    - i. Estimated glomerular filtration rate (GFR) ≥ 45 mL/min using the Cockcroft-Gault formula
- 11. Male patients who are committed to undertaking the following measures for the duration of the study and after the last dose of study drug for the time period specified:

- a. Use a condom during sex while being treated and for 3 months after the last dose of study drug
- b. Do not make semen donations during treatment and for 3 months after the last dose of rucaparib
- c. Those with female partners of childbearing potential may be enrolled if they are:
  - i. Documented to be surgically sterile (ie, vasectomy);
  - ii. Committed to practicing true abstinence during treatment and for 3 months after the last dose of study drug; or
  - iii. Committed to using a highly effective method of contraception (refer to protocol) with their partner during treatment and for 3 months following the last dose of study drug
- 12. Have a life expectancy of at least 6 months

## **Exclusion Criteria:**

Patients will be excluded from participation if any of the following criteria apply:

- 1. Active second malignancy, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
  - a. Patients with a history of malignancy that has been completely treated, and currently with no evidence of that cancer, are permitted to enroll in the study provided all therapy was completed > 6 months prior and/or bone marrow transplant (BMT) > 2 years prior to first dose of rucaparib
- 2. Prior treatment with any PARPi
- 3. Prior treatment with chemotherapy (eg docetaxel, mitoxantrone, cyclophosphamide, platinum-based agents) for mCRPC. Prior treatment with docetaxel (or other taxane chemotherapy) administered for castration-sensitive disease is permitted
- 4. Symptomatic and/or untreated central nervous system (CNS) metastases. Patients with asymptomatic, previously treated CNS metastases are eligible provided they have been clinically stable (not requiring steroids for at least 4 weeks prior to first dose of study drug) and have appropriate scans at screening assessment
- 5. Symptomatic or impending spinal cord compression unless appropriately treated, clinically stable, and asymptomatic
- 6. Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of study drug
- 7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or history of chronic hepatitis B or C, with the exception of patients with sustained virologic response after completion of treatment for hepatitis C
- 8. Received treatment with chemotherapy, antibody therapy, immunotherapy, gene therapy, angiogenesis inhibitors, or experimental drugs within < 14 days prior to first dose of study drug. Treatment with hormonal therapies (with the exception of LHRH analog) must be discontinued at least 7 days prior to the first dose of study drug
- 9. Adverse effect of prior therapy not resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or below with the exception

- of alopecia. Ongoing Grade 2 non-hematologic toxicity related to most recent treatment regimen may be permitted with prior advanced approval from the sponsor
- 10. Initiated low-dose corticosteroid, bisphosphonate, or denosumab therapy or adjusted low-dose corticosteroid, bisphosphonate, or denosumab dose/regimen within < 28 days prior to first dose of study drug. Patients on a stable low-dose corticosteroid, bisphosphonate or denosumab regimen are eligible and may continue treatment
- 11. Non-study related minor surgical procedure within < 5 days, or major surgical procedure within < 21 days, prior to first dose of study drug; in all cases, the patient must be sufficiently recovered and stable before treatment administration
- 12. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry into the study

No waivers of these inclusion or exclusion criteria will be granted by the investigator and the sponsor or its designee for any patient enrolling into the study.

Inclusion/exclusion for entry into the Cross-over Phase of the study are described in the protocol.

#### Randomization

Eligible patients will be randomized 2:1 to receive rucaparib (600 mg BID) or physician's choice (specified prior to randomization) of either docetaxel or AR-directed therapy (abiraterone acetate or enzalutamide, whichever the patient has not yet received). Randomization will occur by a central randomization procedure using an Interactive Response System (IXRS). The following will be included as randomization stratification factors at study entry to ensure treatment groups are balanced:

- ECOG Status 0 vs 1
- Presence of hepatic metastases or not
- BRCA1 vs BRCA2 vs ATM gene mutation

# **Study Treatment**

## Rucaparib:

The starting dose and schedule of rucaparib is 600 mg ingested BID. Patients may take rucaparib with or without food. Each dose should be taken with at least 8 oz (240 mL) of water as close to 12 hours apart as possible, preferably at the same times every day. Rucaparib may be provided as 200, 250 and 300 mg (as free base) dose strength tablets. Tablets should be swallowed whole.

Dose holds or reductions are permitted in the event of unacceptable toxicity.

## Abiraterone acetate plus prednisone:

The starting dose of abiraterone is 1,000 mg orally once a day (QD). No food should be eaten for at least 2 hours before and 1 hour after dosing. Abiraterone should be swallowed whole with water. Prednisone should be administered concomitantly at a dose of 10 mg orally daily.

#### Enzalutamide:

The starting dose of enzalutamide is 160 mg orally QD. Enzalutamide may be taken with or without food. Enzalutamide should be swallowed whole with water.

# **Docetaxel plus prednisone or prednisolone:**

Docetaxel at a dose of 75 mg/m<sup>2</sup> should be administered intravenously (IV) every 3 weeks, for up to a maximum of 10 cycles (whereupon no additional study treatment shall be given, but assessments continue). Docetaxel is given in combination with prednisone or prednisolone 5 mg BID.

Patients will continue with study drug treatment until radiographic disease progression is confirmed by IRR until analysis of the primary endpoint has been performed, or by investigator assessment after analysis of the primary endpoint has been performed and IRR is discontinued, using modified RECIST Version 1.1 and PCWG3 (for bone lesions only) criteria, unequivocal clinical disease progression, unacceptable toxicity or inability to tolerate further treatment, loss to follow-up, or withdrawal of consent.

Dose modifications of comparator drugs are permitted according to the label and local institution treatment guidelines.

If a patient receiving study drug has met criteria for confirmed radiographic disease progression by modified RECIST Version 1.1 and/or PCWG3 criteria, but the patient continues to derive clinical benefit per the investigator, then continuation of treatment will be permitted with additional consent.

#### **Concomitant Medications**

During the study, supportive care (eg, antiemetics; analgesics for pain control) may be used at the investigator's discretion and in accordance with institutional procedures. Supportive care must be recorded for each patient in the appropriate section of the eCRF.

Erythropoietin, darbepoetin alfa, and/or hematopoietic colony-stimulating factors for treatment of cytopenias should be administered per standard of care and according to institutional guidelines. Transfusion thresholds for blood product support will be in accordance with institutional guidelines.

Palliative radiotherapy for the treatment of painful bony metastasis is permitted during the study. Treatment with rucaparib should be held prior to initiation of radiation therapy and until the patient has recovered from any radiation-related toxicity. Radiotherapy to soft-tissue lesions (either target or non-target) renders these inevaluable by RECIST Version 1.1, and is therefore discouraged during the Treatment Phase of the study.

For patients who have not undergone an orchiectomy and are currently being treated with LHRH analogs at the time of consent, therapy must be continued throughout the study.

No other anticancer therapies (including chemotherapy, radiation, antibody, immunotherapy, gene therapy, angiogenesis inhibitors, or other experimental drugs) of any kind will be permitted while the patient is participating in the study with the exception of LHRH analogs and palliative radiotherapy for painful bony metastases.

Initiation of bisphosphonates or other approved bone targeting agents is allowed, if clinically indicated, and should not result in study treatment discontinuation unless patient has radiographic evidence of disease progression.

Herbal and complementary therapies should not be encouraged because of unknown side effects and potential drug interactions.

Based on the results from the cytochrome P450 (CYP) interaction clinical study CO-338-044, rucaparib is a moderate inhibitor of CYP1A2, and a weak inhibitor of CYP2C9, CYP2C19,

and CYP3A, and showed no clinically significant effect on P-gp. Caution should be exercised in the concomitant use of drugs that are sensitive substrates of the above CYP enzymes. Although in vitro rucaparib metabolism mediated by CYP3A4 was slow, a significant contribution of CYP3A4 in vivo cannot be excluded. Caution should be used for concomitant use of strong CYP3A4 inhibitors or inducers.

Patients taking warfarin should have international normalized ratio (INR) monitored regularly according to standard institutional practices, and those patients taking phenytoin should have therapeutic drug level monitored.

In vitro, rucaparib is a potent inhibitor of MATE 1 and MATE2-K, a moderate inhibitor of OCT1, and a weak inhibitor of OCT2. As inhibition of these transporters could decrease renal elimination and decrease liver uptake of metformin, caution is advised when metformin is co-administered with rucaparib.

#### **Treatment Discontinuation Criteria**

A patient must be discontinued from treatment with study drug if <u>any</u> of the following apply:

- unequivocal clinical disease progression;
- unacceptable toxicity or inability to tolerate further treatment;
- loss to follow-up;
- withdrawal of consent.

## **Efficacy Assessments**

Soft tissue (visceral and nodal) disease will be evaluated for evidence of radiographic response based on modified RECIST Version 1.1 criteria. Bone lesions will be followed and evaluated for evidence of radiographic progression based on PCWG3 criteria. Additionally, PSA response will be evaluated.

Tumor assessments will be performed during screening (baseline), at the end of every 8 calendar weeks (± 7 days) relative to Study Day 1 (Week 1) up to 24 weeks, then every 12 calendar weeks (± 7 days), until confirmed radiographic disease progression by modified RECIST Version 1.1 and/or PCWG3 (for bone lesions only) criteria, loss to follow-up, withdrawal, or study closure. Tumor assessments will continue to be performed until radiographic disease progression is confirmed by IRR. After the primary endpoint analysis is performed, confirmation of radiographic progression by IRR will no longer occur and only investigator-assessed radiographic progression performed. If a complete response (CR) or partial response (PR) is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented.

Tumor assessments should consist of clinical examination and appropriate imaging techniques (ie, CT scans of the chest, abdomen, and pelvis with appropriate slice thickness per modified RECIST Version 1.1); other studies (MRI, X-ray, positron emission tomography (PET)/CT, and ultrasound) may also be performed if required. If a site can document that the CT performed as part of a PET/CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast) then the CT portion of the PET/CT can be used for RECIST Version 1.1 measurements. Radionuclide bone scanning (whole body) should be performed using 99mTc-methylene diphosphonate (MDP) or hydroxydiphosphonate (HDP). All sites of disease should be followed and the same methods used to detect lesions at baseline are to be used to follow

the same lesions throughout the clinical study. If a patient has known brain metastases, this disease should be evaluated at each required assessment time.

Copies of CT and bone scans (and other imaging, as appropriate) from the Treatment Phase of the study will be submitted for IRR for all patients. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR. After analysis of the primary endpoint, investigator-assessed radiographic disease progression will be used for cross-over eligibility evaluation. Radiographic assessments from the Cross-over Phase will not be submitted for IRR.

PSA will be measured locally at Screening, each clinic visit, and at the Treatment Discontinuation Visit.

# **Safety Assessments**

Safety and tolerability will be assessed based on the following:

- Incidence, type, seriousness, and severity of AEs reported;
- Clinical laboratory investigations (hematology, serum chemistry and urinalysis);
- Vital signs (blood pressure, pulse, and body temperature);
- 12-lead electrocardiograms (ECGs);
- Physical examinations; and
- ECOG performance status

## **Statistical Methods**

# Sample Size Justification

The total enrollment planned is approximately 400 patients, with approximately 300 patients in the subgroup with a deleterious BRCA1/2 mutation and approximately 100 patients in the subgroup with a deleterious ATM mutation. The median rPFS is assumed to be 6 months for the control arm and 10 months for rucaparib in the subgroup of patients with a deleterious BRCA1/2 mutation and 9 months for rucaparib in the total population. A sample size of approximately 300 patients in the subgroup with a deleterious BRCA1/2 mutation should result in approximately 200 events of rPFS, which will provide approximately 90% power to detect a hazard ratio (HR) of 0.6 at a one-sided 0.025 significance level. A sample size of approximately 400 total patients should result in approximately 270 events of rPFS, which will provide approximately 90% power to detect a HR of 0.67 at a one-sided 0.025 significance level.

# Step-down Procedure of Primary and Secondary Endpoints and General Statistical Considerations

The primary and key secondary endpoints will first be tested among the patients with a deleterious BRCA1/2 mutation and then in the intent-to-treat (ITT) Population (ie, BRCA + ATM) using an ordered step-down multiple comparisons procedure. The primary endpoint of rPFSirr (rPFS by independent radiology review) in the subgroup of patients with a deleterious BRCA1/2 mutation will be tested first at a two-sided 0.05 significance level. If rPFSirr in the subgroup of patients with a deleterious BRCA1/2 mutation is statistically significant, then

rPFSirr will be tested in the ITT Population. Continuing in an ordered step-down manner, the key secondary endpoints of OS and ORR (by IRR) will be tested at the two-sided 0.05 significance level. To preserve the overall Type 1 error rate, statistical significance will only be declared for a secondary endpoint if the primary endpoints and previous secondary endpoints are also statistically significant in the ordered step-down procedure.

Quantitative variables will be summarized using descriptive statistics. For variables registered on a continuous scale, the following will be presented: N, mean, standard deviation (StD), median, minimum and maximum. Categorical variables will be presented using frequencies and percentages. The Kaplan-Meier methodology will be used to summarize time-to-event variables. The stratified HR from the Cox proportional hazards model will be used to estimate the HR between the randomized treatment groups for the primary endpoint.

# **Primary Efficacy Analysis**

rPFSirr is defined as the time from randomization to the first objective evidence of radiographic progression, or death due to any cause (whichever occurs first). Radiographic disease progression includes soft tissue disease progression as per modified RECIST Version 1.1 and confirmed progression of bone disease per PCWG3 criteria. rPFS, as assessed by the investigator (rPFSinv), is defined similarly and will be supportive of the primary endpoint, rPFSirr.

# **Secondary Efficacy Analyses**

Overall survival time will be calculated as the time from randomization to death (by any cause) +1 day. Patients who have not died will be censored on the date the patient was last known to be alive. OS will be analyzed at the time of the primary analysis (interim OS analysis) and again for a final OS analysis when maturity is reached.

ORR is defined as the proportion of patients with a confirmed response of CR or PR using modified RECIST Version 1.1 (ie, CR or PR by IRR assessment and no progression in bone per PCWG3). Per RECIST Version 1.1, to be assigned a best overall response of CR or PR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met.

DOR is defined as the time from the date that a PR or CR is first reported to the time that disease progression is documented including that in bone (modified RECIST Version 1.1/PCWG3 criteria).

Time to PSA progression is defined as the time from randomization to the date that  $a \ge 25\%$  increase and absolute increase of  $\ge 2$  ng/mL above the nadir (or baseline value for patients who did not have a decline in PSA) in PSA was measured. The increase must be confirmed by a second consecutive assessment conducted at least 3 weeks later.

Confirmed PSA response is defined as  $\geq 50\%$  (or  $\geq 90\%$ ) reduction in PSA from baseline to lowest post-baseline PSA result, with a consecutive assessment conducted at least 3 weeks later. PSA response will be calculated for all patients with PSA values at baseline and at least one post-baseline assessment. PSA will be assessed by a local laboratory.

CBR is defined as the combination of CR, PR, and stable disease (SD) as defined by modified RECIST Version 1.1 with no progression in bone per PCWG3 criteria.

## Safety Analyses

AEs, clinical laboratory results, vital signs, ECOG performance status, body weight, and concomitant medications/procedures will be tabulated and summarized. AEs will be

summarized overall and separately for SAEs, AESIs, AEs leading to discontinuation, AEs leading to death, and Grade 3 or higher AEs graded using NCI-CTCAE Version 4.03 or higher. Body weight and vital signs will be summarized descriptively (N, mean, StD, median, minimum, and maximum). ECOG performance status will be summarized categorically. An IDMC will review safety and efficacy data on a periodic basis to ensure an acceptable overall risk and benefit for patients participating in the study.

# **Independent Data Monitoring Committee**

An IDMC with multidisciplinary representation will regularly evaluate benefit-risk during the study, and recommend any potential changes to study conduct. No formal efficacy or futility interim analyses for early stopping are planned; however, OS will be analyzed at the time of the primary analysis (interim OS analysis) and again for a final OS analysis when maturity is reached. The IDMC may recommend that the study be stopped if there is excessive toxicity observed in the rates of serious and/or Grade 3 and 4 AEs.

# **Date of Protocol Amendment 4 Approval:**

18 February 2022

# **TABLE OF CONTENTS**

| 1 | SYNO | OPSIS | | 5 |
|---|---|---|---|---|
| LI | ST OF | IN-TI | EXT TABLES | 23 |
| LI | ST OF | IN-TI | EXT FIGURES | 24 |
| 2 | LIST | OF A | BBREVIATIONS AND DEFINITIONS OF TERMS | 25 |
| 3 | INTR | ODU | CTION | 30 |
| | 3.1 | Inve | stigational Product | 30 |
| | 3.2 | Bac | kground and Rationale for PARP Inhibition | 30 |
| | 3.3 | Met | astatic Castration-resistant Prostate Cancer | 30 |
| | 3. | 3.1 | Treatment of Metastatic, Castration-resistant Prostate Cancer | 31 |
| | 3.4 | Prio | r Experience with Rucaparib | 32 |
| | 3. | 4.1 | Nonclinical Experience with Rucaparib | 32 |
| | 3. | 4.2 | Clinical Experience with Rucaparib | 33 |
| | 3.5 | Rati | onale for this Study of Rucaparib | 43 |
| 4 | STUI | OY OF | BJECTIVES | 45 |
| | 4.1 | Prin | nary Objective | 45 |
| | 4.2 | Seco | ondary Objectives | 45 |
| | 4.3 | Exp | loratory Objectives | 45 |
| 5 | INVE | STIG | ATIONAL PLAN | 46 |
| | 5.1 | Ove | rall Study Design and Plan | 46 |
| | 5. | 1.1 | Pre-Screening Phase | 46 |
| | 5. | 1.2 | Screening Phase | 47 |
| | 5. | 1.3 | Randomization | 47 |
| | 5. | 1.4 | Treatment Phase | 48 |
| | 5. | 1.5 | Post-treatment Phase | 49 |
| | 5. | 1.6 | Cross-over Phase | 50 |
| | 5. | 1.7 | Post-progression Treatment Phase | 50 |
| | 5.2 | Stuc | ly Schema | 50 |
| | 5.3 | End | of Study | 53 |
| 6 | STUI | OY PC | PULATION SELECTION | 53 |
| | 6.1 | Nun | nber of Patients and Sites. | 53 |
| | 6.2 | Incl | usion Criteria | 53 |
| | 6.3 | Exc | lusion Criteria | 55 |
| | 6.4 | | eria for Rucaparib Cross-over Treatment Eligibility Following | |
| | | | iographic Progression on or after Comparator Arm Therapy | |
| | 6.5 | Pati | ents or Partners of Patients Including Those of Reproductive Potential | |
| | 6. | 5.1 | Patients Not on Rucaparib | |
| | 6.6 | Wai | vers of Inclusion/Exclusion Criteria | 58 |

| 7 | STUDY T | REATMENT(S) | 58 |
|---|---|---|---|
| | 7.1 Des | scription of Treatment(s) and Storage | 58 |
| | 7.1.1 | Investigational Drug Product - Rucaparib | 59 |
| | 7.1.2 | Comparator Therapeutic Drug Products | 59 |
| | 7.2 Pac | kaging and Labeling | 59 |
| | 7.2.1 | Rucaparib | 59 |
| | 7.2.2 | Comparator Therapy | 60 |
| | 7.3 Blin | nding | 60 |
| | 7.4 Me | thod of Assigning Patients to Treatment Groups | 60 |
| | 7.5 Pre | paration and Administration of Protocol-specified Treatment | 60 |
| | 7.5.1 | Rucaparib | 61 |
| | 7.5.2 | Single-agent Docetaxel | 64 |
| | 7.5.3 | Single-agent Abiraterone Acetate | 64 |
| | 7.5.4 | Single-agent Enzalutamide | 64 |
| | 7.5.5 | Re-treatment and Dose Modification for All Comparator Therapy | 64 |
| | 7.5.6 | Cross-over to Rucaparib Treatment | 65 |
| | 7.5.7 | Continuation of Study Drug beyond Disease Progression | 65 |
| | 7.6 Tre | atment Compliance | |
| | 7.6.1 | Rucaparib Treatment Compliance | 65 |
| | 7.6.2 | Comparator Therapy Treatment Compliance | 66 |
| | 7.7 Acc | countability of Protocol-specified Treatment | 66 |
| 8 | PRIOR AN | ND CONCOMITANT THERAPY | 67 |
| | 8.1 Sup | pportive Care | 67 |
| | _ | liotherapy | |
| | 8.3 Lut | einizing Hormone-releasing Hormone Analogs | 67 |
| | | ticancer or Experimental Therapy | |
| | 8.5 CY | P450 Isoenzyme Inhibitors, Inducers, and Substrates | 68 |
| | 8.6 The | erapies to Control Bone Loss | 68 |
| | 8.7 An | icoagulants | 68 |
| | | er Concomitant Medications | |
| 9 | STUDY PI | ROCEDURES AND ACTIVITIES BY VISIT | 69 |
| | 9.1 Sch | edule of Assessments | 69 |
| | | ormed Consent. | |
| | 9.3 Pre | -Screening Phase | 79 |
| | | eening Phase | |
| | 9.4.1 | Screening: Up to 28 Days Prior to Randomization: | |
| | 9.4.2 | Screening: Up to 14 Days Prior to Randomization: | |
| | 9.5 Tre | atment Phase | 81 |

| | 9.5 | 5.1 | Patients Randomized to Rucaparib, Physician's Choice of Abiraterone Acetate or Enzalutamide or Cross-over to Rucaparib | <b>Q</b> 1 |
|---|---|---|---|---|
| | 9.5 | 5.2 | Patients Randomized to Physician's Choice of Docetaxel | |
| | 9.6 | | treatment Phase (Randomized Treatment/ Cross-over to Rucaparib) | |
| | 9.6 | | Treatment Discontinuation Visit | |
| | 9.6 | | 28-day Safety Follow-up Visit (Randomized Treatment/ Cross-over to | 00 |
| | | ,. <u> </u> | Rucaparib) | 87 |
| | 9.6 | 5.3 | Long-term Follow-up (Randomized Treatment/ Cross-over to Rucaparib) | 88 |
| | 9.7 | | med Consent for Patients Who Cross-over to Rucaparib after Disease ression on Comparator Treatment | 89 |
| | 9.8 | Scree | ening Prior to Cross-over to Rucaparib | 89 |
| | 9.8 | 3.1 | Ongoing Assessments for Cross-over Patients: | 89 |
| | 9.9 | Meth | ods of Data Collection | |
| | 9.9 | | Medical History and Demographic/ Baseline Characteristics | |
| | 9.10 | | and Concomitant Medication/ Procedure Assessments | |
| | 9.11 | Effic | acy Evaluations | |
| | | 1.1 | Disease/ Tumor Assessments | |
| | 9.12 | | y Evaluations | |
| | _ | 12.1 | Adverse Event Assessment | |
| | | 12.2 | Clinical Laboratory Investigations | |
| | | 12.3 | Vital Signs | |
| | | 12.4 | 12-lead Electrocardiogram. | |
| | | 12.5 | Physical Examinations, Body Weight and Height | |
| | | 12.6 | ECOG Performance Status | |
| | 9.13 | | narker Analysis – FFPE Tumor Tissue | |
| | 9.14 | | narker Analysis – ctDNA/genomic DNA from Blood | |
| | 7.13 | | nacokinetics Evaluation | |
| 10 | 9.16 | | nt-reported Outcomes (Health and Quality of Life Questionnaires) EVENT MANAGEMENT | |
| 10 | 10.1 | | nition of an Adverse Event | |
| | 10.1 | | nition of a Serious Adverse Event. | |
| | 10.2 | | nition of an Adverse Event of Special Interest | |
| | 10.3 | | ts or Outcomes Not Qualifying as Serious Adverse Events | |
| | 10.4 | | cal Laboratory Assessments as Adverse Events and Serious Adverse | ) |
| | 10.5 | | ts | 97 |
| | 10.6 | | nancy or Drug Exposure During Pregnancy | |
| | 10.7 | | rding of Adverse Events, Serious Adverse Events, and Adverse Events of | |
| | | | ial Interest. | 97 |

| | 10 | .7.1 | Onset Date of Adverse Events | 98 |
|---|---|---|---|---|
| | 10 | .7.2 | Resolution Date of Adverse Events | |
| | 10 | .7.3 | Intensity of Adverse Events | 98 |
| | 10 | .7.4 | Causal Relationship of Adverse Events to Study Drug | |
| | 10 | .7.5 | Outcome and Action Taken | |
| | 10.8 | | ow-up of Adverse Events, Serious Adverse Events, and Adverse Events of ial Interest | 100 |
| | 10.9 | | ntial Drug-induced Liver Injury | |
| | 10.10 | Regu | alatory Aspects of Serious Adverse Event and Adverse Events of Special est Reporting | |
| 11 | PLAN | | STATISTICAL METHODS | |
| | 11.1 | | eral Considerations | |
| | 11.2 | | rmination of Sample Size | |
| | 11.3 | | ysis Populations | |
| | 11.4 | | ent Disposition | |
| | 11.5 | | ographics and Baseline Characteristics | |
| | 11.6 | | -down Procedure of Primary and Secondary Endpoints | |
| | 11.7 | | eacy Analyses | |
| | 11 | .7.1 | Primary Efficacy Analysis | |
| | 11 | .7.2 | Secondary Efficacy Analyses | |
| | 11 | .7.3 | Exploratory Efficacy Analyses | 107 |
| | 11.8 | Safe | ty Analyses | 108 |
| | 11 | .8.1 | Adverse Events | 108 |
| | 11 | .8.2 | Clinical Laboratory Evaluations | 109 |
| | 11 | .8.3 | Vital Sign Measurements | 109 |
| | 11.9 | Inter | im Analysis | 110 |
| 12 | PATII | ENT D | DISPOSITION | 110 |
| | 12.1 | Rem | oval of Patients from the Study or Study Drug | 110 |
| 13 | STUD | Y AD | MINISTRATION | 111 |
| | 13.1 | Regu | ulatory and Ethical Considerations | 111 |
| | 13 | .1.1 | Good Clinical Practice. | 111 |
| | 13 | .1.2 | Regulatory Authority Approvals | 112 |
| | 13 | .1.3 | Institutional Review Board or Independent Ethics Committee Approval | 112 |
| | 13.2 | Patie | ent Information and Consent | 113 |
| | 13 | .2.1 | General Aspects of Informed Consent | 113 |
| | 13 | .2.2 | Informed Consent Process | 113 |
| | 13.3 | Patie | ent Confidentiality | 114 |
| | 13.4 | Stud | y Monitoring | 114 |
| | 13.5 | Case | Report Forms and Study Data | 115 |

| 13.6 | Independent Data Monitoring Committee | 116 |
|---|---|---|
| 13.7 | Study Termination and Site Closure | 116 |
| 13.8 | Study Protocol Amendments | 117 |
| 13.9 | Retention of Study Documents | 117 |
| 13.10 | Quality Control and Assurance | 118 |
| 1 | 3.10.1 Protocol Deviations | 118 |
| 1 | 3.10.2 Study Site Training | 118 |
| 1 | 3.10.3 Quality Assurance Audits and Inspections | 118 |
| 1 | 3.10.4 Direct Access to Source Data/ Documents for Audits and Inspections | 118 |
| 13.11 | Clinical Study Report | 119 |
| 13.12 | Publication and Disclosure Policy | 119 |
| 13.13 | Investigator Oversight | 119 |
| 14 REFI | ERENCE LIST | 120 |
| 15 APPI | ENDICES | 125 |
| 15.1 | Appendix 1 - Modified Response Evaluation Criteria in Solid Tumors Criteria (Version 1.1) and Prostate Cancer Working Group 3 Criteria | 126 |
| 15.2 | Appendix 2 - Eastern Cooperative Oncology Group (ECOG) Performance Status Scale | 133 |
| 15.3 | Appendix 3 - Cockcroft-Gault Formula | 134 |
| 15.4 | Appendix 4 - Examples of Sensitive CYP Substrates (not an inclusive list) | 135 |
| 15.5 | Appendix 5 - Brief Pain Inventory – Short Form (BPI-SF) | 136 |
| 15.6 | Appendix 6 - Functional Assessment of Cancer Therapy – Prostate (FACT-P) | 139 |
| 15.7 | Appendix 7 - Euro-Quality of Life 5D 5L (EQ-5D-5L) Patient-reported | |
| | Outcome | 143 |
| 15.8 | Appendix 8 - Analgesic Use Questionnaire | 147 |
| LIST C | F IN-TEXT TABLES | |
| Table 1. | Treatment-emergent AEs (All Grades and ≥ Grade 3) Reported in ≥ 20% of Ovarian Cancer Patients in Combined Studies CO-338-010 and CO-338-017 | 39 |
| Table 2. | Treatment-emergent AEs Reported in ≥ 20% of Patients (All Grades) in Any Treatment Group in Study CO-338-014 - Safety Population | 40 |
| Table 3. | Change from Baseline in Laboratory Parameters in Patients Treated with 600 mg BID Rucaparib (Study CO-338-014) | 42 |
| Table 4. | Rucaparib Dose Reduction Steps | 64 |
| Table 5. | Schedule of Assessments for Patients Randomized to Rucaparib or Physician's Choice of Abiraterone Acetate or Enzalutamide | 70 |
| Table 6. | Schedule of Assessments for Patients Randomized to Physician's Choice of | 73 |

| Table 7. | Schedule of Assessments for Patients Who Cross over to Rucaparib after Physician's Choice Comparator | 76 |
|---|---|---|
| Table 8. | Requirements for Confirmation of Radiographic Disease Progression in Bone per Investigator's Assessment | 91 |
| LIST O | F IN-TEXT FIGURES | |
| Figure 1. | Pre-Screening Study Schema. | 51 |
| Figure 2. | Study Schema: Screening, Treatment, and Post-treatment Phases | 52 |
| Figure 3. | Ordered Step-down Procedure | 105 |

# 2 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| ADP | adenosine diphosphate |
|---|---|
| ADT | androgen deprivation therapy |
| AE | adverse event |
| AESI | adverse event of special interest |
| AIDS | acquired immunodeficiency syndrome |
| ALCOA+ | Attributable, Legible, Contemporaneous, Original or Certified Copy, Accurate, and 'Plus' (+) Complete, Consistent, Enduring, and Available |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| AML | acute myeloid leukemia |
| ANC | absolute neutrophil count |
| ANCOVA | analysis of covariance |
| AR | androgen receptor |
| AST | aspartate aminotransferase |
| ATM | ataxia telangiectasia mutated serine/threonine kinase |
| ATR | ataxia telangiectasia and RAD3-related |
| AUC | area under the concentration-time curve |
| BCRP | breast cancer resistance protein |
| BER | base excision repair |
| BID | twice a day |
| BMT | bone marrow transplant |
| BPI-SF | Brief Pain Inventory–Short Form |
| BRCA | breast cancer 1 or breast cancer 2 gene |
| BRCA1/2 | breast cancer 1 or breast cancer 2 gene |
| BRIP1 | BRCA1-interacting protein |
| BUN | blood urea nitrogen |
| CA-125 | cancer antigen-125 |
| CBR | clinical benefit rate |
| CDK12 | cyclin-dependent kinase 12 |
| CFR | Code of Federal Regulations |
| CHEK2 | checkpoint kinase 2 |
| CI | confidence interval |
| CLIA | Clinical Laboratory Improvement Amendments |
| C <sub>max</sub> | maximum plasma concentration |
| C <sub>min</sub> | trough concentration |
| СМН | Cochran-Mantel-Haenszel |

| CNS | central nervous system |
|----------|--------------------------------------------------|
| $CO_2$ | bicarbonate |
| CR | complete response |
| CRO | contract research organization |
| CSR | clinical study report |
| CT | computed tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ctDNA | circulating cell-free tumor DNA |
| CYP | cytochrome P450 |
| DILI | drug-induced liver injury |
| DNA | deoxyribonucleic acid |
| DOR | duration of response |
| DSB | double-strand breaks |
| EC | European Commission |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EMA | European Medicines Agency |
| EOC | epithelial ovarian cancer |
| EQ-5D-5L | EuroQol 5 dimensions 5 level questionnaire |
| EU | European Union |
| FACT-P | Functional Assessment of Cancer Therapy–Prostate |
| FANCA | Fanconi anemia, complementation group A |
| FDA | Food and Drug Administration |
| FFPE | formalin-fixed paraffin-embedded |
| FSH | follicle-stimulating hormone |
| FTC | fallopian tube cancer |
| gBRCA | germline breast cancer 1 or 2 gene mutation |
| GCIG | Gynecologic Cancer InterGroup |
| GCP | Good Clinical Practice |
| GDPR | General Data Protection Regulation |
| GFR | glomerular filtration rate |
| Hct | hematocrit |
| HDL | high density lipoprotein |
| HDP | hydroxydiphosphonate |
| HDPE | high-density polyethylene |
| | - |

| Hgb | hemoglobin |
|---|---|
| HIPAA | Health Information Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HR | hazard ratio |
| HRD | homologous recombination deficiency |
| HRR | homologous recombination repair |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IDMC | Independent Data Monitoring Committee |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug Application |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| invPFS | investigator-assessed progression-free survival |
| IRB | Institutional Review Board |
| IRR | central independent radiology review |
| ITT | intent-to-treat |
| IUD | intrauterine device |
| IUS | intrauterine hormone-releasing system |
| IV | intravenous(ly) |
| IXRS | Interactive Response System |
| LD | longest diameter |
| LDH | lactate dehydrogenase |
| LDL | low density lipoprotein |
| LHRH | luteinizing hormone-releasing hormone |
| LOH | loss of heterozygosity |
| MATE | multidrug and toxin extrusion protein |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| mCRPC | metastatic castration-resistant prostate cancer |
| MCV | mean corpuscular volume |
| MDP | methylene diphosphonate |
| MDS | myelodysplastic syndrome |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Modified<br>RECIST | Response Evaluation Criteria in Solid Tumors modified according to PCWG3 guidelines (used for evaluation of nodal/visceral disease, excluding bone disease) |

| Modified<br>RECIST/PCWG3 | Response Evaluation Criteria in Solid Tumors modified according to PCWG3 guidelines, combined with evaluation of bone disease according to PCWG3 |
|---|---|
| MRI | magnetic resonance imaging |
| NBN | nibrin |
| NCI | National Cancer Institute |
| OCT | organic cationic transporter |
| ORR | objective response rate |
| OS | overall survival |
| PALB2 | partner and localizer of BRCA2 |
| PARP | poly (ADP-ribose) polymerase |
| PARPi | PARP inhibitor |
| PCWG3 | Prostate Cancer Working Group Guidelines Version 3 |
| PD | progressive disease (in context of disease monitoring) |
| PD | pharmacodynamic (in context of pharmacology discussion) |
| PET | positron emission tomography |
| PFS | progression-free survival |
| P-gp | P-glycoprotein |
| PIS | Patient Information Sheet |
| PK | pharmacokinetic |
| PPC | primary peritoneal cancer |
| PPI | proton pump inhibitor |
| PR | partial response |
| PRO | patient-reported outcome |
| PSA | prostate-specific antigen |
| PT | Preferred Term |
| PV | pharmacovigilance |
| QD | once a day |
| RAD51B | RAD51 homolog B |
| RAD51C | RAD51 homolog C |
| RAD51D | RAD51 homolog D |
| RBC | red blood cell |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| rPFS | radiographic progression-free survival |
| rPFSinv | radiographic progression-free survival by the investigator |
| rPFSirr | radiographic progression-free survival by IRR |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| sBRCA | somatic breast cancer gene 1 or 2 mutation |

| SD | stable disease |
|---|---|
| SOC | system organ class |
| SOP | standard operating procedure |
| SSB | single-strand break |
| StD | standard deviation |
| SUSAR | suspected unexpected serious adverse reactions |
| tBRCA | tumor tissue mutation in BRCA1 or BRCA2, includes gBRCA and sBRCA |
| TEAE | treatment-emergent adverse event |
| TMZ | temozolomide |
| UDP | uridine diphosphate |
| UGT1A1 | UDP-glucuronosyl transferase 1A1 |
| ULN | upper limit of normal |
| Upper case<br>gene/protein<br>names | Gene and protein names should be in italics and plain text, respectively, based on HUGO Gene Nomenclature Committee guidelines. However, in this document mutations which occur at both the gene and protein level are often discussed. Therefore for enhanced readability, gene and protein names are written in plain text |
| US | United States |
| VAS | visual analog scale |
| WBC | white blood cells |
| WHO | World Health Organization |
| XO | cross-over |

## 3 INTRODUCTION

# 3.1 Investigational Product

Rucaparib (CO-338) is a small molecule inhibitor of poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) being developed for the treatment of cancer associated with homologous recombination deficiency (HRD). Rucaparib has been shown to potently inhibit PARP-1, PARP-2, and PARP-3 and has demonstrated activity in cells, animal models and patients with a breast cancer gene 1 or 2 (BRCA1 and BRCA2) mutations in both clinical and nonclinical studies.

Clovis Oncology, Inc. is developing rucaparib for oral administration in patients with metastatic castration-resistant prostate cancer (mCRPC) associated with HRD, including patients with a deleterious mutations in BRCA1, BRCA2 and ataxia telangiectasia mutated serine/threonine kinase (ATM) and other homologous recombination repair (HRR) gene mutations.

# 3.2 Background and Rationale for PARP Inhibition

Deoxyribonucleic acid (DNA) is constantly damaged by both endogenous and exogenous (environmental) assaults. Endogenous causes include spontaneous base changes, replication errors, and oxygen-free radicals. Exogenous agents of DNA damage include chemicals and both ultraviolet and ionizing radiation. A common type of DNA damage is the formation of DNA single-strand breaks (SSBs). Normal cells repair SSBs in DNA through a process known as base excision repair (BER). While there are several variations of BER, all pathways rely on the activity of PARP enzymes. In humans, the PARP family encompasses 17 enzymes, of which PARP-1 is the best characterized.<sup>22</sup> SSBs that are not repaired result in stalled replication forks and the development of double-strand breaks (DSBs), which are in turn repaired by HRR, a complex process involving multiple proteins, including BRCA1 and BRCA2, as well as RAD51, Fanconi anemia core complex, ATM, and ataxia telangiectasia and RAD3-related (ATR) protein, among others. Thus, HRR processes act as a functional buffer to enable normal cells to survive the effects of PARP and BER inhibition and overcome DSB in DNA. Homologous recombination defects or PARP inhibition on their own can be overcome by a cell, but the combination is fatal, a concept termed "synthetic lethality", which forms the basis of the therapeutic approach of using PARP inhibition to kill cancer cells with HRD. 1-3

# 3.3 Metastatic Castration-resistant Prostate Cancer

Prostate cancer is the most common malignancy among men in the United States (US), and the second-most common cause of cancer-related mortality, with approximately 30,000 men dying of the disease each year. Based upon GLOBOCAN 2012 estimates, prostate cancer is the second leading malignancy diagnosis and fifth leading cause of death in men worldwide, with 307,000 deaths estimated in 2012. The course of prostate cancer from diagnosis to death is often a series of clinical states progressing from localized disease to mCRPC, a disease state characterized by resistance to standard androgen deprivation therapies and that accounts for the majority of prostate cancer deaths.

HRD has been observed in many carcinomas, including prostate cancer. Men with a germline mutation in BRCA2 are at increased risk for developing prostate cancer, estimated at 2.5 to 8.6-fold compared with non-carriers. 6 Men with prostate cancer and a germline mutation in BRCA2 typically develop disease at a younger age, have more aggressive features and higher mortality rates; while less common in prostate cancer, germline mutations in BRCA1 are also associated with more aggressive disease. In addition to germline mutations in breast cancer 1 or breast cancer 2 gene (BRCA1/2), somatic mutations in BRCA1/2 and other HRR genes have been shown to occur in advanced prostate cancer. A large genomic study of mCRPC identified a 12.7% rate of mutation/deletion in BRCA2 (of which over 90% was biallelic), half of which was a germline mutation in BRCA2; a 7% rate of loss of ATM, an approximately 5% mutation rate of cyclin-dependent kinase 12 (CDK12), a previously-reported positive regulator of BRCA genes, and lower rates of mutation of BRCA1, Fanconi anemia, complementation group A (FANCA), RAD51 homolog B (RAD51B), RAD51 homolog C (RAD51C), and other HRR genes. Overall, almost 23% of tumors were found to have a mutation in at least one HRR gene, and over 19% of tumors had either a BRCA1/2 or ATM mutation, suggesting that in principle a significant percentage of patients with mCRPC may benefit from approaches exploiting a deficiency in homologous recombination repair, such as treatment with a PARP inhibitor (PARPi).8 A recent clinical study reported that 16 of 49 evaluable patients with advanced heavily pre-treated mCRPC had a response to the PARPi, olaparib. Response was defined as a Response Evaluation Criteria in Solid Tumors (RECIST) partial response (PR) or complete response (CR), circulating tumor cell reduction from 5 or more to less than 5 per 7.5 mL of blood, or 50% decrease in prostate-specific antigen (PSA). Fourteen of the 16 responders had a mutation in a HRR gene, most commonly BRCA2 and ATM. These findings provide compelling evidence for use of a PARPi in a selected population of mCRPC patients with predicted loss-of-function mutations in HRR genes such as BRCA1/2 and ATM.

# 3.3.1 Treatment of Metastatic, Castration-resistant Prostate Cancer

Androgen deprivation therapy (ADT) is the standard first-line systemic treatment for metastatic prostate cancer. It is highly active with clinical, radiographic and PSA responses for most patients – but almost all men will eventually progress to mCRPC. Over the last 10 years, multiple therapies have been shown to confer a survival benefit for patients with mCRPC and were approved on this basis, including docetaxel, cabazitaxel, Sipuleucel-T, radium Ra 223 dichloride, and two agents that target the androgen receptor (AR) pathway, abiraterone acetate and enzalutamide. More recently, abiraterone has demonstrated a survival advantage for patients with metastatic high-risk castration-sensitive prostate cancer, and in separate studies, both enzalutamide and apalutamide have demonstrated improvement in metastasis-free survival in patients with non-metastatic castration-resistant prostate cancer. 16, 17

Based on their tolerability and proven efficacy in the pre-chemotherapy setting, abiraterone acetate and enzalutamide have become common first-line therapies for mCRPC; however, patients progress on these agents after a median duration of 16 to18 months treatment. Response rates to a second regimen of AR-directed therapy are low, <sup>18-21</sup> therefore systemic chemotherapy is often considered as the next treatment option for patients who have progressed on AR-directed therapy. Docetaxel (75 mg/m² every 3 weeks) plus prednisone demonstrated good activity (45% PSA response rate and 19.2 months overall survival [OS]) in chemotherapy-naïve mCRPC patients who progressed on ADT, but has generally been replaced by abiraterone acetate and

enzalutamide as first-line treatment for mCRPC. Docetaxel appears to be less effective in the post-abiraterone or enzalutamide setting, with median progression-free survival (PFS) of approximately 4.5 months. <sup>19</sup> It is also associated with significant toxicity, including Grade 3/4 neutropenia, fatigue, sensory neuropathy, stomatitis, diarrhea and fatigue. <sup>14</sup> Cabazitaxel plus prednisone is a treatment option following docetaxel-based treatment based on demonstrated OS benefit versus mitoxantrone (median of 15.1 versus 12.7 months, hazard ratio [HR] 0.70 (95% confidence interval [CI] 0.59-0.83, p < 0.0001) in mCRPC patients who progressed on both ADT and docetaxel therapy, but it is also associated with significant Grade 3/4 neutropenia and diarrhea. <sup>23</sup> Radium Ra 223 dichloride received approval for treatment of mCRPC based on OS benefit (median of 14 versus 11.2 months for placebo) in patients who had bone, but not visceral disease. <sup>24</sup> Sipuleucel-T extended median OS in mCRPC by 4.1 months compared to placebo, <sup>25</sup> but its effectiveness is not known in the post-abiraterone/enzalutamide and post-docetaxel setting. Both agents are generally well-tolerated and thus reasonable treatment options for patients prior to receiving treatment with chemotherapy or for patients with bone-only disease.

Nevertheless, novel therapies that provide robust clinical benefit and have a good safety profile are still needed for patients with advanced mCRPC, and a targeted therapy such as a PARPi for the subset of patients who exhibit features of HRD represents an attractive option.

# 3.4 Prior Experience with Rucaparib

Refer to the current rucaparib Investigator's Brochure (IB) for the latest relevant nonclinical and clinical information regarding rucaparib, including the status of ongoing and completed clinical studies.

An overview of data from nonclinical and clinical studies with rucaparib are summarized below. More current additional detail is provided in the rucaparib Investigator's Brochure (IB). A summary of the benefits and risks of rucaparib treatment are also provided in the rucaparib IB. The nonclinical and clinical data and benefits and risks of rucaparib have been consistent over time.

## 3.4.1 Nonclinical Experience with Rucaparib

The results from nonclinical studies are consistent with the anticipated mechanism of action and pharmacological effects of PARP inhibition.

Pharmacological assessment demonstrated that rucaparib is a potent and selective inhibitor of PARP-1, PARP-2, and PARP-3 and has robust and durable in vitro and in vivo activity in multiple BRCA1/2 mutant cell lines and xenograft models. Rucaparib was also active in a BRCA wild-type model, consistent with in vitro data suggesting that rucaparib is active in cells with other defects in HRR through synthetic lethality. In vitro screens suggested that rucaparib has a limited potential for off-target effects. Safety pharmacology studies suggest that when given orally, rucaparib poses a low risk for causing neurobehavioral and cardiac effects in patients.

In pharmacokinetic (PK) studies, rucaparib demonstrated species-dependent oral bioavailability, moderate plasma protein binding, and large volumes of distribution in nonclinical species. As a P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) substrate, rucaparib

demonstrated minimal penetration of rucaparib-derived radioactivity through the blood-brain barrier. In vitro data suggested slow metabolism by cytochrome P450 (CYP) enzymes, with CYP2D6 and to a lesser extent CYP1A2 and CYP3A4 contributing to the metabolism of rucaparib. Rucaparib was mainly excreted in feces in rats and dogs. In vitro, rucaparib reversibly inhibited CYP1A2, CYP2C19, CYP2C9, and CYP3A, and to a lesser extent CYP2C8, CYP2D6, and UDP-glucuronosyltransferase 1A1 (UGT1A1). Rucaparib induced CYP1A2, and down-regulated CYP2B6 and CYP3A4 in human hepatocytes at clinically relevant exposures. Rucaparib is a potent inhibitor of multidrug and toxin extrusion protein 1 (MATE1) and MATE2-K, a moderate inhibitor of organic cationic transporter 1 (OCT1), a weak inhibitor of OCT2, and may inhibit P-gp and BCRP in the gut.

Oral dosing of rucaparib in single and repeat dose toxicity studies in rats and dogs resulted in toxicity to the hematopoietic, lymphopoietic, and gastrointestinal systems. These toxicities were generally both reversible upon recovery and predictive of toxicities observed in patients. Rucaparib was shown to be clastogenic in an in vitro chromosomal aberration assay suggesting potential genotoxicity in humans. Reproductive and development toxicity studies in rat showed that rucaparib caused maternal toxicity and was embryo-toxic. Although no rucaparib related effects on sperm total count, density, motility, or morphology were identified, based on published studies, PARP inhibitors have the potential to impair spermatogenesis and reduce fertility. <sup>26-29</sup>

# 3.4.2 Clinical Experience with Rucaparib

Rucaparib has been evaluated in Phase 1, 2, and 3 clinical studies and is being evaluated in ongoing Phase 1, 2, and Phase 3 clinical studies. The early clinical program assessed safety and efficacy of rucaparib in patients with malignancies commonly treated with chemotherapeutic agents. Initially, an intravenous (IV) formulation of rucaparib was administered in combination with a variety of chemotherapies; later, the oral formulation of rucaparib was administered in combination with chemotherapy and as a monotherapy. The oral formulation as monotherapy is the focus of current development efforts. The IV formulation is no longer in use.

On 19 December 2016, under priority and expedited review, the US Food and Drug Administration (FDA) granted accelerated approval for the marketing of rucaparib (Rubraca®) for monotherapy treatment of patients with deleterious breast cancer susceptibility gene (BRCA) mutation (germline and/or somatic) associated advanced ovarian cancer who have been treated with 2 or more chemotherapies and on 06 April 2018 Rubraca was approved for use as monotherapy maintenance treatment for adult patients with recurrent epithelial ovarian (EOC), fallopian tube cancer (FTC), or primary peritoneal cancer (PPC) who are in response (complete or partial) to platinum-based chemotherapy. On 29 May 2018, the European Commission (EC) authorized oral rucaparib as monotherapy treatment of adult patients with platinum-sensitive, relapsed or progressive, BRCA-mutated (germline and/or somatic), high-grade EOC, FTC, or PPC, who have been treated with 2 or more prior lines of platinum-based chemotherapy, and who are unable to tolerate further platinum-based chemotherapy.

The latest summary information on indications and ongoing/completed clinical studies is provided in the rucaparib IB. Information below is current as of 27 August 2020.

Six studies (A4991002, A4991005, A4991014, CO-338-010, CO-338-023 [RUCAPANC], and CO-338-045 [ADME]) have been completed and 6 studies in addition to the one described in this protocol are ongoing (CO-338-014 [ARIEL3], CO-338-017 [ARIEL2], CO-338-043 [ARIEL4], CO-338-044 [DDI], CO-338-052 [Phase 2 mCRPC], and CO-338-078 [hepatic impairment study]).

Details of all completed, ongoing, and planned studies are described briefly below. Additional information is provided in the rucaparib IB.

# **Completed Studies**

- A4991002: a Phase 1 open-label, dose-escalation study of IV rucaparib in combination with temozolomide (TMZ) in patients with advanced solid tumors (Part 1) or malignant melanoma (Part 2).
- A4991005: a Phase 2, open-label study of IV rucaparib in combination with TMZ in patients with metastatic melanoma.
- A4991014: a Phase 1, open-label, dose-escalation study of IV and oral rucaparib administered with different chemotherapeutic agents in patients with an advanced solid tumor.

CO-338-023 (RUCAPANC): a Phase 2, single-arm, open-label study of monotherapy oral rucaparib as treatment for patients with previously treated locally advanced or metastatic pancreatic ductal adenocarcinoma and a known deleterious BRCA mutation.

- CO-338-010: 3-part, open-label, Phase 1/2 study of monotherapy oral rucaparib.
  - Part 1: a Phase 1 portion evaluating PK and safety of escalating doses of rucaparib in patients with solid tumors; this portion identified 600 mg twice a day (BID) as the recommended starting dose for future studies (n = 56; completed).
  - Part 2: a Phase 2 portion evaluating the efficacy and safety of rucaparib in patients with relapsed, high-grade ovarian cancer associated with a BRCA mutation.
    - Part 2A enrolled patients with a gBRCA mutation who had received 2 to 4 prior treatment regimens (n = 42; enrollment complete).
    - Part 2B enrolled patients with a gBRCA or sBRCA mutation who received at least 3 prior chemotherapy regimens (n = 12; enrollment complete).
  - Part 3: a Phase 2 portion in patients with a relapsed solid tumor associated with a BRCA mutation in order to characterize the PK, food effect, and safety profile of a higher dose strength tablet (n = 26; enrollment complete).
- CO-338-045 (ADME study): a Phase 1 mass balance study of  $[^{14}C]$ -rucaparib in patients with an advanced solid tumor (n = 6; completed).

# **Ongoing Studies**

• CO-338-017 (ARIEL2): a 2-part open-label Phase 2 study of monotherapy oral rucaparib for treatment of relapsed, high-grade ovarian cancer patients. It is designed to identify tumor characteristics that may predict sensitivity to rucaparib. Patients will be classified into

molecularly-defined subgroups, including tumor BRCA (tBRCA, inclusive of both germline and somatic BRCA) and BRCA-like, by a prospectively defined genomic signature.

- Part 1 enrolled patients with platinum-sensitive, relapsed disease who received  $\geq 1$  prior platinum regimen (n = 204; enrollment complete).
- Part 2 enrolled patients with relapsed disease who received at least 3 prior chemotherapy regimens (n = 287 enrollment complete).
- CO-338-014 (ARIEL3): a Phase 3, randomized, double-blind study of monotherapy oral rucaparib versus placebo as switch maintenance treatment in patients with platinum-sensitive-, relapsed, high-grade ovarian cancer who achieved a response to platinum-based chemotherapy (n = 564 [randomized patients; rucaparib n = 375; placebo n = 189]; enrollment complete).
- CO-338-043 (ARIEL4): a Phase 3, randomized study of rucaparib versus chemotherapy in patients with relapse, BRCA-mutant, high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer (n = 345 planned).
- CO-338-044 (DDI study): a 2-part, Phase 1, open-label, multiple-probe drug-drug interaction (DDI) study to determine the effect of rucaparib on PK of caffeine, S-warfarin-, omeprazole, midazolam, and digoxin in patients with advanced solid tumors in Part 1, followed by optional continued treatment with rucaparib in Part 2 (n = 17; enrollment complete).
- CO-338-052 (TRITON2): a Phase 2 study evaluating rucaparib for treatment of patients with mCRPC whose tumors are associated with HRD by enrolling mCRPC patients with mutations in BRCA1/2, ATM, or other HRR genes. All patients will be required to have progressed on prior AR-targeted therapy (abiraterone acetate, enzalutamide, or investigational AR-targeted agent) and also have progressed after one prior taxane-based chemotherapy for mCRPC (n = 350 planned; enrollment ongoing)
- CO-338-078 (hepatic impairment study): a Phase 1, clinical pharmacology study in patients with an advanced solid tumor and normal or moderately impaired hepatic function to assess the effect of hepatic function on rucaparib PK.

# 3.4.2.1 Overview of Pharmacokinetics and Drug-Drug Interactions

An overview of data are provided below and described in detail in the rucaparib IB.

Assessment of rucaparib PK in cancer patients showed an approximate dose proportional exposure after once a day (QD) or BID dosing, rapid absorption with maximum plasma concentration ( $C_{max}$ ) achieved within 1.5 to 6 hours, and distribution into tissue. The oral bioavailability was 36% and elimination ranged from 11 to 29.8 hours. Rucaparib was moderately bound to human plasma proteins in vitro.

At a dose of 600 mg BID rucaparib, steady state was achieved after approximately 1 week. The absolute oral bioavailability was 37.2%. In the presence of a high-fat meal, there was a slight delay in absorption, but an overall increase in exposure and oral bioavailability (51.7% [fed] vs. 36.2% [fasted]).

In vitro, CYP enzymes were shown to contribute to rucaparib metabolism. In a preliminary assessment of rucaparib metabolism in patients, rucaparib biotransformation pathways included hydroxylation or oxidation, N-demethylation, deamination, and phase II methylation. A
carboxylic acid metabolite (M324) and a phase II N-methylated metabolite of M324 (M338) were identified as major metabolites.

#### POPULATION PK ANALYSES

Drug interactions with rucaparib as a substrate were assessed in a population PK analysis. CYP2D6 phenotypes (poor metabolizers, intermediate metabolizers, normal metabolizers, and ultra-rapid metabolizers) and CYP1A2 phenotypes (normal metabolizers and hyperinducers) did not significantly impact the steady-state exposure of rucaparib at 600 mg BID. Concomitant administration of strong CYP1A2 or CYP2D6 inhibitors did not significantly impact rucaparib PK. Current smokers had overlapping rucaparib exposures as compared to nonsmokers and former smokers. Collectively, the results suggest that CYP1A2 and CYP2D6 play limited role in rucaparib metabolism in vivo, and no rucaparib dose adjustment is needed when concomitantly administered with CYP1A2 or CYP2D6 inhibitors.

In vitro, rucaparib is a substrate of P-gp and BCRP. Concomitant usage of strong P-gp inhibitors did not affect rucaparib PK. Effect of BCRP inhibition on rucaparib PK has not been studied. Concomitant treatment with proton pump inhibitors (PPIs) did not show clinically significant effect on rucaparib PK. No dose modification is recommended based on use PPIs.

#### EFFECT OF RUCAPARIB ON THE PHARMACOKINETICS OF OTHER DRUGS

In the "cocktail" drug-drug interaction study CO-338-044, the effects of steady-state rucaparib at 600 mg BID on CYP1A2, CYP2C9, CYP2C19, CYP3A, and P-gp were evaluated with single oral doses of sensitive probes (caffeine, S-warfarin, omeprazole, midazolam, and digoxin, respectively). Data suggest that rucaparib is a moderate inhibitor of CYP1A2, a weak inhibitor of CYP2C9, CYP2C19, and CYP3A. Rucaparib also marginally inhibited P-gp in the gut but the effect is unlikely clinically significant. Details and results of study CO-338-044 are provided in the rucaparib IB.

#### 3.4.2.2 Overview of Efficacy

An overview of data are provided below and described in detail in the rucaparib IB.

Efficacy analysis was based on pooled efficacy data from 106 patients with BRCA mutant ovarian cancer, who received two or more prior chemotherapy regimens, and who initiated treatment with rucaparib at 600 mg BID in Part 2A of Study CO-338-010 and Parts 1 and 2 of Study CO-338-017. The enrollment cut-off date was 1 October 2015 (all 42 patients enrolled) and the visit data cut-off date was 30 November 2015 for Study CO-338-010 Part 2A. The enrollment cut-off was a 1 October 2015 and the visit data cut-off was 29 February 2016 for Part 1 (24 patients) and Part 2 (40 patients) of Study CO-338-017.

Efficacy data indicate that many patients with advanced ovarian cancer associated with a BRCA1/2 gene mutation and who had two or more prior therapies achieve RECIST Version 1.1 and/or Gynecologic Cancer InterGroup (GCIG) cancer antigen-125 (CA-125) responses. The confirmed objective response rate (ORR) per RECIST Version 1.1 by investigator review was 53.8% (57/106) and the confirmed response by RECIST Version 1.1 or GCIC CA-125 was

70.8% (75/106). The confirmed ORR per RECIST Version 1.1 by independent review was 41.5% (44/106).

In addition, patients without a BRCA1/2 gene mutation in tumor tissue are also deriving benefit, with 43% achieving RECIST Version 1.1 and/or GCIG CA-125 responses.

In the Phase 3, randomized, double-blind study of monotherapy oral rucaparib versus placebo as switch maintenance treatment in patients with platinum-sensitive, relapsed, high-grade ovarian cancer who achieved a response to platinum-based chemotherapy (ARIEL3), the primary efficacy endpoint was investigator-assessed PFS (invPFS) by RECIST Version 1.1. Three patient populations (tBRCA, HRD, and intent-to-treat [ITT]) were evaluated in a step-down analysis.

The primary endpoint was achieved as of 15 April 2017 with a highly statistically significant difference in invPFS between rucaparib treatment as compared to placebo for each of the 3 stratified primary efficacy analysis populations (p < 0.0001 for each population). The median invPFS in the tBRCA population was 16.6 months (95% CI, 13.4-22.9) for the rucaparib group and 5.4 months (95% CI, 3.4-6.7) for the placebo group. Additional data in HRD and ITT populations are available in the rucaparib IB.

For each of the 3 populations, the confirmed investigator-assessed ORR, per RECIST Version 1.1, in patients with measurable disease at baseline was statistically significantly higher in the rucaparib group compared to the placebo group. In the tBRCA population, the confirmed ORR was 15/40~(37.5%) for the rucaparib group and 2/23~(8.7%) for the placebo group (p = 0.0055). Additional data in HRD and ITT populations are available in the rucaparib IB.

Three mCRPC patients with a BRCA mutation received rucaparib monotherapy in Study CO-338-010 or under named patient access, most of whom experienced tumor stabilization, decrease of PSA levels, and symptom improvement.

#### 3.4.2.3 Overview of Safety

An overview of data are provided below and described in detail in the rucaparib IB.

# **Integrated Safety Analysis in the Treatment Setting (Studies CO-338-010 and CO-338-017)**

An integrated safety analysis, based on pooled safety data from 545 patients in Study CO-338-010 (Parts 2A and 2B) and Study CO-338-017 (ARIEL2; Parts 1 and 2) with relapsed ovarian cancer who were treated with 600 mg BID monotherapy rucaparib, was performed and a summary of treatment-emergent adverse events (TEAEs), overall and ≥ Grade 3, is presented in Table 1. This analysis includes data as of 1 September 2017. Overall, the median duration of treatment was 160.0 days (approximately 5.3 months; range, 2 to 1234 days).

The most common TEAEs reported were primarily mild to moderate (Grade 1 to 2) in severity and included gastrointestinal disorders (nausea [78.5%], vomiting [45.9%], constipation [37.6], abdominal pain (32.5%), and diarrhea [32.3%]), asthenia/fatigue (75.0%), anemia/decreased haemoglobin (44.0%), ALT/AST increased (39.3%), decreased appetite (38.3%), and dysgeusia (36.7%).

The most common treatment-related TEAEs reported were primarily mild to moderate (Grade 1 to 2) in severity and included nausea (68.3), asthenia/fatigue (67.0%), anemia/decreased haemoglobin (38.9%), alanine aminotransferase (ALT)/aspartate aminotransferase (AST) increased (36.5%), dysgeusia (34.1%), and vomiting (31.6%) as described in greater detail in the rucaparib IB.

The most common TEAEs  $\geq$  Grade 3 were anemia/decreased hemoglobin (24.2%), asthenia/fatigue (11.7%), ALT/AST increased (10.8%), thrombocytopenia/decreased platelets (6.1%), and nausea (5.3%). As of the data cut-off date, approximately 9% of patients had discontinued due to a treatment-related TEAE.

In addition, photosensitivity has been reported in some patients. Photosensitivity was initially reported in the Phase 1 dose-escalation portion of Study CO-338-010 (n = 6; 10.7%) and based on these reports of photosensitivity, guidance for sun protection was included in rucaparib clinical studies. Of 917 patients with advanced ovarian cancer treated with rucaparib 600 mg BID in Studies CO-338-014 (ARIEL3), CO-338-010, and CO-338-017 (ARIEL2), 118 patients (12.9%) experienced photosensitivity, of whom 2 patients (0.2%) experienced ≥ Grade 3 photosensitivity as described in the rucaparib IB. Patients should use typical precautions when going outside, such as applying sunscreen (sun protection factor 50 or greater) and/or covering exposed skin with clothing and wearing a hat and sunglasses.

Effects on cardiac channel activity in vitro and a comprehensive assessment of the effects of rucaparib on electrocardiogram (ECG) parameters in cancer patients demonstrated a low risk of cardiac effects by rucaparib.

Table 1.

| Preferred Term <sup>a</sup> | 600 mg BID Rucaparib (N = 409) <sup>b</sup><br>n (%) | |
|---|---|---|
| | All Grades | ≥ Grade 3 |
| Nausea | 428 (78.5) | 29 (5.3) |
| Asthenia/fatigue <sup>c</sup> | 409 (75.0) | 64 (11.7) |
| Vomiting | 250 (45.9) | 23 (4.2) |
| Anemia/decreased hemoglobin <sup>c</sup> | 240 (44.0) | 132 (24.2) |
| ALT/AST increased <sup>c</sup> | 214 (39.3) | 59 (10.8) |
| Decreased appetite | 209 (38.3) | 16 (2.9) |
| Constipation | 205 (37.6) | 8 (1.5) |
| Dysgeusia | 200 (36.7) | 1 (0.2) |
| Abdominal pain | 177 (32.5) | 22 (4.0) |
| Diarrhoea | 176 (32.3) | 11 (2.0) |
| Thrombocytopenia/decreased platelets <sup>c</sup> | 128 (23.5) | 33 (6.1) |
| Blood creatinine increased | 120 (22.0) | 3 (0.6) |
| Dypsnoea | 120 (22.0) | 5 (0.9) |

Treatment-emergent AEs (All Grades and ≥ Grade 3) Reported in

Note: Data are presented by decreasing frequency for TEAEs of all grades, all causality.

**Abbreviations:** ALT = alanine aminotransferase; AST = aspartate aminotransferase; BID = twice a day; MedDRA = Medical Dictionary for Regulatory Activities; N or n = number of patients; TEAE = treatment-emergent adverse event.

- <sup>a</sup> Preferred Terms were based on MedDRA dictionary (version 18.1).
- The data presented in this table are from: all ovarian cancer patients treated with rucaparib 600 mg BID and enrolled in Parts 2A and 2B of Study CO-338-010 and Parts 1 and 2 of Study CO-338-017, with a data cut-off date of 1 September 2018.
- c Combined MedDRA preferred terms

# Safety in the Maintenance Setting (Study CO-338-014 [ARIEL3])

As of the 15 April 2017 cut-off date for Study CO-338-014 (ARIEL3), a total of 561 patients were treated with at least 1 dose of study drug (372 patients in the rucaparib group and 189 patients in the placebo group). The median duration of treatment was 8.3 months (range: 0-35) in the rucaparib group and 5.5 months (range, 0 to 35) in the placebo group.

The TEAEs that occurred in  $\geq$  20% of patients (all grades) in either treatment group are summarized by Preferred Term (PT) in Table 2. The most common TEAEs that occurred in the rucaparib group were nausea (75.3%), asthenia/fatigue (69.4%), dysgeusia (39.2%), and anemia/low or decreased hemoglobin (37.4%). Although greater incidences of these most common TEAEs occurred with rucaparib treatment compared to placebo, the TEAEs reported for the placebo group provide a general context of what events are prevalent in this patient

population without treatment. The most common TEAEs that reported in the placebo group were nausea (36.5%), asthenia/fatigue (43.9%), abdominal pain (25.9%), and constipation (23.8%).

Grade 3 or higher TEAEs are also summarized in Table 2. Approximately half (56.2%) of the patients treated with rucaparib experienced a TEAE of Grade 3 or higher compared to approximately 15% of placebo patients. For patients in the rucaparib group, 2 TEAEs that were Grade 3 or higher had an incidence of > 10%: anemia/low or decreased hemoglobin (18.8%) and increased ALT/AST (10.5%). No Grade 4 events of increased ALT/AST were reported.

Table 2. Treatment-emergent AEs Reported in ≥ 20% of Patients (All Grades) in Any Treatment Group in Study CO-338-014 - Safety Population

| | All G | rades | ≥ Grade 3 <sup>a</sup> | |
|---|---|---|---|---|
| Preferred Term(s) | Rucaparib<br>(N = 372)<br>n (%) | Placebo<br>(N = 189)<br>n (%) | Rucaparib<br>(N = 372)<br>n (%) | Placebo<br>(N = 189)<br>n (%) |
| Number of Patients With at Least One TEAE | 372 (100) | 182 (96.3) | 209 (56.2) | 28 (14.8) |
| Nausea | 280 (75.3) | 69 (36.5) | 14 (3.8) | 1 (0.5) |
| Asthenia/Fatigue | 258 (69.4) | 83 (43.9) | 25 (6.7) | 5 (2.6) |
| Dysgeusia | 146 (39.2) | 13 (6.9) | 0 | 0 |
| Anemia and/or low/decreased hemoglobin | 139 (37.4) | 11 (5.8) | 70 (18.8) | 1 (0.5) |
| Constipation | 136 (36.6) | 45 (23.8) | 7 (1.9) | 2 (1.1) |
| Vomiting | 136 (36.6) | 28 (14.8) | 15 (4.0) | 2 (1.1) |
| ALT/AST Increased | 126 (33.9) | 7 (3.7) | 39 (10.5) | 0 |
| Diarrhea | 118 (31.7) | 41 (21.7) | 2 (0.5) | 2 (1.1) |
| Abdominal pain | 111 (29.8) | 49 (25.9) | 9 (2.4) | 1 (0.5) |
| Thrombocytopenia and/or low/decreased platelets | 104 (28.0) | 5 (2.6) | 19 (5.1) | 0 |
| Decreased appetite | 87 (23.4) | 26 (13.8) | 2 (0.5) | 0 |

**Abbreviations**: ALT = alanine aminotransferase; AST = aspartate aminotransferase; CTCAE = Common Terminology Criteria for Adverse Events; NCI = National Cancer Institute; TEAE = treatment-emergent adverse event.

The laboratory abnormalities were consistent with the TEAEs, with decreased hemoglobin, increased ALT, increased AST, and increased serum creatinine, most common (Table 3). Decreased platelets, neutrophils, leukocytes, lymphocytes, and increased cholesterol were observed to a lesser extent (Table 3).

A decrease in hemoglobin (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] Grade 1 to 4) from baseline was observed in 61% of patients (Grade 3, 13%). A decrease in lymphocytes, platelets, or neutrophils from baseline to a worsening CTCAE Grade occurred in 24%, 40%, and 35% of all patients, respectively). A shift to CTCAE Grade 3 or greater lymphocytes, platelets, or neutrophils was observed in 5%, 2%, and 6%, of all patients, respectively.

Notable shifts from baseline were observed for creatinine, ALT, AST, and cholesterol concentrations in the majority of patients. An increase in ALT or AST from baseline to a

<sup>&</sup>lt;sup>a</sup> NCI CTCAE grade.

worsening CTCAE grade was observed in 73% and 61% of patients, respectively. A shift to CTCAE Grade 3 or greater ALT or AST was observed in 7% and 1% of all patients, respectively.

Increases in ALT/AST are a known self-limiting effect of rucaparib treatment; therefore, management of these elevations was specified within the protocol. Elevations in ALT/AST were generally not accompanied by a concomitant elevation in bilirubin outside the normal range, and no cases met Hy's Law criteria for drug-induced liver injury. Continued dosing with rucaparib in the presence of Grade 3 ALT/AST elevations is permitted if there are no other signs of liver toxicity.

An increase in serum creatinine from baseline to a worsening CTCAE grade occurred in 43% of patients (0.3% Grade 3) using an updated version of the CTCAE (ie, version 5). In CTCAE version 4.03, any increase in creatinine above the baseline value is assessed as a Grade 1 toxicity (1 to 1.5 x baseline value) and almost all patients exhibit a shift from baseline creatinine. In CTCAE version 5, Grade 1 for increased creatinine is based on values greater than the upper limit of normal (ULN). The elevations were observed early in treatment (Day 15 of Cycle 1) and then stabilized with continued rucaparib treatment. Serum creatinine levels decreased with interruption or discontinuation of rucaparib, and increase again with resumption of treatment.

An increase in total cholesterol from baseline to a worsening CTCAE grade occurred in 41% of all patients (4% Grade  $\geq$  3).

Overall, rucaparib safety data at a dose of 600 mg BID in patients with ovarian cancer in Study CO-338-014 in the maintenance setting were consistent with the combined safety data in patients with ovarian cancer from Studies CO-338-010 and CO-338-017 in the treatment setting.

Table 3. Change from Baseline in Laboratory Parameters in Patients Treated with 600 mg BID Rucaparib (Study CO-338-014)

| | | nparib<br>=372) | Placebo<br>(N=189) | |
|---|---|---|---|---|
| Shift in CTCAE Grade (r | 1 [%]) <sup>a</sup> | | • | |
| | Grade 1-4 | Grade 3-4 | Grade 1-4 | Grade 3-4 |
| Decrease in hemoglobin <sup>b</sup> | 224 (61.0) | 46 (12.5) | 24 (12.7) | 2 (1.1) |
| Decrease in lymphocytes <sup>b, c</sup> | 87 (23.7) | 17 (4.6) | 31 (16.5) | 5 (2.7) |
| Decrease in neutrophils <sup>b, c</sup> | 128 (34.9) | 23 (6.3) | 32 (17.0) | 4 (2.1) |
| Decrease in platelets <sup>b</sup> | 145 (39.5) | 8 (2.2) | 15 (8.0) | 0 |
| Shift in CTCAE Grade (r | 1 [%]) <sup>a</sup> | | | |
| | Grade 1-4 | Grade 3-4 | Grade 1-4 | Grade 3-4 |
| Increase in ALT <sup>b</sup> | 267 (72.8) | 24 (6.5) | 7 (3.7) | 0 |
| Increase in AST <sup>c, d</sup> | 223 (60.9) | 3 (0.8) | 7 (3.7) | 0 |
| Increase in alkaline phosphatase <sup>b</sup> | 116 (31.6) | 1 (0.3) | 10 (5.3) | 0 |
| Increase in bilirubin <sup>b</sup> | 34 (9.3) | 1 (0.3) | 3 (1.6) | 0 |
| Increase in cholesterol <sup>b</sup> | 152 (41.4) | 15 (4.1) | 39 (20.6) | 0 |
| Hyperglycemia <sup>b</sup> | 125 (34.1) | 6 (1.6) | 54 (28.6) | 0 |
| Increase in creatinine <sup>b, e</sup> | 156 (42.5) | 1 (0.3) | 14 (7.4) | 0 |

**Abbreviations**: ALT = alanine aminotransferase; AST = aspartate aminotransferase; CTCAE = Common Terminology Criteria for Adverse Events; ULN = upper limit of normal

- Shifts are based on worst grade experienced on treatment and patients who had at least a 1 grade shift from baseline.
- b rucaparib n = 367.
- placebo n = 188.
- d rucaparib n = 366.
- Evaluated using CTCAE, v5 where Grade 1 is > ULN-1.5 ULN; Grade 2 is > 1.5  $\times$  baseline to 3.0  $\times$  baseline or > 1.5  $\times$  ULN to 3.0  $\times$  ULN; Grade 3 is > 3.0  $\times$  baseline or > 3.0  $\times$  ULN to 6.0  $\times$  ULN; and Grade 4 is > 6.0  $\times$  ULN.

#### **Adverse Events of Special Interest**

Myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) are considered adverse events of special interest (AESI), as these events have been observed in patients exposed to cytotoxic chemotherapy (eg, platinum and anthracyclines) used for treatment of ovarian cancer as well as with PARP inhibitors, including rucaparib. Patients in rucaparib clinical studies diagnosed with MDS or AML had significant confounding risk factors including prior cytotoxic chemotherapy, and in some cases a deleterious BRCA mutation, which increases the risk of developing cancer(s). Based on these confounding factors, there is insufficient scientific evidence to conclude that MDS and AML are causally related to rucaparib. More information on AESIs of MDS/AML experienced by patients in rucaparib clinical studies is provided in the rucaparib IB.

Adverse events (AEs) of pneumonitis have been reported with PARP inhibitor treatment, including in clinical trials evaluating rucaparib. Currently, however, there is a lack of understanding of a mechanistic link between pneumonitis and PARP inhibitor treatment, and causality assessment is often confounded by lack of a consistent clinical pattern as well as other pre-disposing factors, such as cancer and/or metastases in lungs, underlying pulmonary disease, smoking history, and/or previous chemotherapy and radiotherapy. Clovis Oncology is seeking to understand whether or not there is a relationship between pneumonitis and rucaparib treatment; thus, Clovis Oncology is designating pneumonitis as an AESI to gather data to enable a thorough evaluation and assessment of the event and associated terms specified in Section 10.7. Also, refer to the rucaparib IB for information regarding the AESI of pneumonitis.

# 3.5 Rationale for this Study of Rucaparib

Homologous recombination deficiency has been observed in many carcinomas, including prostate cancer. Men with a germline mutation in BRCA2 are at increased risk for developing prostate cancer, estimated at 2.5 to 8.6-fold compared with non-carriers. Men with prostate cancer and a germline mutation in BRCA2 typically develop disease at a younger age, have more aggressive features and higher mortality rates; while less common in prostate cancer, germline mutations in BRCA1 are also associated with more aggressive disease. Deleterious germline mutations in other HRR genes, including ATM, checkpoint kinase 2 (CHEK2), RAD51 homolog D (RAD51D) and partner and localizer of BRCA2 (PALB2), have also been reported. In addition to germline mutations, somatic mutations in the HRR genes BRCA1, BRCA2 and ATM, and other much less frequent mutations in BRCA1-interacting protein 1 (BRIP1), CDK12, CHEK2, FANCA, nibrin (NBN), PALB2, RAD51B, and RAD51C have been observed in advanced prostate cancer. Researched

Nonclinical evaluation has demonstrated sensitivity of BRCA1 and BRCA2 homozygous mutant cell lines to rucaparib and other PARP inhibitors (see Section 4.1 of the Investigator's Brochure). In addition, sensitivity to PARP inhibition has also been observed in cells deficient or depleted in other components of HRR, including ATM.<sup>31</sup> This sensitivity is the result of synthetic lethality in homologous recombination deficient cells (like BRCA-mutant tumors) when exposed to a PARPi.

Rucaparib, olaparib, niraparib, and talazoparib, similar agents in the growing class of PARP inhibitors in clinical development, have demonstrated clinical activity in several studies as a single agent for treatment of ovarian, prostate, and breast cancer associated with a BRCA mutation (germline or somatic), as well as in patients without a BRCA mutation.<sup>9, 32-40</sup>

The response to PARP inhibitors in mCRPC patients has been explored in several Phase 1 studies. Fong et al. provided the first description of a BRCA mutant prostate cancer patient responding to PARPi therapy. In a Phase 1 dose-escalation study of olaparib, three mCRPC patients were enrolled, of which one patient was a germline BRCA2 mutation carrier. This BRCA mutant mCRPC patient had a > 50% reduction in his PSA level, resolution of bone metastases, and treatment duration > 1 year. The two mCRPC patients without a germline BRCA mutation did not demonstrate a similar response.

Sandhu et al. reported on a cohort of four patients with germline BRCA2-mutant advanced prostate cancer treated with either olaparib (three patients) or niraparib (one patient).<sup>42</sup> In the patients treated with olaparib, PSA and radiographic responses lasting 34 and 26 months were noted in two patients, and stable disease (SD) of 10 months was noted in the third. The patient treated with niraparib demonstrated primary resistance and quickly progressed; the total duration for niraparib treatment in that patient was 6 weeks.

Olaparib was further evaluated in mCRPC in several Phase 2 studies. In one study that enrolled multiple tumor types, Kaufman et al. (2014) reported efficacy data for eight BRCA mutant mCRPC patients who had received a median number of two prior therapies. All patients had experienced disease progression following hormonal therapy; 75% had received prior docetaxel, and 50% had received prior platinum (carboplatin or cisplatin). Four patients had a confirmed PR (confirmed RECIST Version 1.1 ORR = 50%) and two patients (25%) had a best response of SD. Overall duration of response (DOR) was 327 days, PFS was 7.2 months and median OS was 18.4 months.

More recently, olaparib demonstrated compelling clinical activity in a Phase 2 open-label investigator-sponsored study<sup>9</sup> evaluating mCRPC patients with evidence of HRD. In the Trial of PARP Inhibition in Prostate Cancer (TOPARP) study, which enrolled 50 mCRPC patients who received prior docetaxel (100%), abiraterone or enzalutamide (98%), and cabazitaxel (58%), olaparib demonstrated an ORR of 33% in 49 evaluable patients. Response was defined as any of the following: response according to modified RECIST Version 1.1; at least 50% reduction in PSA level; or a confirmed reduction in the circulating tumor-cell count from 5 or more cells per 7.5 mL of blood to less than 5 cells per 7.5 mL. The ORR in patients with a mutation in a DNA repair gene (n = 16) was 88%, including 7/7 patients with a BRCA2 mutation and 4/5 patients with an ATM mutation. Median radiographic PFS (rPFS) and OS in patients classified as biomarker positive (with HRR gene mutation) were 9.8 months and 13.8 months, respectively, compared to 2.7 months and 7.5 months for patient classified as biomarker negative (no HRR gene mutation).

To date, rucaparib has exhibited clinical activity and an acceptable safety profile when administered as monotherapy. Details of the rucaparib clinical studies and efficacy data are further described in Section 3.4.2 and Section 3.4.2.2, as well an in the IB (Sections 5.1 and 5.3). Complete and partial responses, as defined by RECIST Version 1.1 criteria, as well as durable SD, have been observed in patients with ovarian, breast and pancreatic cancer treated with monotherapy rucaparib. Robust efficacy has been observed in ovarian cancer patients with a BRCA mutation (germline and somatic) (Section 3.4.2.2) and in patients who have a BRCA-like tumor (ie, did not have a BRCA mutation, but had a high percentage of tumor genome loss of heterozygosity [LOH]), including patients with a deleterious mutations in RAD51C or RAD51D. Three mCRPC patients with a BRCA mutation received rucaparib monotherapy in Study CO-338-010 or under named patient access, most of whom experienced tumor stabilization, decrease of PSA levels, and symptom improvement. Rucaparib monotherapy has an established and manageable safety profile. Taken together, nonclinical and clinical data with rucaparib and other PARP inhibitors provide a compelling evidence for use of rucaparib in a selected population of mCRPC patients with predicted loss-of-function mutations in HRR genes such as BRCA1/2 and ATM.

#### 4 STUDY OBJECTIVES

# 4.1 Primary Objective

The primary objective of this study is:

To assess the efficacy of rucaparib versus physician's choice of treatment based on rPFS in mCRPC patients with HRD who progressed on prior AR-directed therapy and have not yet received chemotherapy in the castration-resistant setting.

# 4.2 Secondary Objectives

The secondary objectives of this study are:

- To assess OS
- To assess ORR using modified RECIST Version 1.1 in patients with measurable (nodal or visceral) disease
- To assess DOR using modified RECIST Version 1.1 in patients with measurable (nodal or visceral) disease
- To assess time to PSA progression
- To assess PSA response  $\geq 50\%$  (all patients)
- To assess PSA response  $\geq 90\%$  (all patients)
- To evaluate Patient-reported Outcome (PRO) using the following instruments:
  - EuroQol 5 dimensions 5 level questionnaire (EQ-5D-5L),
  - Functional Assessment of Cancer Therapy—Prostate (FACT-P),
  - Analgesic drug score, and
  - Brief Pain Inventory—Short Form (BPI-SF)
- To assess clinical benefit rate (CBR)
- To assess sparse PK
- To assess safety and tolerability

# 4.3 Exploratory Objectives

Exploratory objectives in this study are:

- To assess concordance in BRCA/ATM gene mutation status in matched Pre-Screening biopsy tissue, archival primary and metastatic tumor tissue, and plasma circulating cell-free tumor DNA (ctDNA)
- To assess changes in the molecular profile over time of matched pre and post-treatment tumor or plasma samples
- To evaluate LOH in metastatic disease site biopsy and archival primary and metastatic tumor tissue samples
- To evaluate mechanisms of response and resistance in ctDNA and progression tumor tissue samples.

## 5 INVESTIGATIONAL PLAN

## 5.1 Overall Study Design and Plan

This is a Phase 3, multicenter, randomized, study of rucaparib versus physician's choice of second-line AR-directed therapy (abiraterone acetate or enzalutamide) or docetaxel as treatment for mCRPC patients with histologically or cytologically confirmed adenocarcinoma who have progressed on one prior AR-directed therapy (abiraterone acetate, enzalutamide, apalutamide, or investigational AR-targeted agent) and have not yet received chemotherapy in the castration-resistant setting. Progression is defined according to the Prostate Cancer Working Group Guidelines Version 3 (PCWG3) criteria as a rise in PSA, new or progressive disease by modified RECIST Version 1.1 (Appendix 1), or two new lesions by radionuclide bone scan. Patients who received prior PARPi treatment will be excluded. This study will enroll mCRPC patients with a deleterious mutation in BRCA1/2 or ATM genes. Deleterious mutations are defined as protein-truncating mutations, large protein-truncating rearrangements, splice site mutations, deleterious missense mutations, and homozygous deletions. Mutations may be detected by local testing, with the result documented in the patient's medical record, or may be detected through central testing provided by the sponsor during Pre-Screening. For local test results, the classification of the mutation as deleterious must be documented in the patient's medical record. The primary endpoint is rPFS using modified RECIST Version 1.1/PCWG3 criteria by central independent radiology review (IRR; rPFSirr).

This study consists of a Pre-Screening Phase (Section 5.1.1), Screening Phase (Section 5.1.2), Randomization (Section 5.1.3), Treatment Phase (Section 5.1.4) and Post-Treatment Phase (Section 5.1.5). Patients will receive rucaparib monotherapy or physician's choice of comparator therapy (pre-designated prior to randomization) in the Treatment Phase, and will undergo procedures and assessments including regular safety and efficacy evaluations during the entire conduct of the study. Patients randomized to the control arm will have the opportunity to receive treatment with rucaparib in the Cross-over Phase of the study, after confirmation of radiographic progression (see Section 5.1.6).

## 5.1.1 Pre-Screening Phase

The Pre-Screening Phase is to identify eligible deleterious BRCA1/2 or ATM gene mutations through central testing of tumor tissue and plasma. Patients who have a qualifying deleterious BRCA1/2 or ATM gene mutation identified through local testing need not enter Pre-Screening and the patient should proceed to the Screening Phase.

To enter Pre-Screening, patients should have evidence of radiographic or biochemical disease progression, and be eligible for this study as their immediate next therapy. Patient tissue and plasma samples should be submitted simultaneously during Pre-Screening. Tissue submitted for Pre-Screening testing should be from a newly obtained metastatic biopsy, if there is a lesion suitable for biopsy and the patient consents to this procedure. If a metastatic biopsy is not feasible, archival tissue samples should be submitted. To reduce the chance of test failure, archival tissue should be < 3 years old. If plasma or tissue samples result in test failure, sites are encouraged to submit additional samples, as available, in order to obtain a successful test result. Patients who have a qualifying deleterious BRCA1/2 or ATM gene mutation identified during

Pre-Screening may proceed to the Screening Phase. A study schema for the Pre-Screening Phase is provided in Figure 1.

In the event that a deleterious BRCA1/2 or ATM gene mutation is identified in plasma or tumor tissue during the Pre-Screening Phase, the patient may be referred by the investigator for genetic counseling and potential germline testing per institutional guidelines. If the patient chooses to have germline testing performed, this result will be entered in the clinical trial database for this study.

During the Pre-Screening Phase, unless otherwise required by local regulations, serious adverse events (SAEs) which are related to protocol-mandated assessments will be reported.

### 5.1.2 Screening Phase

After providing consent to participate, patients with a deleterious BRCA1/2 or ATM gene mutation will undergo Screening assessments within 28 days prior to the first dose of study drug. Patients will undergo procedures and assessments during the Screening Phase as described in Section 9.3.

During the Screening Phase, unless otherwise required by local regulations, SAEs which are related to protocol-mandated assessments will be reported.

Additional screening assessments will include collection of the patient's medical information and demographics, physical exam, laboratory safety assessments, tumor assessments, PRO instruments, and blood and tissue samples to support exploratory objectives as described in Section 9.3.

Randomization will require prospective sponsor (or designee) review and confirmation of eligibility, including, but not limited to:

- BRCA/ATM gene test result by either local or central testing
- details of prior therapy for prostate cancer
- screening laboratory assessments

#### 5.1.3 Randomization

Following confirmation of all eligibility criteria in the Screening Phase, patients will be randomized 2:1 to receive rucaparib or physician's choice of docetaxel or AR-directed therapy (abiraterone acetate or enzalutamide, whichever the patient has not yet received). The physician's choice of agent in the control arm must be prespecified prior to randomization. Randomization will occur by a central randomization procedure using an Interactive Response System (IXRS), which is described in more detail in Section 7.4. Study treatment must be initiated within 3 days after randomization, unless approved by sponsor or designee.

#### 5.1.4 Treatment Phase

During the treatment phase, patients will receive rucaparib or physician's choice (pre-designated prior to randomization) of docetaxel or AR-directed therapy (abiraterone acetate or enzalutamide) and be monitored for safety and efficacy as described in Section 9.5.

Rucaparib will be administered as 600 mg orally BID. Abiraterone acetate will be administered as 1,000 mg orally QD, with prednisone administered concomitantly at a dose of 10 mg orally daily. Enzalutamide will be administered as 160 mg orally QD. Docetaxel will be administered at a dose of 75 mg/m<sup>2</sup> IV every 3 weeks in combination with prednisone or prednisolone, given orally, 5 mg BID, for up to a maximum of 10 cycles.

Patients will receive the same therapy, as appropriate, throughout the Treatment Phase, or in the case of docetaxel up to a maximum of 10 cycles whereupon no additional study treatment shall be given, but all assessments will continue to be performed until criteria for treatment discontinuation are met. PRO assessments should also be collected at every visit.

Tumor assessments by computed tomography (CT)/magnetic resonance imaging (MRI) and bone scans will be performed during the Screening Phase, at the end of every 8 calendar weeks ( $\pm 7$  days) from Study Day 1 (Week 1) up to 24 weeks and every 12 calendar weeks ( $\pm 7$  days) thereafter, and at the Treatment Discontinuation Visit, if applicable. Modified RECIST Version 1.1 criteria will be used to document radiographic response in soft tissue (visceral and nodal) disease and PCWG3 criteria will be used to document radiographic progression in bone lesions. If a CR or PR is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented. Radiographic tumor assessment (using the same methodology as was used at initial study screening [eg, CT scan and bone scan]) will continue until radiographic disease progression is confirmed, irrespective of whether the patient has discontinued study drug treatment or initiated subsequent anticancer therapy. Any drug modifications (interruption, dose reduction, or discontinuation) should be documented in the electronic case report form (eCRF) and source documents. If study treatment is interrupted, tumor assessments will not be delayed and will proceed on the regular study schedule. Copies of all radiographic scans will be submitted for IRR until after the analysis of the primary endpoint has been performed, at which time IRR will be discontinued and all radiographic scans will be evaluated by the investigator for radiographic progression. The sponsor will inform investigators when submission of scans for IRR should discontinue.

Patients will receive study drug until radiographic disease progression is confirmed by IRR until analysis of the primary endpoint has been performed, or by investigator assessment after analysis of the primary endpoint has been performed and IRR is discontinued, based on modified RECIST Version 1.1 and PCWG3 (for bone lesions only) criteria, unequivocal clinical disease progression, unacceptable toxicity or inability to tolerate further treatment, loss to follow-up, or withdrawal of consent. Patients in the docetaxel arm will receive study drug for a maximum of 10 cycles only and so may not be actively on treatment at the time of disease progression. PSA rise without evidence of confirmed radiographic progression is strongly discouraged as a criterion to start a new systemic antineoplastic therapy during the first 12 weeks of therapy and is discouraged as a criterion to start a new systemic antineoplastic therapy throughout the study. Palliative radiation for the treatment of painful bony metastases and initiation of bisphosphonates

or other approved bone-targeting agents are allowed and should not result in discontinuation of study drug therapy.

Patient safety will be monitored on a regular basis using procedures and assessments described in Section 9 and Section 13.4. Safety and efficacy data will be periodically reviewed by the Independent Data Monitoring Committee (IDMC) as described in Section 13.6.

#### 5.1.5 Post-treatment Phase

The date and reason for cessation of study drug must be documented in the eCRF and source documents as soon as possible. Patients will undergo procedures and assessments during the Post-treatment Phase as described in Section 9.6. Upon treatment discontinuation, patients will have a Treatment Discontinuation Visit (Section 9.6.1), a 28-day Follow-up Visit (Section 9.6.2), and then will proceed to long-term follow-up (Section 9.6.3). An optional tumor biopsy will be collected prior to the start of subsequent anticancer therapy from patients who experience radiographic or unequivocal clinical disease progression and who provide appropriate consent. For patients who had their last tumor assessment  $\geq 8$  weeks ( $\geq 12$  weeks if previous scan was after 24 weeks on study) prior to the Treatment Discontinuation Visit, a tumor assessment must be performed.

If study drug was discontinued for reasons other than centrally confirmed radiographic disease progression, tumor assessments (using the same methodology as was used at initial study screening [eg, CT scan]) will continue until radiographic disease progression is confirmed by IRR. Similarly, PRO will continue to be collected during this time and until radiographic disease progression is confirmed by IRR. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator, as well as collection of PRO, as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR.

Ongoing SAEs, AESIs, and treatment-related Grade 3/4 AEs will be followed until either resolution or stabilization has been determined or until lost to follow-up.

After the 28-day Follow-up Visit, only SAEs assessed as potentially related to study drug should be reported per Clovis Oncology Pharmacovigilance (PV) requirements and captured in the Clovis Oncology PV database.

After the 28-day Follow-up Visit, **AESIs of MDS and AML**, **irrespective of causality, should be reported** per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

• AESIs of pneumonitis or similar events (ie, interstitial lung disease, pulmonary fibrosis, acute interstitial pneumonitis, alveolitis necrotizing, alveolitis, hypersensitivity pneumonitis, and organizing pneumonia) should be reported up to, but not beyond, the 28-Day Follow-up Visit (28-days after the last dose of rucaparib). After the 28-day Follow-up Visit, only pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements.

All patients will be followed for survival and subsequent treatments every 12 weeks ( $\pm$  14 days) relative to the last dose of study drug until death, loss to follow-up, withdrawal of consent, or study closure.

#### 5.1.6 Cross-over Phase

Patients randomized to comparator therapy will be given the opportunity to cross over to receive rucaparib therapy after radiographic progression is confirmed by IRR until analysis of the primary endpoint has been performed, or by investigator assessment after analysis of the primary endpoint has been performed and IRR is discontinued. After providing consent, patients will be assessed to ensure eligibility criteria are met for the Cross-over Phase (see protocol Section 6.4). If eligible, the patient will have protocol assessments for a Treatment Discontinuation Visit performed when treatment to which the patient is randomized has been completed or is discontinued and then will have protocol assessments per the rucaparib Treatment Phase. Radiographic assessments from the Cross-over Phase will not be submitted for IRR either before or after the analysis of the primary endpoint has been performed. The patient will also have all Post-Treatment Phase assessments completed after discontinuing cross-over rucaparib, including a second Treatment Discontinuation Visit.

### 5.1.7 Post-progression Treatment Phase

If a patient demonstrates radiographic progression while receiving treatment with study drug, but continues to derive clinical benefit per investigator assessment, then continuation of treatment beyond progression is permitted. In such cases, the patient must consent prior to continuing treatment with study drug.

# 5.2 Study Schema

The Pre-Screening Phase study schema is provided in Figure 1.

The study schema for Screening, Treatment, and Post-treatment Phases is provided in Figure 2.

Figure 1. Pre-Screening Study Schema



- \* Patients should be demonstrating radiographic or biochemical progression in order to enter the Pre-Screening and Screening Phases
- \*\* Metastatic biopsy (preferred) or archival tissue; tissue samples should be < 3 years old

Figure 2. Study Schema: Screening, Treatment, and Post-treatment Phases



# 5.3 End of Study

The study will close when the required number of rPFS events has been observed and sufficient follow-up for OS events has occurred. At the time the decision is made to close the study, individual patients who are continuing to benefit from treatment with rucaparib and who do not meet any of the criteria for withdrawal, will have the option of receiving rucaparib via another access mechanism. If a patient is continuing to receive benefit from physician's choice standard-of-care at the time of a decision to close the study, the study site treating the patient may remain open until discontinuing the treatment or the patient qualifies for cross-over to rucaparib. The option of receiving rucaparib via another access mechanism will be available if the patient is tolerating their rucaparib regimen and meets the requirements for entering the alternative access mechanism. In addition, if there are patients for whom long-term follow-up information is being collected, these patients may transition to have their long-term follow-up information captured via another mechanism.

The sponsor may discontinue the study early for any reason as noted in Section 13.7.

#### **6 STUDY POPULATION SELECTION**

#### 6.1 Number of Patients and Sites

The total enrollment planned for this study is approximately 400 patients. A total of approximately 300 patients with a deleterious BRCA1/2 gene mutation will be randomized and approximately 100 patients with a deleterious ATM gene mutation may be randomized. These patients will be recruited from approximately 150 sites worldwide. Patients will be randomized 2:1 to receive rucaparib or physician's choice of either docetaxel or second-line AR-directed therapy (abiraterone acetate or enzalutamide, whichever the patient has not yet received).

#### 6.2 Inclusion Criteria

Eligible patients must meet the following inclusion criteria. Unless otherwise specified, the criteria below apply to all patients:

- 1. Have signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form (ICF) prior to any study-specific evaluation
- 2. Male  $\geq$  18 years of age at the time the ICF is signed
- 3. Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma of the prostate (pure small-cell histologies or pure high-grade neuroendocrine histologies are excluded; neuroendocrine differentiation is allowed) that is metastatic
- 4. Surgically or medically castrated, with serum testosterone levels of ≤ 50 ng/dL (1.73 nM). If currently being treated with luteinizing hormone–releasing hormone (LHRH) analogs (patients who have not undergone an orchiectomy), therapy must be continued throughout the study
- 5. Eligible for treatment with physician's choice of comparator treatment, selected prior to randomization, per the corresponding prescribing information
- 6. Evidence of disease progression after treatment with one prior next-generation AR-targeted therapy (abiraterone acetate, enzalutamide, apalutamide, or investigational AR-targeted

- agent); treatment with the older anti-androgen therapies such as bicalutamide, flutamide, and nilutamide are not counted toward this limit
- 7. Disease progression after initiation of most recent therapy is based on <u>any</u> of the following criteria:
  - a. Rise in PSA: a minimum of two consecutive rising levels, with an interval of ≥ 1 week between each determination. The most recent screening measurement must have been ≥ 2 ng/mL
  - b. Transaxial imaging: new or progressive soft tissue masses on CT or MRI scans as defined by modified RECIST Version 1.1
  - c. Radionuclide bone scan: at least two new metastatic lesions
- 8. All patients must have a deleterious gene mutation in BRCA1/2 or ATM. Mutations may be identified by local testing or through central testing by the sponsor of plasma or tumor tissue. For local test results, the classification of the mutation as deleterious must be documented in the patient's medical record
- 9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Appendix 2)
- 10. Have adequate organ function confirmed by the following clinical laboratory values obtained within 14 days prior to the first dose of study drug:
  - a. Bone Marrow Function
    - i. ANC  $> 1.5 \times 10^9/L$
    - ii. Platelets  $> 100 \times 10^9/L$
    - iii. Hemoglobin ≥ 10 g/dL independent of transfusion within 14 days
  - b. Hepatic Function
    - i. AST and ALT  $\leq 3 \times$  the ULN
    - ii. Bilirubin  $\leq 1.5 \times \text{ULN}$  ( $\leq 2 \times \text{ULN}$  if hyperbilirubinemia is due to Gilbert's syndrome)
  - c. Renal Function
    - i. Estimated glomerular filtration rate (GFR) ≥ 45 mL/min using the Cockcroft-Gault formula (Appendix 3)
- 11. Male patients who are committed to undertaking the following measures for the duration of the study and after the last dose of study drug for the time period specified:
  - a. Use a condom during sex while being treated and for 3 months after the last dose of study drug.
  - b. Do not make semen donations during treatment and for 3 months after the last dose of rucaparib,
  - c. Those with female partners of childbearing potential may be enrolled if they are:
    - i. Documented to be surgically sterile (ie, vasectomy);
    - ii. Committed to practicing true abstinence during treatment and for 3 months after the last dose of study drug; or
    - iii. Committed to using a highly effective method of contraception (refer to Section 6.5) with their partner during treatment and for 3 months following the last dose of study drug
- 12. Have a life expectancy of at least 6 months

#### 6.3 Exclusion Criteria

Patients who meet any of the following criteria will be excluded from the study:

- 1. Active second malignancy, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
  - a. Patients with a history of malignancy that has been completely treated, and currently with no evidence of that cancer, are permitted to enroll in the study provided all therapy was completed > 6 months prior and/or bone marrow transplant (BMT) > 2 years prior to first dose of rucaparib
- 2. Prior treatment with any PARPi
- 3. Prior treatment with chemotherapy (eg docetaxel, mitoxantrone, cyclophosphamide, platinum-based agents) for mCRPC. Prior treatment with docetaxel (or other taxane chemotherapy) administered for castration-sensitive disease is permitted
- 4. Symptomatic and/or untreated central nervous system (CNS) metastases. Patients with asymptomatic, previously treated CNS metastases are eligible provided they have been clinically stable (not requiring steroids for at least 4 weeks prior to first dose of study drug) and have appropriate scans at screening assessment
- 5. Symptomatic or impending spinal cord compression unless appropriately treated, clinically stable, and asymptomatic
- 6. Pre-existing duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of study drug
- 7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or history of chronic hepatitis B or C, with the exception of patients with sustained virologic response after completion of treatment for hepatitis C
- 8. Received treatment with chemotherapy, antibody therapy, immunotherapy, gene therapy, angiogenesis inhibitors, or experimental drugs within < 14 days prior to first dose of study drug. Treatment with hormonal therapies (with the exception of LHRH analog) must be discontinued at least 7 days prior to the first dose of study drug
- 9. Adverse effect of prior therapy not resolved to CTCAE Grade 1 or below with the exception of alopecia. Ongoing Grade 2 non-hematologic toxicity related to most recent treatment regimen may be permitted with prior advanced approval from the sponsor
- 10. Initiated low-dose corticosteroid, bisphosphonate, or denosumab therapy or adjusted low-dose corticosteroid, bisphosphonate, or denosumab dose/regimen within < 28 days prior to first dose of study drug. Patients on a stable low-dose corticosteroid, bisphosphonate, or denosumab regimen are eligible and may continue treatment
- 11. Non-study related minor surgical procedure within < 5 days, or major surgical procedure within < 21 days, prior to first dose of study drug; in all cases, the patient must be sufficiently recovered and stable before treatment administration
- 12. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry into the study

# 6.4 Criteria for Rucaparib Cross-over Treatment Eligibility Following Radiographic Progression on or after Comparator Arm Therapy

To be eligible for participation in the cross-over part of the study, patients must fulfill the following criteria and should initiate treatment with rucaparib  $\leq$  28 days after the date of the radiographic disease assessment by which progression is confirmed by IRR until analysis of the primary endpoint has been performed. Treatment with rucaparib may be permitted > 28 days after the date of the radiographic disease assessment by which progression is confirmed by IRR with prior advanced approval from the sponsor, and all cross-over eligibility criteria are met (Note: Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR. After analysis of the primary endpoint, investigator-assessed radiographic disease progression will be used for cross-over eligibility evaluation):

- 1. Receive sponsor approval to cross-over from comparator therapy to rucaparib treatment
- 2. Received the last dose of comparator therapy at least 14 days prior to initiation of rucaparib treatment (7 days prior for abiraterone acetate or enzalutamide)
- 3. Have adequate organ function confirmed by the following local laboratory values  $\leq$  14 days prior to first dose of rucaparib:
  - a. Bone Marrow Function
    - i. ANC  $\geq 1.5 \times 10^9/L$
    - ii. Platelets  $> 100 \times 10^9/L$
    - iii. Hemoglobin  $\geq 9$  g/dL independent of transfusion within 14 days
  - b. Hepatic Function
    - i. AST and ALT  $\leq 3 \times ULN$
    - ii. Bilirubin  $\leq 1.5 \times \text{ULN}$  ( $< 2 \times \text{ULN}$  if hyperbilirubinemia is due to Gilbert's syndrome)
  - c. Renal Function
    - i. Estimated GFR  $\geq$  45 mL/min using the Cockcroft-Gault formula (Appendix 3)
- 4. All Grade 3 and 4 hematologic and non-hematologic toxicities (except alopecia, nausea, vomiting, or adequately controlled diarrhea) resolved to baseline or ≤ CTCAE Grade 1
- 5. Male patients who are committed to undertaking the following measures for the duration of the study and after the last dose of rucaparib for the time period specified:
  - a. Use a condom during sex while being treated and for 3 months after the last dose of rucaparib,
  - b. Do not make semen donations during treatment and for 3 months after the last dose of rucaparib,
  - c. Those with female partners of childbearing potential may cross-over if they are:
    - i Documented to be surgically sterile (ie, vasectomy);
    - ii Committed to practicing true abstinence during treatment and for 3 months after the last rucaparib dose; or
    - iii Committed to using a highly effective method of contraception (refer to Section 6.5) with their partner during treatment and for 3 months following the last dose of rucaparib

- 6. Have an ECOG performance status of 0 to 1 (Appendix 2).
- 7. Written consent on an Institutional Review Board (IRB)/ Independent Ethics Committee (IEC)-approved ICF

In addition, any of the following will exclude patients from receiving rucaparib in the cross-over part of the study:

- 1. Adverse effect of comparator therapy not resolved to CTCAE Grade 1 or below with the exception of alopecia. Ongoing Grade 2 non-hematologic toxicity related to comparator therapy may be permitted with prior approval from the sponsor
- 2. Received treatment with chemotherapy, hormonal therapy (with the exception of LHRH analog), radiation (other than palliative radiation for treatment of painful bony metastases), antibody therapy, immunotherapy, gene therapy, angiogenesis inhibitors, or experimental drugs after discontinuation of study comparator therapy. Patients requiring urgent intervening systemic anticancer therapy, may be permitted to cross over, provided that criteria for unequivocal clinical progression are confirmed per Section 12.1, in consultation with the sponsor, prior to initiation of intervening systemic anticancer therapy
- 3. Non-study-related minor surgical procedure within < 5 days, or major surgical procedure within < 21 days, prior to first dose of rucaparib in cross-over; in all cases, the patient must be sufficiently recovered and stable before treatment administration
- 4. Withdrawal of consent during treatment with the comparator arm therapy
- 5. Presence of any other condition that may increase the risk associated with study participation and, in the opinion of the investigator, would make the patient inappropriate for continuing in the study with cross-over to rucaparib treatment (including general noncompliance with study procedures during treatment with the comparator arm therapy, per investigator judgement)

# 6.5 Patients or Partners of Patients Including Those of Reproductive Potential

Male patients are required to use a condom during sex with a partner to avoid the possibility of exposure of the partner to rucaparib.

Male patients must not make semen donations for 3 months after the last dose of rucaparib.

Male patients of reproductive potential must avoid pregnancy in partners who are women of childbearing potential, and such partners should not be considering getting pregnant during the study and for at least 3 months after treatment is discontinued or longer if requested by local authorities. Patients will be instructed to notify the investigator if pregnancy of female partner is discovered either during or within 3 months of completing treatment with study drug.

Male patients are considered to be of reproductive potential unless permanently sterile by bilateral orchiectomy, or with appropriate post-vasectomy documentation of absence of sperm in ejaculate.

Female partners are considered to be of childbearing potential unless one of the following applies:

- Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 mIU/mL or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state: or
- Considered to be permanently sterile. Permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy.

Male patients of reproductive potential must practice highly effective methods (failure rate < 1% per year when used consistently and correctly) of contraception with their female partners, if of reproductive potential, during treatment and for 3 months following the last dose of study drug or longer if requested by local authorities. Highly effective contraception includes:

- Ongoing use of combined (estrogen- and progestogen-containing) hormonal contraception oral, injectable, or transdermal, associated with inhibition of ovulation;
- Ongoing use of progesterone-only oral, injectable, or implantable contraceptives associated with inhibition of ovulation;
- Placement of an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS);
- Bilateral tubal occlusion;
- Sexual abstinence as defined as complete or true abstinence, acceptable only when it is the usual and preferred lifestyle of the patient; periodic abstinence (eg, calendar, symptothermal, post-ovulation methods) is not acceptable.

#### 6.5.1 Patients Not on Rucaparib

Patients must practice the contraception requirements listed above and additionally apply appropriate requirements for treatment with physicians' choice of comparator according to product labelling and local practice.

#### 6.6 Waivers of Inclusion/Exclusion Criteria

No waivers of these inclusion or exclusion criteria will be granted by the investigator and the sponsor or its designee for any patient enrolling into the study.

# 7 STUDY TREATMENT(S)

# 7.1 Description of Treatment(s) and Storage

This study will assess the investigational drug rucaparib compared to comparator therapy using a randomized 2:1 study design.

# 7.1.1 Investigational Drug Product - Rucaparib

Rucaparib camsylate (also known as CO-338) is an oral formulation with a molecular weight of 555.67 Daltons. Rucaparib tablets for oral administration will be supplied to the study sites by the sponsor. The starting dose of rucaparib is 600 mg ingested BID. A brief description of the investigational product is provided below with details in the Pharmacy Guidelines.

| Drug Name: | Rucaparib |
|---|---|
| INN: | Rucaparib |
| Formulation: (strengths expressed as free base) | Tablet; film coated; 200 mg (blue, round, debossed with C2), 250 mg (white, rounded diamond shape, debossed with C25), 300 mg (yellow, oval, debossed with C3) |
| How Supplied: | 200, 250, and 300 mg (as free base) strength tablets in HDPE or equivalent with child-resistant caps. Patients may receive one or more strengths. |
| Storage Conditions: | 15 to 30° C (59 to 86° F). |

Abbreviation: HDPE = high density polyethylene; INN = International Nonproprietary Name.

### 7.1.2 Comparator Therapeutic Drug Products

Single-agent chemotherapy will consist of docetaxel given at a dose of 75 mg/m<sup>2</sup> docetaxel IV every 3 weeks given in combination with oral prednisone or prednisolone 5 mg BID, for up to a maximum of 10 cycles.

The starting dose of abiraterone is 1,000 mg orally QD. No food should be eaten for at least 2 hours before and for one hour after dosing. Prednisone should be administered concomitantly at a dose of 10 mg orally daily. Abiraterone should be swallowed whole with water.

The starting dose of enzalutamide is 160 mg orally QD. Enzalutamide may be taken with or without food. Enzalutamide should be swallowed whole with water.

Each of these individual drugs will either be procured by the study site or supplied by the sponsor. Each product will be stored according to the manufacturer's prescribing information/product packaging and as described in the Pharmacy Guidelines.

Please refer to the pharmacy manual for further details.

# 7.2 Packaging and Labeling

# 7.2.1 Rucaparib

Rucaparib tablets are provided in 60-count high-density polyethylene (HDPE) bottles with child-resistant caps and should be stored in the provided containers between 15° to 30°C (59 to 86°F). Patients will be dispensed one or more strengths depending on their current dose of rucaparib. The number of bottles of each strength dispensed will be sufficient to supply at least 28 days of treatment until the next study drug dispensing visit.

Rucaparib bottles will be labelled in accordance with local regulatory requirements.

## 7.2.2 Comparator Therapy

Depending on local health authority guidelines, the comparator therapy agents will be obtained through commercial supply, the site pharmacy, or from the sponsor, depending on region. The packaging and labeling will vary depending on the source of the supply.

Products will be labeled to meet local country requirements. Where sites source their own comparator therapies, they are responsible for the quality and security of the supply and for ensuring it is appropriately labeled and dispensed in compliance with local regulations.

# 7.3 Blinding

This is an open-label study; the study drugs will not be blinded or masked to the investigator or patient, so each will know the treatment being administered. A Blinding Plan will be put in place to limit the knowledge of aggregate efficacy data by sponsor personnel.

# 7.4 Method of Assigning Patients to Treatment Groups

Patients will be randomly assigned to treatment groups via IXRS. The following will be included as randomization stratification factors at study entry to ensure treatment groups are balanced; ECOG performance status and presence of hepatic metastases are important prognostic indicators in this patient population.<sup>44, 45</sup>

- ECOG Status 0 vs 1
- Presence of hepatic metastases or not
- BRCA1 vs BRCA2 vs ATM mutation

The investigator should have experience using the comparator therapy that is selected.

Study treatment must be initiated within 3 days after randomization unless otherwise agreed between investigator and sponsor (or designee).

# 7.5 Preparation and Administration of Protocol-specified Treatment

The investigator will be responsible for distributing study drug to all patients. Study drug (ie, rucaparib or comparator therapy) will be assigned by the IXRS according to the patient's randomization assignment.

The IXRS will manage all study drug supplied by the sponsor. The system should be accessed to record each dispensation of rucaparib and each administration of the comparator therapies according to the patient's randomized treatment. Guidelines for the use of the IXRS will be provided to study sites. Study sites should follow local guidelines for the handling of comparator therapy.

## 7.5.1 Rucaparib

The starting dose of rucaparib is 600 mg ingested BID. Patients may take rucaparib with or without food. Each dose should be taken with at least 8 oz (240 mL) of water. Tablets should be swallowed whole without crushing or chewing. Tablet strength combinations shall be determined by the IXRS system.

Patients should take rucaparib doses as close to 12 hours apart as possible, preferably at the same times every day. If a patient misses a dose (ie, does not take it within 4 hours of the scheduled time), the patient should skip the missed dose and resume taking rucaparib with the next scheduled dose. Missed or vomited doses should not be made up.

Dosing with rucaparib may be held or reduced as described in Section 7.5.1.1 and Section 7.5.1.2.

Patients will be provided a sufficient quantity of study drug for 28 days with a small overage. Patients will be instructed to bring their rucaparib tablets and all containers (empty, partially used, and/or unopened) to the next scheduled visit for reconciliation by site personnel. Partially used bottles may be returned to the patient according to local guidelines.

#### 7.5.1.1 Rucaparib Dose Modification Criteria

Treatment with rucaparib should be held if any of the following are observed and a dose reduction should be considered or implemented.

- Grade 3 or 4 hematologic toxicity
- Grade 3 or 4 non-hematologic toxicity (except for alopecia, nausea, vomiting, or diarrhea
  adequately controlled with systemic antiemetic/antidiarrheal medication administered in
  standard doses according to the study center routines). Grade 3 or Grade 4 ALT/AST
  elevations should be managed as described below.
- At the discretion of the investigator, rucaparib may be held or continued if new or worsening unexplained pulmonary symptoms suggestive of pneumonitis (including, but not limited to, dyspnea) occur and while evaluation to rule out pneumonitis or confirm such a diagnosis as well as etiology are ongoing; these events should be managed as described below.
- In addition, and at the discretion of the investigator, the dose of rucaparib may be held and/or reduced for Grade 2 toxicity not adequately controlled by concomitant medications and/or supportive care.

# MANAGEMENT OF ANEMIA INCLUDING EVALUATION FOR MDS/AML AND FOLLOW-UP OF PATIENTS WHO DISCONTINUE TREATMENT WITH ONGOING ANEMIA

- If the patient develops anemia CTCAE Grade ≥ 3, rucaparib treatment should be held until the anemia resolves to CTCAE Grade ≤ 2 whereupon daily dosing may then be resumed at either the same dose or a lower dose, per investigator discretion.
- If a patient has persistent CTCAE Grade 3 anemia despite study drug interruption, and the anemia is considered related to the patient's underlying prostate cancer (eg, patient has

- extensive bony disease or history of disease-related anemia), then resumption of study drug may be considered, if the patient was benefiting from treatment in the opinion of the investigator
- If the duration of dosing is interrupted for > 14 consecutive days due to anemia CTCAE Grade ≥ 3, treatment should be permanently discontinued, unless otherwise agreed between the investigator and the sponsor.
- In addition, if anemia CTCAE Grade ≥ 3 persists for > 14 consecutive days, or a dependence upon blood transfusion occurs, then weekly complete blood counts should be performed until resolution of the event.
- If, after 42 days of interruption of rucaparib, the anemia has not recovered to CTCAE Grade ≤ 1 then the patient should be referred to a hematologist and analysis of the bone marrow with cytogenetic studies are recommended according to standard hematologic practice.
  - The bone marrow analysis should include a bone marrow aspirate (for cellular morphology, cytogenetic analysis, and flow cytometry) and a core biopsy (for bone marrow cellularity).

#### MANAGEMENT OF RUCAPARIB TREATMENT-EMERGENT ALT/AST ELEVATIONS

- Grade 4 ALT/AST elevations: hold rucaparib until values have returned to Grade 2 or better, then resume rucaparib with a dose reduction. Monitor liver function tests weekly for 3 weeks after rucaparib has been restarted.
- Grade 3 ALT/AST elevations, in the absence of other signs of liver dysfunction, should be managed as follows:
  - Monitor liver function tests weekly until resolution to  $\leq$  Grade 2.
  - Continuation of rucaparib with elevation of ALT/AST up to Grade 3 is permitted provided bilirubin is < ULN.
  - If patient has Grade 3 ALT/AST and continues on rucaparib, and levels do not decline within 2 weeks or they continue to rise, treatment interruption and resolution to ≤ Grade 2 will be required before rucaparib can be resumed, either at the current dose or at a reduced dose.

For patients who meet treatment interruption guidelines above, treatment with rucaparib should be held until the toxicity resolves to  $\leq$  CTCAE Grade 2. Dosing BID may then be resumed at either the same dose or a lower dose, per investigator discretion. If treatment is resumed at the same dose, and the patient experiences the same toxicity, treatment should be interrupted, then resumed at a reduced dose following resolution of the event to  $\leq$  CTCAE Grade 2. If the patient continues to experience toxicity, additional dose reduction steps are permitted; however, the investigator must consult with the sponsor's medical monitor before reducing to 300 mg BID. If a patient continues to experience toxicity despite dose reduction steps to 300 mg BID, or if dosing with rucaparib is interrupted for > 14 consecutive days due to toxicity, treatment should be discontinued, unless otherwise agreed between the investigator and the sponsor.

Drug-induced liver injury (DILI) is described in the US FDA Guidance for Industry, Drug-Induced Liver Injury: Premarketing Clinical Evaluation, <sup>46</sup> and should be referenced when managing treatment-emergent ALT/AST elevations.

Rucaparib treatment must be interrupted if biochemical criteria for suspected DILI are met, according to presence of the following laboratory abnormalities:

ALT or AST 
$$> 3 \times ULN$$
  
and  
Bilirubin  $> 2 \times ULN$ 

While treatment is interrupted, the patient should be evaluated for the presence of confounding factors including malignant disease in the liver, coadministration of other suspect drugs, cholestasis, and viral or autoimmune hepatitis that could have caused the laboratory abnormalities. Other laboratory investigations of liver function such as international normalized ratio (INR) should be implemented as indicated. If no alternative cause is identified, rucaparib must be permanently discontinued.

All cases of possible DILI must be reported as SAEs (see Section 10.9) and will be followed until all abnormalities have returned to normal or to baseline levels, or an alternative cause is found to explain the combination of the increased transaminases and bilirubin.

#### MANAGEMENT OF NEW OR WORSENING PULMONARY SYMPTOMS

If new or worsening unexplained pulmonary symptoms suggestive of pneumonitis (including, but not limited to, dyspnea) occur, or a deterioration of pulmonary function is observed, and/or radiologic abnormality is detected in the lungs, and this occurs in the absence of any clear diagnosis, a diagnostic workup (including high resolution CT scan) in consultation with a pulmonologist should be performed in order to rule out pneumonitis. During this time, treatment with rucaparib may be interrupted or continued per investigator discretion.

Following investigation, if pneumonitis is <u>not</u> confirmed, treatment with rucaparib may be resumed/continued as deemed appropriate by the investigator and in accordance with the study protocol directions for management of AEs. All confirmed events of pneumonitis should be treated as appropriate per medical judgement and institutional guidelines. If the event resolves and retreatment with rucaparib is being considered, please consult the Sponsor's Medical Monitor. Retreatment with rucaparib may be resumed at the current or a reduced dose, if appropriate.

Refer to Sections 10.3 and 10.7 of the protocol for additional information regarding classification and reporting of pneumonitis (and associated events) as an AESI.

#### 7.5.1.2 Rucaparib Dose Modification

Dose reduction steps are presented in Table 4.

Dose re-escalation upon resolution of toxicity to  $\leq$  CTCAE Grade 1 is permitted at the discretion of the investigator.

Dose modifications (interruption, reduction, re-escalation) must be recorded for each patient in the appropriate section of the eCRF.

Table 4. Rucaparib Dose Reduction Steps

| Starting Dose | 600 mg BID |
|-----------------------------|------------|
| Dose Level - 1 | 500 mg BID |
| Dose Level - 2 | 400 mg BID |
| Dose Level - 3 <sup>a</sup> | 300 mg BID |

Abbreviation: BID = twice a day.

#### 7.5.1.3 General Restrictions

Photosensitivity has been observed in patients treated with rucaparib. Patients should avoid spending time in direct sunlight because they burn more easily during treatment with rucaparib. When outdoors, patients should use typical precautions such as applying sunscreen (sun protection factor 50 or greater) and/or covering exposed skin with clothing and wearing a hat and sunglasses.

## 7.5.2 Single-agent Docetaxel

Handling, preparation, administration, precautions, and restrictions for the use of docetaxel are to follow Prescribing Information provided in the Pharmacy Guidelines or approved institutional or local guidelines.

# 7.5.3 Single-agent Abiraterone Acetate

Handling, preparation, administration, precautions, restrictions and other information for the use of each drug are in the Prescribing Information provided in the Pharmacy Guidelines or approved institutional or local guidelines.

#### 7.5.4 Single-agent Enzalutamide

Handling, preparation, administration, precautions, restrictions and other information for the use of each drug are in the Prescribing Information provided in the Pharmacy Guidelines or approved institutional or local guidelines.

# 7.5.5 Re-treatment and Dose Modification for All Comparator Therapy

In the event of toxicities, dose delays and modifications should occur in accordance with the highest toxicity observed per the recommendations and guidelines provided in the approved Prescribing Information provided in the Pharmacy Guidelines or according to institutional guidelines or local dose reduction protocols. Dose modifications (interruption, reduction, re-escalation) must be recorded for each patient in the appropriate section of the eCRF.

<sup>&</sup>lt;sup>a</sup> Consult with the sponsor's medical monitor before reducing to dose level 3. Further dose reduction may be possible, but requires consultation with the sponsor's medical monitor.

### 7.5.6 Cross-over to Rucaparib Treatment

Patients initially randomized to comparator therapy have the option to cross-over to rucaparib treatment upon radiographic disease progression, following sponsor (or designee) approval of the radiology report confirming disease progression by IRR, and meeting eligibility for the cross-over as listed in Section 6.4.

Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR. After analysis of the primary endpoint, investigator-assessed radiographic disease progression will be used for cross-over eligibility evaluation. Patients may cross-over to rucaparib treatment upon radiographic disease progression, following sponsor (or designee) approval of the radiology report confirming disease progression by the investigator, and provided the patient meets eligibility criteria for cross-over as listed in Section 6.4.

Patients who cross-over to receive rucaparib will continue to have all protocol-required assessments as described in Section 9. Cross-over to rucaparib can occur only after toxicities related to the comparator have resolved or sufficiently stabilized and the patient meets all criteria for initiation of treatment with rucaparib. Initiation of treatment with rucaparib should normally occur within 28-days following the scan date resulting in confirmed radiographic disease progression. Deviations from this timeline must be confirmed with the Sponsor.

## 7.5.7 Continuation of Study Drug beyond Disease Progression

If a patient (either per initial randomization or after cross-over) has met the criteria for radiographic disease progression, but continues to derive clinical benefit per investigator assessment, then continuation of treatment is permitted with additional consent. Clinical scenarios where continuation of study drug treatment after radiographic progression may be considered include a patient in whom radiographic progression develops slowly while disease-related symptoms remain well controlled, a patient who experiences progression in a site of disease that is unlikely to adversely affect prognosis (eg, enlargement of a solitary lymph node), or a patient with general disease control but limited progression in sites of disease that can be managed with local therapies such as surgery or radiation. In such cases, the decision to continue must be documented in the medical notes prior to continuing treatment. Patients continuing to receive study drug will need to provide additional consent and will continue to have all protocol-required assessments as described in Section 9, with the exception of radiographic assessments which may be performed per local standard of care.

# 7.6 Treatment Compliance

# 7.6.1 Rucaparib Treatment Compliance

Study site personnel will review dosing information with the patient (or legally authorized representative) on scheduled clinic visit days, providing instructions regarding dose, dose frequency and the number of tablets to be taken for each dose. Patients (or legally authorized representative) will be instructed to keep all unused containers (empty, partially used, and/or

unopened) for accountability at the next scheduled clinic visits. A compliance check and tablet count will be performed by study personnel during clinic visits. Study site personnel will record compliance information in the eCRF.

Every effort should be made to ensure patients return to the clinic with their study drug containers/unused study drug at each study drug dispensation visit. Study site personnel should conduct a verbal review of dosing with the patient and document the discussion in the patient's medical record. This may serve as source documentation for the purpose of entering dosing data in the appropriate eCRF.

### 7.6.2 Comparator Therapy Treatment Compliance

Comparator therapy will be managed by the study site for each patient following the institutional guidelines or Prescribing Information for each agent.

For abiraterone and enzalutamide, study site personnel will review dosing information with the patient (or legally authorized representative) on scheduled clinic visit days, providing instructions regarding dose, dose frequency and the number of tablets/capsules to be taken for each dose. Patients (or legally authorized representative) will be instructed to keep all unused containers (empty, partially used, and/or unopened) for accountability for any product provided by the sponsor at the next scheduled clinic visits. A compliance check and tablet/capsule count will be performed by study personnel during clinic visits. Study site personnel will record compliance information in the eCRF.

Every effort should be made to ensure patients return to the clinic with their study drug containers/unused study drug at each study drug dispensation visit. Study site personnel should conduct a verbal review of dosing with the patient and document the discussion in the patient's medical record. This may serve as source documentation for the purpose of entering dosing data in the appropriate eCRF.

For docetaxel, site personnel should record dosing data (changes, interruptions, etc.) in the source records and in the appropriate eCRF.

# 7.7 Accountability of Protocol-specified Treatment

Study personnel will maintain accurate records of study drug receipt, dispensation, use, return, destruction, and reconciliation for study drugs provided by the sponsor. The IXRS will be used to manage study drug inventory at all sites. In order to function properly, the system will require real-time entry of study drug receipt, dispensation, destruction, etc. by study personnel at the study site.

The site is responsible for the return or destruction of study drug supplied by the sponsor as required. Authorization to destroy study drug at the site that has not been dispensed to a patient (eg, expired study drug), must be requested from the sponsor prior to destruction. Any study drug supplied by the sponsor accidentally or deliberately destroyed must be accounted for. All study drug containers must be accounted for prior to their destruction at the study center, according to institutional procedures for disposal of cytotoxic chemotherapeutic drugs. Unused study drug

containers should be destroyed on-site if possible. If destruction on site is not possible, supply should be returned to the drug depot.

During the course of the study and at completion of the study, the number of study drug containers received, dispensed, returned, and destroyed must be reconciled.

For comparator therapy that is sourced locally, the study site should follow local drug accountability practices.

#### 8 PRIOR AND CONCOMITANT THERAPY

Patients who have received prior treatment with a PARPi including IV or oral rucaparib, prior treatment with chemotherapy (eg docetaxel, mitoxantrone, cyclophosphamide, platinum-based agents) for mCRPC are not eligible to participate in this study. Prior treatment with docetaxel (or other taxane chemotherapy) administered for castration-sensitive disease is permitted.

All procedures performed (eg, thoracentesis, etc.) during the study must be documented in the eCRF.

# 8.1 Supportive Care

During the study, supportive care (eg, antiemetics; analgesics for pain control) may be used at the investigator's discretion and in accordance with institutional procedures. Supportive care must be recorded for each patient in the appropriate section of the eCRF.

Continuation of low-dose corticosteroid therapy that has been stable prior to study entry is permitted (see Section 6.3). A low dose is considered 5-15 mg/day of prednisone or prednisolone, and 0.5-3 mg/day of dexamethasone. For corticosteroids administered in combination with comparator therapy during the study, see Section 7.1.2.

Erythropoietin, darbepoetin alfa, and/or hematopoietic colony-stimulating factors for treatment of cytopenias should be administered according to institutional guidelines. Transfusion thresholds for blood product support will be in accordance with institutional guidelines.

# 8.2 Radiotherapy

Palliative radiotherapy for the treatment of painful bony metastasis is permitted during the study. Treatment with rucaparib should be held prior to initiation of radiation therapy and until the patient has recovered from any radiation related toxicity. Radiotherapy to soft-tissue lesions (either target or non-target) renders these inevaluable by RECIST Version 1.1, and is therefore discouraged during the Treatment Phase of the study.

# 8.3 Luteinizing Hormone-releasing Hormone Analogs

For patient who have not undergone an orchiectomy and are currently being treated with LHRH analogs at the time of consent, therapy must be continued throughout the study.

# 8.4 Anticancer or Experimental Therapy

No other anticancer therapies (including chemotherapy, radiation [except for palliative radiotherapy to bone metastases], antibody therapy, immunotherapy, gene therapy, angiogenesis inhibitors, or other experimental drugs) of any kind will be permitted while the patient is taking study treatment in the study (ie, unless in follow-up). Prior treatment with anticancer therapies must have been completed at least 14 days prior to the first dose of study drug. Prior treatment with hormonal therapies (with the exception of LHRH analog) must be discontinued at least 7 days prior to the first dose of study drug.

# 8.5 CYP450 Isoenzyme Inhibitors, Inducers, and Substrates

Based on the results from the CYP interaction clinical study CO-338-044, rucaparib is a moderate inhibitor of CYP1A2, and a weak inhibitor of CYP2C9, CYP2C19, and CYP3A. Caution should be used in patients on rucaparib taking concomitant medicines that are sensitive substrates of CYP1A2, CYP2C9, and/or CYP3A (Appendix 4). Patients taking phenytoin, a CYP2C9 substrate with a narrow therapeutic window, should have therapeutic drug level monitored while using concomitantly with rucaparib.

Although in vitro rucaparib metabolism mediated by CYP3A4 was slow, a significant contribution of CYP3A4 in vivo cannot be excluded. Caution should be used for concomitant use of strong CYP3A4 inhibitors or inducers.

# 8.6 Therapies to Control Bone Loss

Patients cannot have initiated denosumab or bisphosphonate therapy or adjusted bisphosphonate or demosumab dose/regimen within 28 days prior to first dose of study drug. Patients on a stable denosumab or bisphosphonate regimen are eligible and may continue treatment. Initiation of bisphosphonates or other approved bone targeting agents if clinically indicated is allowed, and should not result in study treatment discontinuation unless patient has radiographic evidence of disease progression.

# 8.7 Anticoagulants

Rucaparib is a weak inhibitor of CYP2C9 in vivo. Caution should be exercised in patients receiving rucaparib and concomitant warfarin (Coumadin). Patients taking warfarin should have INR monitored regularly per standard institutional practice.

## 8.8 Other Concomitant Medications

Therapies considered necessary for the patient's well-being may be given at the discretion of the investigator and should be documented in the eCRF. Other concomitant medications, except for analgesics, chronic treatments for concomitant medical conditions, or agents required for life-threatening medical problems, should be avoided. Herbal and complementary therapies should not be encouraged because of unknown side effects and potential drug interactions, but any taken by the patient should be documented appropriately in the eCRF.

Rucaparib marginally increased digoxin AUC by 20%. Caution should be exercised for patients receiving rucaparib and requiring concomitant medication with digoxin. Patients taking digoxin should have their digoxin levels monitored after starting rucaparib and then regularly per standard clinical practice.

In vitro, rucaparib is a potent inhibitor of MATE 1 and MATE2-K, a moderate inhibitor of OCT1, and a weak inhibitor of OCT2. As inhibition of these transporters could decrease renal elimination and liver uptake of metformin, caution is advised when metformin is co-administered with rucaparib.

## 9 STUDY PROCEDURES AND ACTIVITIES BY VISIT

#### 9.1 Schedule of Assessments

Table 5 and Table 6 summarize the procedures and assessments to be performed for patients randomized to rucaparib or physician's choice of comparator during the study.

Table 7 summarizes the procedures and assessments for patients in the Cross-over Phase. Study procedures and assessments should be performed as close to the scheduled time as possible, but within  $\pm$  3 days of the scheduled time unless otherwise stated. Tumor assessment visits are scheduled relative to Study Day 1.

Table 5. Schedule of Assessments for Patients Randomized to Rucaparib or Physician's Choice of Abiraterone Acetate or Enzalutamide

| | | | | | Treatment Phase | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure <sup>a</sup> | Pre-<br>screening<br>Phase | Screening | ization | Week 1 | | | | Week 9 &<br>every 4 weeks<br>thereafter | Post-Treatment Phase | | | |
| | | Day -28 to<br>Day -1 | Day -14<br>to<br>Day - | Randomization | Stud<br>y<br>Day 1 <sup>b</sup> | Study<br>Day 15 | Study<br>Day 29 | Study<br>Day 43 | Day 57 & every 28 days thereafter | Freatment<br>Discontin-<br>uation <sup>w</sup> | | Long-term<br>Follow-up |
| Informed Consent | Xc | X | | | | | | | | | | |
| BRCA1/2, ATM gene mutation<br>assessment from ctDNA blood and tumor<br>sample <sup>c, d</sup> | X <sup>c</sup> | | | | | | | | | | | |
| Medical/Oncology History <sup>e</sup> | | X | | | | | | | | | | |
| Blood samples for plasma ctDNA analysis <sup>f</sup> | | X | | | X | | | | | X | | |
| Physical Examination, Weight, Height <sup>g</sup> | | X | | | X | X | X | X | X | X | X | |
| Vital Signs <sup>h</sup> | | X | | | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>i</sup> | | X | | | | | | | | X | | |
| Prior/Concomitant Medications/Procedures | | X | | | X | X | X | X | X | X | X | |
| Tumor Assessment/CT/MRI/Bone Scan <sup>j</sup> | | X | | | | | | | $X^k$ | $X^{l}$ | $X^{l}$ | $X^{l}$ |
| Archival Primary/ Metastatic Tumor<br>Tissue Sample for retrospective testing <sup>m</sup> | | X | | | | | | | | | | |
| Patient-reported outcome (BPI-SF, analgesic drug score, FACT-P, EQ-5D-5L) <sup>n</sup> | | | X | | X | | X | | X | X | X | X |
| ECOG Performance Status | | | X | | X | X | X | X | X | X | X | |
| Serum Testosterone | | X | | | | | | | | | | |
| PSA Measurement <sup>o</sup> | | X | | | X | | X | | X | X | | |
| Clinical Laboratory Assessments <sup>p</sup> | | | X | | X | X | X | X | X | X | X | |
| Pharmacogenomic blood sample <sup>q</sup> | | | | | X | | | | | | | |
| Randomization to Study Treatment | | | | X | | | | | | | | |
| Study Drug Dispensation | | | | | X | | X | | X | | | |
| Adverse Events <sup>r</sup> | (X) | (X) | (X) | | X | X | X | X | X | X <sup>s</sup> | Xs | |
| Plasma PK Sample (Rucaparib patients only) | | | | | | | X <sup>t</sup> | | X <sup>t</sup> | | | |

| Post-progression Tumor Biopsy | X <sup>u</sup> | | |
|---------------------------------|----------------|---|---|
| (Optional) | | | |
| Subsequent Treatments, AESIs, & | | X | X |
| Survival | | | |

Abbreviations: AESI = adverse event of special interest, ALP = alkaline phosphatase, ALT = alanine transaminase, AML = acute myeloid leukemia, ANC = absolute neutrophil count, AST = aspartate transaminase, ATM = ataxia telangiectasia mutated serine/threonine kinase, BRCA1/2 = breast cancer 1 or breast cancer 2 gene, BPI-SF = Brief Pain Inventory – Short Form, BUN = blood urea nitrogen, CO<sub>2</sub> = bicarbonate, CR = complete response, CT = computer tomography, ctDNA = circulating cell-free tumor DNA, DNA = deoxyribonucleic acid, ECG = electrocardiogram, ECOG = Eastern Cooperative Oncology Group, EQ-5D-5L = EuroQol 5 dimensions 5 level questionnaire, FACT-P = Functional Assessment of Cancer Therapy-Prostate, Hct = hematocrit, HDL = high density lipoprotein, HDP = hydroxydiphosphonate, Hgb = hemoglobin, INR = international normalized ratio, LDL= low density lipoprotein, MCH = mean corpuscular hemoglobin, MCHC = mean corpuscular hemoglobin concentration, MCV = mean corpuscular volume, MDP = methylene diphosphonate, MDS = myelodysplastic syndrome, MRI = magnetic resonance imaging, PET = positron emission tomography, PK = pharmacokinetic, PR = partial response, PV = Pharmacovigilance, RBC = red blood cell count, RECIST = Response Evaluation Criteria in Solid Tumors. SAE = serious adverse event. WBC = white blood cells

- a The study visit window is ±3 days, unless noted otherwise for a particular assessment. Study visits should take into account the patient's study drug supply.
- b First dose of study drug is designated as Study Day 1 and must occur within 3 days after randomization. Procedures required on Study Day 1 may be omitted if completed ≤ 3 days earlier during the Screening Phase with the exception of ctDNA which will be collected during Pre-Screening and must be collected during Screening and on Study Day 1.
- Pre-Screening is for central testing of plasma ctDNA and tumor tissue samples to identify patients with qualifying deleterious BRCA1/2 and ATM gene mutations. To enter Pre-Screening, patients should have evidence of radiographic or biochemical disease progression, and be eligible for this study as their immediate next therapy. Both plasma ctDNA and tumor tissue samples should be submitted simultaneously. If plasma or tissue testing results in failure, additional samples may be submitted, as available. Pre-Screening requires a separate informed consent form.
- d Tissue for Pre-Screening should be from biopsy or resection specimen from metastatic tumor, if there is a lesion suitable for biopsy. A biopsy or resection of a visceral or nodal site of metastasis is preferred; however a biopsy of primary tumor or of a site of bony metastasis is also acceptable (soft tissue biopsy preferred over bone site biopsy). If a metastatic biopsy is not feasible, archival tissue samples can be submitted. Archival tissue for Pre-Screening should be < 3 years old. Submission of a tumor block with a tumor content ≥ 30% with a minimum of 80% nucleated cellular content should be provided.
- <sup>e</sup> Includes demographic information. Patient's medical record must include prior treatments received, dates of administration, date of progression and how assessed, PSA and radiology reports.
- f Blood samples for plasma ctDNA analysis during Screening, before dosing on Study Day 1, and at Treatment Discontinuation are for pharmacodynamic assessments and companion diagnostic development. Plasma ctDNA is required on Study Day 1 even when it was previously collected.
- g Height at screening only.
- h Vital signs (blood pressure, pulse, and temperature) to be taken on drug administration days, after the patient has been resting for at least 5 minutes.
- i Heart rate, pulse rate, QRS, QT, QTc, and rhythm. Investigator to review results and assess as normal or abnormal (clinically significant or not clinically significant). ECGs to be repeated as clinically indicated.
- Tumor assessments to consist of clinical examination and appropriate imaging techniques (CT scans of the chest, abdomen and pelvis, with appropriate slice thickness); CT with contrast is preferred, non-contrast may be used where clinically indicated. MRI may be used in place of CT scan if requested by local authorities. Where indicated for neurological symptoms, MRI of spine and skull to be conducted. Radionuclide bone scanning (whole body) using 99mTc-MDP or HDP. Other studies, such as PET/CT, may also be performed. The same methods used to detect lesions at baseline are to be used to follow the same lesions throughout the clinical study. If a patient has known brain metastases, this disease should be evaluated at each required assessment.
- bisease assessment by CT/MRI and bone scans will be performed during screening, during the treatment phase, and Treatment Discontinuation, and if applicable, during follow up. Modified RECIST Version 1.1/PCWG3 criteria will be used. Tumor assessments will occur at the end of every 8 weeks from Study Day 1, up to 24 weeks (Study Weeks 9, 17, 25) and then every 12 weeks thereafter (Study weeks 37, 49, 61, etc.). If a CR or PR is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented.
- Radiographic assessments should continue for all patients until <u>central</u> confirmation of radiographic progression, including any patient who discontinued from study treatment for reason other than disease progression or death. Tumor assessments should be performed during the Treatment Discontinuation Visit, 28-day Follow-up, or during Long-term Follow-up if the reason was other than central radiographically confirmed disease progression and it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since the last assessment. Tumor assessments should continue on schedule (ie, every 8 or 12 weeks) during Long-term Follow-up until central radiographically confirmed disease progression. After the primary endpoint analysis is performed central confirmation of radiographic progression will no longer occur; radiographic progression and confirmation of disease progression will be performed by the investigator.
- m If archival primary or metastatic tumor tissue was not submitted during Pre-Screening, a specimen should be submitted during the Screening Phase or after enrollment for retrospective testing by the central laboratory. Archival tissue submitted during Screening for retrospective testing can be > 3 years old. Refer to the Pathology Charter for detailed sample handling instructions.
- The BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments must be completed prior to other scheduled study procedures and dosing (if applicable). During long-term follow up, if possible, PROs to be collected to coincide on days when tumor assessments are performed. PRO assessments should continue to be collected until confirmed radiologic disease progression.
- <sup>o</sup> All PSA measurements are performed by the local laboratory.
- P Clinical laboratory assessments will be done locally. Hematology should include RBC and parameters (Hgb, Hct, MCV, MCH, MCHC) and reticulocyte count, WBC and differential (with ANC), and platelet count. Serum chemistry should include total protein, albumin, creatinine for estimating GFR using the Cockcroft Gault formula, BUN or urea, total bilirubin, ALP, ALT, AST, LDH, lipid panel (total cholesterol, LDL, HDL, and triglycerides), glucose, sodium, potassium, chloride, CO<sub>2</sub>, calcium, and phosphorus. Fasting is not required. Urinalysis should include protein, glucose, blood, pH, and ketones. Microscopic evaluation to assess abnormal findings, if clinically warranted by investigator.
- <sup>q</sup> If pharmacogenomic sample is not collected prior to Study Day 1, it must be collected as soon as possible thereafter.
- AEs (inclusive of SAEs and AESIs) occurring after first dose of study drug through to 28 days after last dose of study drug will be recorded. In addition, SAEs occurring after signing of ICF that were related to a Pre-Screening or Screening procedure will also be reported.
- Ongoing SAEs, AESIs and Grade 3/4 AEs will be followed to resolution or stabilization. SAEs/AESIs are collected per Clovis Oncology PV guidelines and reported in the Clovis Oncology PV database through the 28-day Follow-up Visit after the last dose of rucaparib. Ongoing SAEs and AESIs at the time of the 28-day Follow-up Visit will be followed to resolution, stabilization, or lost to follow-up. After this visit, only SAEs considered as potentially related to study drug, (including pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug), and AESIs of MDS and AML irrespective of causality, should be reported.
- PK within 1 hour prior to the morning dose on Study Day 29, Day 57, Day 85, and Day 113. The PK sample should be collected close to 12 hours post the last dose (even if the morning dose on the specified visit days is not administered).
- <sup>u</sup> Optional tumor biopsy should be collected from patients at time of disease progression. Refer to the Pathology Charter for detailed sample handling instructions.
- All patients discontinued from treatment, regardless of reason, should be followed for subsequent treatments and survival every 12 weeks relative to the last dose of study drug until death, loss to follow-up, withdrawal of consent from study, or closure of the study. Follow-up can be performed via the telephone and can be completed to coincide with scheduled tumor assessments and/or PRO during this period.
- Patients eligible for cross-over to rucaparib will have a Treatment Discontinuation Visit after discontinuation of comparator therapy, but are not required to complete the 28-day follow-up visit on their original study treatment.

Table 6. Schedule of Assessments for Patients Randomized to Physician's Choice of Docetaxel

| | | | | | Treatment Phase | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Screeni | ization | Week<br>1 | Week 1<br>and every<br>3 weeks<br>thereafter | Week 1<br>and every<br>4 weeks<br>thereafter | Week 9<br>and every<br>8 weeks<br>thereafter | Post-Treatment Phase | | | |
| Procedurea | Pre-<br>screening<br>Phase | Day -28<br>to<br>Day -1 | Day -14<br>to<br>Day -1 | Randomization | Study<br>Day 1 | Study Day 1 and every 21 days thereafter | Study Day 1 and every 28 days thereafter | Study Day 57 and every 56 days thereafter | Treatment<br>Discontinuati<br>on' | 28-day<br>Follow-<br>up <sup>v</sup> | Long-t<br>erm<br>Follow<br>-up |
| Informed Consent | X <sup>c</sup> | X | | | | | | | | | |
| BRCA1/2, ATM gene mutation assessment from ctDNA blood and tumor sample <sup>c, d</sup> | X° | | | | | | | | | | |
| Medical/Oncology History <sup>e</sup> | | X | | | | | | | | | |
| Blood samples for plasma ctDNA analysis <sup>f</sup> | | X | | | X | | | | X | | |
| Physical Examination, Weight,<br>Height <sup>g</sup> | | X | | | | X | | | X | X | |
| Vital Signs <sup>h</sup> | | X | | | | X | | | X | X | |
| 12-lead ECG <sup>i</sup> | | X | | | | | | | X | | |
| Prior/Concomitant Medications/Procedures | | X | | | | X | | | X | X | |
| Tumor Assessment/CT/MRI/Bone<br>Scan <sup>j</sup> | | X | | | | | | $X^k$ | $X^{l}$ | $X^{l}$ | $X^{l}$ |
| Archival Primary/ Metastatic<br>Tumor Tissue Sample for<br>retrospective testing <sup>m</sup> | X | | | | | | | | | | |
| Patient-reported outcome (BPI-SF, analgesic drug score, FACT-P, EQ-5D-5L) <sup>n</sup> | | | X | | | | X | | X | X | X |
| ECOG Performance Status | | | X | | | X | | | X | X | _ |
| Serum Testosterone | | X | | | | | | | | | |
| PSA Measurement <sup>o</sup> | | X | | | | X | | | X | | |
| Clinical Laboratory Assessments <sup>p</sup> | | | X | | | X | | | X | X | |
| Pharmacogenomic blood sample <sup>q</sup> | | | | | X | | | | | | |
| Randomization to Study | | | | X | | | | | | | |
| Treatment | | | | | | | | | | | |

| Docetaxel Administration | | | | X | | | | |
|---|---|---|---|---|---|---|---|---|
| Adverse Events <sup>r</sup> | (X) | (X) | (X) | X | X | $X^{s}$ | Xs | |
| Post-progression Tumor Biopsy (Optional) | | | | | | $X^{t}$ | | |
| Subsequent Treatments, AESIs, & Survival <sup>u</sup> | | | | | | | X | X |

Abbreviations: AESI = adverse event of special interest, ALP = alkaline phosphatase, ALT = alanine transaminase, ANC = absolute neutrophil count, AML = acute myeloid leukemia, AST = aspartate transaminase, ATM = ataxia telangiectasia mutated serine/threonine kinase, BRCA1/2 = breast cancer 1 or breast cancer 2 gene, BPI-SF = Brief Pain Inventory - Short Form, BUN = blood urea nitrogen, CO<sub>2</sub> = bicarbonate, CR = complete response, CT = computer tomography, ctDNA = circulating cell-free tumor DNA, DNA = deoxyribonucleic acid, ECG = electrocardiogram, ECOG = Eastern Cooperative Oncology Group, EQ-5D-5L = EuroQol 5 dimensions 5 level questionnaire, FACT-P = Functional Assessment of Cancer Therapy-Prostate, Hct = hematocrit, HDL= high density lipoprotein, HDP = hydroxydiphosphonate, Hgb = hemoglobin, INR = international normalized ratio, LDL= low density lipoprotein, MCH = mean corpuscular hemoglobin, MCHC = mean corpuscular hemoglobin concentration, MCV = mean corpuscular volume, MDP = methylene diphosphonate, MDS = myelodysplastic syndrome, MRI = magnetic resonance imaging, PET = positron emission tomography, PR = partial response, PV = Pharmacovigilance, RBC = red blood cell count, RECIST = Response Evaluation Criteria in Solid Tumors, SAE = serious adverse event. WBC = white blood cells

- a The study visit window is ±3 days, unless noted otherwise for a particular assessment. Study visits should take into account the patient's study drug supply.
- First dose of study drug is designated as Study Day 1 and **must occur within 3 days after randomization**. Procedures required on Study Day 1 may be omitted if completed ≤ 3 days earlier during the Screening Phase with the exception of ctDNA which will be collected during Pre-Screening and must be collected during Screening and on Study Day 1. Docetaxel administration will continue up to a maximum of 10 cycles (whereupon no study treatment shall be given, but assessments continue).
- Pre-Screening is for central testing of plasma ctDNA and tissue samples to identify patients with qualifying deleterious BRCA1/2 or ATM gene mutations. To enter Pre-Screening, patients should have evidence of radiographic or biochemical disease progression, and be eligible for this study as their immediate next therapy. Both plasma ctDNA and tumor tissue samples should be submitted simultaneously. If plasma or tissue testing results in failure, additional samples may be submitted, as available. Pre-Screening requires a separate informed consent form.
- d Tissue for Pre-Screening should be from biopsy or resection specimen from metastatic tumor, if there is a lesion suitable for biopsy. A biopsy or resection of a visceral or nodal site of metastasis is preferred; however a biopsy of primary tumor or of a site of bony metastasis is also acceptable (soft tissue biopsy preferred over bone site biopsy). If a metastatic biopsy is not feasible, archival tissue samples can be submitted. Archival tissue for Pre-Screening should be < 3 years old. Submission of a tumor block with a tumor content ≥ 30% with a minimum of 80% nucleated cellular content should be provided.
- <sup>e</sup> Includes demographic information. Patient's medical record must include prior treatments received, dates of administration, date of progression and how assessed, PSA and radiology reports.
- f Blood samples for plasma ctDNA analysis during Screening, before dosing on Study Day 1, and at Treatment Discontinuation are for pharmacodynamic assessments and companion diagnostic development. Plasma ctDNA is required on Study Day 1 even when it was previously collected.
- g Height at screening only.
- h Vital signs (blood pressure, pulse, and temperature) to be taken on drug administration days, after the patient has been resting for at least 5 minutes.
- Heart rate, pule rate, QRS, QT, QTc, and rhythm. Investigator to review results and assess as normal or abnormal (clinically significant or not clinically significant). ECGs to be repeated as clinically indicated.
- Tumor assessments to consist of clinical examination and appropriate imaging techniques (CT scans of the chest, abdomen and pelvis, with appropriate slice thickness); CT with contrast is preferred, non-contrast may be used where clinically indicated. MRI may be used in place of CT scan if requested by local authorities. Where indicated for neurological symptoms, MRI of spine and skull to be conducted. Radionuclide bone scanning (whole body) using 99mTc-MDP or HDP. Other studies, such as PET/CT, may also be performed. The same methods used to detect lesions at baseline are to be used to follow the same lesions throughout the clinical study. If a patient has known brain metastases, this disease should be evaluated at each required assessment.

- Disease assessment by CT/MRI and bone scans will be performed during screening, during the treatment phase, and Treatment Discontinuation, and if applicable, during follow up. Modified RECIST Version 1.1/PCWG3 criteria will be used. End of every 8 weeks from Study Day 1, up to 24 weeks (Study Weeks 9, 17, 25) and then every 12 weeks thereafter (Study weeks 37, 49, 61, etc.). If a CR or PR is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented.
- Radiographic assessments should continue for all patients until <u>central</u> confirmation of radiographic progression, including any patient who discontinued from study treatment for reason other than disease progression or death. Tumor assessments should be performed during the Treatment Discontinuation Visit, 28-day Follow-up, or during Long-term Follow-up if the reason was other than radiographically confirmed disease progression and it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since the last assessment. Tumor assessments should continue on schedule (ie, every 8 or 12 weeks) during Long-term Follow-up until central radiographically confirmed disease progression. After the primary endpoint analysis is performed central confirmation of radiographic progression will no longer occur; radiographic progression and confirmation of disease progression will be performed by the investigator.
- m If archival primary or metastatic tumor tissue is not submitted during Pre-Screening, a specimen should be submitted during the Screening Phase or after enrollment for retrospective testing by the central laboratory. Archival tissue submitted during Screening for retrospective testing can be > 3 years old. Refer to the Pathology Charter for detailed sample handling instructions.
- The BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments must be completed every 4 weeks (±7 days) prior to other scheduled study procedures and dosing (if applicable). During long-term follow up, if possible, PROs to be collected to coincide on days when tumor assessments are performed. Collection of PROs at any other study visit within 7 days of the scheduled time point is permitted. PRO assessments should continue to be collected until confirmed radiologic disease progression.
- <sup>o</sup> All PSA measurements are performed by the local laboratory.
- P Clinical laboratory assessments will be done locally. Hematology should include RBC and parameters (Hgb, Hct, MCV, MCH, MCHC) and reticulocyte count, WBC and differential (with ANC), and platelet count. Serum chemistry should include total protein, albumin, creatinine for estimating GFR using the Cockcroft Gault formula, BUN or urea, total bilirubin, ALP, ALT, AST, LDH, lipid panel (total cholesterol, LDL, HDL, and triglycerides), glucose, sodium, potassium, chloride, CO<sub>2</sub>, calcium, and phosphorus. Fasting is not required. Urinalysis should include protein, glucose, blood, pH, and ketones. Microscopic evaluation to assess abnormal findings, if clinically warranted by investigator.
- <sup>q</sup> If pharmacogenomic sample is not collected prior to Study Day 1, it must be collected as soon as possible thereafter.
- AEs (inclusive of SAEs and AESIs) occurring after first dose of study drug through to 28 days after last dose of study drug will be recorded. In addition, SAEs occurring after signing of ICF that were related to a Pre-Screening or Screening procedure will also be reported.
- Ongoing SAEs, AESIs and Grade 3/4 AEs will be followed to resolution or stabilization. SAEs/AESIs are collected per Clovis Oncology PV guidelines and reported in the Clovis Oncology PV database through the 28-day Follow-up Visit after the last dose of rucaparib. Ongoing SAEs and AESIs at the time of the 28-day Follow-up Visit will be followed to resolution, stabilization, or lost to follow-up. After this visit, only SAEs considered as potentially related to study drug (including pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug), and AESIs of MDS and AML irrespective of causality, should be reported.
- Optional tumor biopsy should be collected from patients at time of disease progression. Refer to the Pathology Charter for detailed sample handling instructions.
- <sup>u</sup> All patients discontinued from treatment, regardless of reason, should be followed for subsequent treatments and survival every 12 weeks relative to the last dose of study drug until death, loss to follow-up, withdrawal of consent from study, or closure of the study. Follow-up can be performed via the telephone and can be completed to coincide with scheduled tumor assessments and/or PRO during this period.
- Patients eligible for cross-over to rucaparib will have a Treatment Discontinuation Visit after discontinuation of comparator therapy, but are not required to complete the 28-day follow-up visit on their original study treatment.

Table 7. Schedule of Assessments for Patients Who Cross over to Rucaparib after Physician's Choice Comparator

| | | | | 7 | reatment Pl | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| XO-Screening Phase | | XO-Week<br>1 | XO-Week | XO-Week<br>5 | XO-Week 7 | XO-Week<br>9 & every<br>4 weeks<br>thereafter | Post-Trea | atment Ph | ase | |
| Procedure <sup>a</sup> | Day -28 to<br>Day -1 | Day -14<br>to<br>Day -1 | XO-Study<br>Day 1 <sup>b</sup> | XO-Study<br>Day 15 | XO-Study<br>Day<br>29 | XO-Study<br>Day 43 | XO-Day 57<br>& every<br>28 days<br>thereafter | Treatment<br>Discontinuation | 28-day<br>Follow<br>-up | Long-<br>term<br>Follow-up |
| Cross-over Informed Consent | X | | | | | | | | | |
| Blood samples for plasma ctDNA analysis | | | X | | | | | X | | |
| Physical Examination,<br>Weight, Height <sup>c</sup> | X | | X | X | X | X | X | X | X | |
| Vital Signs <sup>d</sup> | X | | X | X | X | X | X | X | X | |
| 12-lead ECG <sup>e</sup> | X | | | | | | | X | | |
| Prior/Concomitant Medications/Procedures | X | | X | X | X | X | X | X | X | |
| Tumor<br>Assessment/CT/MRI/Bone<br>Scan <sup>f</sup> | X | | | | | | Xg | $X^{ m h}$ | X <sup>h</sup> | $X^{h}$ |
| Patient-reported outcome<br>(BPI-SF, analgesic drug<br>score, FACT-P, EQ-5D-5L) <sup>i</sup> | | X | X | | X | | X | X | X | X |
| ECOG Performance Status | | X | X | X | X | X | X | X | X | |
| Serum Testosterone | X | | | | | | | | | |
| PSA Measurement <sup>j</sup> | X | | X | | X | _ | X | X | | |
| Clinical Laboratory<br>Assessments <sup>k</sup> | | X | X | X | X | X | X | X | X | |
| Study Drug Dispensation | | | X | | X | | X | | | |
| Adverse Events <sup>1</sup> | (X) | (X) | X | X | X | X | X | X <sup>m</sup> | X <sup>m</sup> | |
| Post-progression Tumor<br>Biopsy (Optional) | | | | | | | | X <sup>n</sup> | | |
| Subsequent Treatments,<br>AESIs, & Survival <sup>o</sup> | | | | | | | | | X | X |

Abbreviations: AESI = adverse event of special interest, ALP = alkaline phosphatase, ALT = alanine transaminase, AML = acute myeloid leukemia, ANC = absolute neutrophil count, AST = aspartate transaminase, BPI-SF = Brief Pain Inventory – Short Form, BUN = blood urea nitrogen, CO<sub>2</sub> = bicarbonate, CR = complete response, CT = computer tomography, ctDNA = circulating cell-free tumor DNA, DNA = deoxyribonucleic acid, ECG = electrocardiogram, ECOG = Eastern Cooperative Oncology Group, EQ-5D-5L = EuroQol 5 dimensions 5 level questionnaire, FACT-P = Functional Assessment of Cancer Therapy-Prostate, Hct = hematocrit, HDL= high density lipoprotein, HDP = hydroxydiphosphonate, Hgb = hemoglobin, INR = international normalized ratio, LDL= low density lipoprotein, MCH = mean corpuscular hemoglobin, MCHC = mean corpuscular hemoglobin concentration, MCV = mean corpuscular volume, MDP = methylene diphosphonate, MDS = myelodysplastic syndrome, MRI = magnetic resonance imaging, PET = positron emission tomography, PK = pharmacokinetic, PR = partial response, PV = Pharmacovigilance, RBC = red blood cell count, RECIST = Response Evaluation Criteria in Solid Tumors, SAE = serious adverse event, WBC = white blood cells

- a The study visit window is ±3 days, unless noted otherwise for a particular assessment. Study visits should take into account the patient's study drug supply.
- b First dose of study drug is designated as XO-Study Day 1. Procedures required on XO-Study Day 1 may be omitted if completed ≤ 3 days earlier during the Screening Phase.
- c Height at screening only.
- d Vital signs (blood pressure, pulse, and temperature) to be taken on drug administration days, after the patient has been resting for at least 5 minutes.
- <sup>e</sup> Heart rate, pulse rate, QRS, QT, QTc, and rhythm. Investigator to review results and assess as normal or abnormal (clinically significant or not clinically significant). ECGs to be repeated as clinically indicated.
- Tumor assessments to consist of clinical examination and appropriate imaging techniques (CT scans of the chest, abdomen and pelvis, with appropriate slice thickness); CT with contrast is preferred, non-contrast may be used where clinically indicated. MRI may be used in place of CT scan if requested by local authorities. Where indicated for neurological symptoms, MRI of spine and skull to be conducted. Radionuclide bone scanning (whole body) using 99mTc-MDP or HDP. Other studies, such as PET/CT, may also be performed. The same methods used to detect lesions at baseline are to be used to follow the same lesions throughout the clinical study. If a patient has known brain metastases, this disease should be evaluated at each required assessment.
- Disease assessment by CT/MRI and bone scans will be performed during screening, during the treatment phase, and Treatment Discontinuation, and if applicable, during follow up. Modified RECIST Version 1.1/PCWG3 criteria will be used. Tumor assessments will occur at the end of every 8 weeks from XO-Study Day 1, up to 24 weeks (XO-Study Weeks 9, 17, 25) and then every 12 weeks thereafter (XO-Study weeks 37, 49, 61, etc.). If a CR or PR is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented.
- h Radiographic assessments should continue for all patients until confirmation of radiographic progression by investigator assessment, including any patient who discontinued from study treatment for reason other than disease progression or death. Tumor assessments should be performed during the Treatment Discontinuation Visit, 28-day Follow-up, or during Long-term Follow-up if the reason was other than radiographically confirmed disease progression and it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since the last assessment. Tumor assessments should continue on schedule (ie, every 8 or 12 weeks) during Long-term Follow-up until radiographically confirmed disease progression by investigator assessment.
- The BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments must be completed prior to other scheduled study procedures and dosing (if applicable). During long-term follow up, if possible, PROs to be collected to coincide on days when tumor assessments are performed. PRO assessments should continue to be collected until radiologic disease progression is confirmed by investigator assessment.
- All PSA measurements are performed by the local laboratory.
- k Clinical laboratory assessments will be done locally. Hematology should include RBC and parameters (Hgb, Hct, MCV, MCH, MCHC) and reticulocyte count, WBC and differential (with ANC), and platelet count. Serum chemistry should include total protein, albumin, creatinine for estimating GFR using the Cockcroft Gault formula, BUN or urea, total bilirubin, ALP, ALT, AST, LDH, lipid panel (total cholesterol, LDL, HDL, and triglycerides), glucose, sodium, potassium, chloride, CO2, calcium, and phosphorus. Fasting is not required. Urinalysis should include protein, glucose, blood, pH, and ketones. Microscopic evaluation to assess abnormal findings, if clinically warranted by investigator.
- AEs (inclusive of SAEs and AESIs) occurring after first dose of study drug through to 28 days after last dose of study drug will be recorded. In addition, SAEs occurring after signing of ICF that were related to a Pre-Screening or Screening procedure will also be reported.

- Ongoing SAEs, AESIs and Grade 3/4 AEs will be followed to resolution or stabilization. SAEs/AESIs are collected per Clovis Oncology PV guidelines and reported in the Clovis Oncology PV database through the 28-day Follow-up Visit after the last dose of rucaparib. Ongoing SAEs and AESIs at the time of the 28-day Follow-up Visit will be followed to resolution, stabilization, or lost to follow-up. After this visit, only SAEs considered as potentially related to study drug (including pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug), and AESIs of MDS and AML irrespective of causality, should be reported.
- Deprive a contraction of the Pathology Charter for detailed sample handling instructions.
- All patients discontinued from treatment, regardless of reason, should be followed for subsequent treatments and survival every 12 weeks relative to the last dose of study drug until death, loss to follow-up, withdrawal of consent from study, or closure of the study. Follow-up can be performed via the telephone and can be completed to coincide with scheduled tumor assessments and/or PRO during this period.

## 9.2 Informed Consent

Patients are required to sign the Pre-Screening ICF prior to undergoing any Pre-Screening activities (ie, deleterious BRCA1/2 or ATM gene mutation testing), and are required to sign the Screening ICF prior to undergoing any other Screening assessments. Obtaining written informed consent does not signify the start of the Screening Phase as it begins when the first study-specific screening activity is performed.

The investigator or their designee shall discuss with each patient the nature of the study and its requirements. The information on the IRB/IEC approved consent form should be translated and communicated in the language the patient (or legally authorized representative) can understand.

Additionally, patients undergoing tumor tissue biopsy during Pre-Screening at the time of radiographic disease progression/randomized treatment discontinuation must provide additional consent for this procedure.

Patients who cross-over to treatment with rucaparib after confirmed radiographic disease progression must provide additional consent to continue treatment, as well as sponsor (or designee) approval of the radiology report confirming disease progression and eligibility. Details regarding cross-over to rucaparib are described in Section 9.7.

Patients with radiographic disease progression who are still receiving benefit and are allowed to continue study drug must also provide consent for continued treatment.

## 9.3 Pre-Screening Phase

Following written informed consent, and unless otherwise specified, the following assessments will be performed prior to Screening. Pre-Screening procedures may be repeated in the event of test failure.

Pre-screening is for central testing of plasma ctDNA and tumor tissue samples to identify patients with qualifying deleterious BRCA1/2 and ATM gene mutations. Patients with deleterious BRCA1/2 or ATM gene mutation identified through local testing need not enter Pre-Screening. To enter Pre-Screening, patients should have evidence of radiographic or biochemical disease progression, and be eligible for this study as their immediate next therapy. Patients must sign the Pre-Screening ICF.

## During Pre-Screening:

- Submit patient plasma sample for ctDNA analysis and tissue samples simultaneously
- Tissue should be from a newly obtained metastatic biopsy, if there is a lesion suitable for biopsy. A biopsy or resection of a visceral or nodal site of metastasis is preferred; however, a biopsy of primary tumor or of a site of bony metastasis is also acceptable.
- If a metastatic biopsy is not feasible, archival tissue samples can be submitted. Archival tissue should be < 3 years old. The most recently collected tumor tissue sample available that is of adequate quality (at least 30% tumor content with a minimum of 80% nucleated cellular content) should be provided.

• If plasma or tissue samples result in test failure, sites are encouraged to submit additional samples, as available, in order to obtain a successful test result

A central laboratory test result or a local laboratory test result is required for subsequent Screening of these patients

Refer to the Pathology Charter for detailed tissue sample handling instructions.

SAE monitoring is ongoing during Pre-Screening (only report if related to Pre-Screening procedures).

# 9.4 Screening Phase

Following written informed consent, and unless otherwise specified, the following assessments will be performed prior to randomization within the allowable windows of time as indicated below. Assessments performed within the specified windows, but prior to patient signing informed consent, are acceptable only if confirmed to have been standard of care. Screening procedures may be repeated if the findings/results are considered invalid or not representative of the patient's baseline medical status. When screening procedures are repeated, the rationale should be documented in the source file.

## 9.4.1 Screening: Up to 28 Days Prior to Randomization:

- Serum testosterone level measurement
- PSA measurement
- Medical/oncology history, including demographic information
- Plasma sample for ctDNA
- Physical examination by body system, including height and weight
- Vital signs (blood pressure, pulse, and body temperature)
- 12-lead ECG
- Prior and concomitant medications, any surgical/ medical procedures
- Tumor assessment: assessments should consist of clinical examination and appropriate imaging techniques (preferably CT scans of the chest, abdomen, and pelvis with appropriate slice thickness per modified RECIST Version 1.1); other studies (MRI, X-ray, positron emission tomography [PET]/CT, and ultrasound) may be performed if required. Radionuclide bone scanning (whole body) should be performed using 99mTc-methylene diphosphonate (MDP) or hydroxydiphosphonate (HDP). The same methods used to detect lesions at baseline are to be used to follow the same lesions throughout the clinical study.
  - If a patient has known brain metastases, this disease should be evaluated at each required assessment
- Archival primary and metastatic tumor tissue (if available, and not already submitted to the central laboratory) for retrospective testing by the central laboratory. Archival tissue samples > 3 years old are allowed for retrospective testing purposes. Samples may be submitted after enrollment. Refer to the Pathology Charter for detailed tissue sample handling instructions.

• SAE monitoring (only report if related to screening procedures)

# 9.4.2 Screening: Up to 14 Days Prior to Randomization:

- PRO collected using the BPI-SF (Appendix 5), FACT-P (Appendix 6), EQ-5D-5L (Appendix 7), and analgesic drug score instruments (Appendix 8); complete before other procedures
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis; see Section 9.12.2)
- ECOG performance status (Appendix 2);
- SAE monitoring (only report if related to screening procedures)

## 9.5 Treatment Phase

Patients are to be randomized to receive either rucaparib or the physician's choice of comparator therapy (Section 5.1.3) through IXRS after meeting eligibility criteria (Sections 6.2 and 6.3) and having completed screening assessments (Section 9.3).

The first dose of study drug must be administered  $\leq 3$  days after randomization and the day of first dose is Study Day 1.

During the treatment period, patients randomized to rucaparib will receive oral rucaparib tablets which should be taken BID at 600 mg/dose with 8 oz (240 mL) of water with or without food. At each study visit, the first dose of rucaparib will be taken in the clinic, with the remaining doses self-administered by the patient at home. Patients should take rucaparib at about the same time every day and should inform the clinic staff of any changes to their dose and timing of self-administration of oral rucaparib.

The choice of comparator therapy is at the discretion of the investigator from the regimens described in this protocol and must be specified prior to randomization. Refer to Sections 7.5.2 to 7.5.4 for dosing details.

Patients initially randomized and treated with comparator who have crossed over to rucaparib following radiographic progression will be required to sign a cross-over ICF as described in Section 9.7, meet eligibility criteria for the cross-over described in Section 6.4, and have sponsor (or designee) approval prior to crossing over to rucaparib treatment. Patients who cross-over to rucaparib will follow the procedures/assessments described in Section 9.8, Sections 9.5.1.1 to 9.5.1.5, Section 9.6.1, and Section 9.6.2.

- 9.5.1 Patients Randomized to Rucaparib, Physician's Choice of Abiraterone Acetate or Enzalutamide or Cross-over to Rucaparib
- 9.5.1.1 Study Day 1 (Week 1) and Cross-over Study Day 1 (XO Week 1)

The following procedures/assessments will be completed for all patients randomized to rucaparib or physician's choice of abiraterone acetate or enzalutamide (whichever the patient has not yet received) or cross-over to rucaparib <u>before</u> initiation of treatment on Study Day 1. Procedures

required on Study Day 1/ Cross-over Study Day 1 may be omitted if completed  $\leq$  3 days earlier during the Screening Phase.

- PRO collected using the BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments; complete before other procedures
- Physical examination, including weight
- Vital Signs
- Concomitant medications and procedures
- PSA measurement
- ECOG performance status
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- Plasma sample for ctDNA (required on Study Day 1 even if collected at any time during the Pre-Screening or Screening Phase)
- Blood sample for pharmacogenomic analysis (not required for patients crossing over to rucaparib)
- AE (inclusive of SAE and AESI) monitoring
- Study drug dispensation (rucaparib, abiraterone acetate, enzalutamide). Enough study drug will be dispensed to patient in sufficient quantity to last until the next study drug dispensation visit.

Site personnel will account for study drug that is administered or dispensed to the patient during the study visit and document appropriately.

## 9.5.1.2 Study Day 15 (Week 3) and Cross-over Day 15 (XO-Week 3)

The following procedures will be completed:

- Physical examination, including weight
- Vital signs
- Concomitant medications and procedures
- ECOG performance status
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- AE (inclusive of SAE and AESI) monitoring

Patients will keep all unused containers (empty, partially used, and/or unopened) and return with them to the study site for accountability/compliance review at the next visit. In the event of toxicities, re-treatment or dose modification will be according to the criteria described in Sections 7.5.1.1 and 7.5.5.

## 9.5.1.3 Study Day 29 (Week 5) and Cross-over Day 29 (XO-Week 5)

Patients randomized to rucaparib will be instructed to refrain from taking their first dose of rucaparib at home on the day of their visit to collect plasma samples for PK. Cross-over patients will not have plasma samples for PK collected.

Plasma samples for PK analysis should be collected before the morning dose as close to 12 hours after the previous dose as possible. If the start of the next dose is delayed, the PK sample should still be collected during this visit instead of the delayed start of the next treatment cycle.

The following procedures will be completed:

- PRO collected using the BPI-SF, analgesic drug score, FACT-P, EQ-5D-5L instruments; complete before other procedures
- Physical examination, including weight
- Vital signs
- Concomitant medications and procedures
- ECOG performance status
- PSA measurement
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- Plasma sample for PK analyses (patients initially randomized to rucaparib only, PK is not required for patients who cross-over to rucaparib)
- AE (inclusive of SAE and AESI) monitoring
- Study drug dispensation (rucaparib, abiraterone acetate, enzalutamide). Enough study drug will be dispensed to patient in sufficient quantity to last until the next study drug dispensation visit.

Patients will keep all unused containers (empty, partially used, and/or unopened) and return with them to the study site for accountability/compliance review at the next visit. In the event of toxicities, re-treatment or dose modification will be according to the criteria described in Sections 7.5.1.1 and 7.5.5.

## 9.5.1.4 Study Day 43 (Week 7) and Cross-over Study Day 43 (XO-Week 7)

The following procedures will be completed:

- Physical examination, including weight
- Vital signs
- Concomitant medications and procedures
- ECOG performance status
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)

- AE (inclusive of SAE and AESI) monitoring
- 9.5.1.5 Study Day 57 (Week 9) and Cross-over Day 57 (XO-Week 9), and Every 28 Days Thereafter

Patients randomized to rucaparib will be instructed to refrain from taking their first dose of rucaparib at home on the day of their visit to collect plasma samples for PK. Cross-over rucaparib patients will not collect PK samples.

Plasma samples for PK analysis should be collected before the morning dose on Study Day 57, Study Day 85, and Study Day 113 as close to 12 hours after the previous dose as possible. If the start of the next dose is delayed, the PK sample should still be collected during this visit instead of the delayed start of the next dose.

The following procedures will be completed:

- PRO collected using the BPI-SF, analgesic drug score, FACT-P, EQ-5D-5L instruments; complete before other procedures
- Physical examination, including weight
- Vital signs
- Tumor assessment scans at the end of every 8 calendar weeks ( $\pm$  7 days) for the first 24 weeks (Weeks 9, 17, 25), and then every 12 calendar weeks ( $\pm$  7 days) thereafter (Weeks 37, 49, 61, etc.)
- Concomitant medications and procedures
- ECOG performance status
- PSA measurement
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- Plasma sample for PK analyses (patients initially randomized to rucaparib only, PK is not required for patients who cross-over to rucaparib)
- AE (inclusive of SAE and AESI) monitoring
- Study drug dispensation (rucaparib, abiraterone acetate, enzalutamide). Enough study drug will be dispensed to patient in sufficient quantity to last until the next study drug dispensation visit.

Patients will keep all unused containers (empty, partially used, and/or unopened) and return with them to the study site for accountability/compliance review at the next visit. In the event of toxicities, re-treatment or dose modification will be according to the criteria described in Sections 7.5.1.1 and 7.5.5.

## 9.5.2 Patients Randomized to Physician's Choice of Docetaxel

## 9.5.2.1 Study Day 1 (Week 1) and Every 21 Days Thereafter

The following procedures/assessments will be completed for patients randomized to physician's choice of docetaxel <u>before</u> initiation of treatment on Study Day 1. Procedures required on Study Day 1 may be omitted if completed  $\leq$  3 days earlier during the Screening Phase.

- Physical examination, including weight
- Vital Signs
- Concomitant medications and procedures
- PSA measurement
- ECOG performance status
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- AE (inclusive of SAE and AESI) monitoring
- Docetaxel administration
  - Docetaxel administration will continue up to a maximum of 10 cycles (whereupon no study treatment shall be given, but assessments continue).

## 9.5.2.2 Study Day 1 (Week 1)

- Plasma sample for ctDNA (required on Study Day 1 even if collected at any time during the Pre-Screening or Screening Phase)
- Blood sample for pharmacogenomic analysis

## 9.5.2.3 Study Day 1 (Week 1) and Every 28 Days Thereafter

- PRO collected using the BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments; complete before other procedures (every 28 days ±7 days)
- AE (inclusive of SAE, and AESI) monitoring

## 9.5.2.4 Study Day 57 (Week 9) and Every 56 Days Thereafter

• Tumor assessment scans at the end of every 8 calendar weeks (± 7 days) for the first 24 weeks (Weeks 9, 17, 25), and then every 12 calendar weeks (± 7 days) thereafter (Weeks 37, 49, 61, etc.)

# 9.6 Post-treatment Phase (Randomized Treatment/ Cross-over to Rucaparib)

## 9.6.1 Treatment Discontinuation Visit

Upon randomized treatment discontinuation, regardless of the reason, patients will have a Treatment Discontinuation Visit.

However, patients with radiographic disease progression by modified RECIST Version 1.1 and/or PCWG3 criteria (for bone lesions), as assessed by IRR, but still receiving benefit per the investigator, may be considered for treatment continuation. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator, including to assess for consideration to continue treatment; scans will no longer be submitted to or read by IRR. The sponsor will inform investigators when submission of scans for IRR should discontinue. These patients will continue cycles of study drug as described starting in Sections 9.5.1.5 and 9.5.2.3, and a Treatment Discontinuation Visit as described below will occur at the end of all study treatment. In such cases, the patient must consent prior to continuing treatment with study drug.

Patients who continue treatment on study drug after radiographic disease progression will have the option of tumor tissue biopsy collection at time of first disease progression on study (requires additional consent). Tumor tissue will be processed locally as formalin-fixed paraffin-embedded (FFPE) tissue. Refer to the Pathology Charter for detailed sample handling instructions. Patients on comparator arms may be evaluated for eligibility to cross-over to treatment as described in Sections 6.4 and 9.8.

Patients who cross-over to rucaparib will complete a Treatment Discontinuation Visit after discontinuation of comparator therapy, and will then complete a second Treatment Discontinuation Visit after discontinuation of rucaparib.

The following procedures will be performed when treatment to which the patient is randomized and/or cross-over to rucaparib has been completed or is discontinued:

- PRO collected using the BPI-SF, analgesic drug score, FACT-P, and EQ-5D-5L instruments; complete before other procedures
- Physical examination, including weight
- Vital Signs
- 12-lead ECG
- Tumor assessment if it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since the last assessment and the reason for treatment discontinuation was other than disease progression confirmed by IRR for the randomized Treatment Phase and by investigator assessment for the Cross-over Phase. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR.

- Concomitant medications and procedures
- ECOG performance status
- PSA measurement
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)
- Plasma sample for ctDNA
- AE (inclusive of SAE, and AESI) monitoring
- Optional tumor tissue biopsy collection from the time of disease progression (radiographic or clinical) / randomized treatment discontinuation and prior to the initiation of any subsequent anticancer therapy (requires additional consent). Tumor tissue will be processed locally as FFPE tissue. Refer to Section 9.13 for more information and to the Pathology Charter for detailed sample handling instructions.

# 9.6.2 28-day Safety Follow-up Visit (Randomized Treatment/ Cross-over to Rucaparib)

The following procedures will be performed for all patients at  $28 (\pm 3)$  days after the last dose of randomized study drug and/or cross-over to rucaparib.

Patients initially randomized to rucaparib and patients who cross-over to receive rucaparib after comparator therapy will have a safety follow-up visit  $28 (\pm 3)$  days after the last dose of rucaparib and continue with long-term follow-up. (Section 9.6.3).

Patients randomized to comparator therapy who do not cross-over to receive rucaparib will have a safety follow up visit  $28 (\pm 3)$  days after the last dose of comparator and continue with long-term follow-up (Section 9.6.3).

- PRO collected using the BPI-SF, analgesic pain score, FACT-P, and EQ-5D-5L instruments; complete before other procedures
- Physical examination, including weight
- Vital Signs
- Tumor assessment only if it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since the last assessment for those patients that have not had radiographic progression (by central assessment for the randomized Treatment Phase and by investigator assessment for the Cross-over Phase). Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR.
- Concomitant medications and procedures
- ECOG performance status
- Clinical laboratory assessments (hematology, serum chemistry [fasting is <u>not</u> required], urinalysis)

- AE monitoring (<u>Note</u>: all SAEs, AESIs, and treatment-related Grade 3/4 AEs are to be followed to outcome [Section 10.8] if longer than the 28-day follow-up period); and
- Information collected for subsequent treatments

Patients who do not withdraw from the study at this visit will continue with long-term follow-up as described in Section 9.6.3.

## 9.6.3 Long-term Follow-up (Randomized Treatment/ Cross-over to Rucaparib)

Patients randomized to rucaparib who complete a safety follow-up visit  $28 \pm 3$  days after the last dose of rucaparib will continue in long-term follow-up as described below.

Patients randomized to comparator therapy who discontinue treatment due to radiographic disease progression and are ineligible or do not consent to cross-over to rucaparib treatment will continue in long-term follow-up as described below, after a safety follow-up visit.

Patients randomized to comparator therapy who discontinue treatment before radiographic disease progression and complete a safety follow-up visit  $28 \pm 3$  days after the last dose of randomized chemotherapy will continue in long-term follow-up as described below. At the time of radiographic disease progression, the patient may be eligible and consent to cross-over to treatment with rucaparib. The patient may also be ineligible or not consent to cross-over to rucaparib treatment and will continue in long-term follow-up.

Patients who cross-over to rucaparib treatment will follow the procedures beginning in Section 9.7. These patients will have appropriate follow-up visits after discontinuation of cross-over rucaparib treatment.

Patients in long-term follow-up will undergo the following assessments:

- If applicable, tumor assessment (using the same methodology as was used at initial study screening [eg, CT and bone scan]) when the reason for treatment discontinuation was other than death or disease progression based on radiographic assessment and it has been ≥ 8 weeks (≥ 12 weeks if previous scan was after 24 weeks on study) since last scan or disease progression was noted on the last scan. Tumor assessment should continue to be performed at the end of every 8 calendar weeks (±7 days) relative to Study Day 1 (Week 1) up to 24 weeks, then every 12 calendar weeks (±7 days), until confirmed radiographic disease progression by modified RECIST Version 1.1 and/or PCWG3 (for bone lesions only) criteria, as assessed by IRR for the randomized Treatment Phase, until analysis of the primary endpoint has been performed, and by investigator assessment for the Cross-over Phase, loss to follow-up, withdrawal, or study closure. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or read by IRR.
  - PRO assessments will also continue and coincide on days when tumor assessments are performed until confirmed radiographic disease progression for the randomized Treatment Phase or the Cross-over Phase. PRO using the BPI-SF (Appendix 5), FACT-P

(Appendix 6), EQ-5D-5L instruments (Appendix 7), and analgesic drug score (Appendix 8).

- All patients discontinued from treatment, regardless of reason, will be followed and information collected for subsequent treatments and survival every 12 weeks (± 14 days) from last dose of study drug until death, loss to follow-up, withdrawal of consent from study, or closure of the study. Follow-up can be performed via the telephone and can be completed to coincide with scheduled tumor assessments and/or PRO during this period.
- SAEs related to study drug and AESIs are to be reported as specified in Section 10.7.

# 9.7 Informed Consent for Patients Who Cross-over to Rucaparib after Disease Progression on Comparator Treatment

Patients who initially received comparator treatment and then cross-over to treatment with rucaparib after radiographic disease progression is confirmed by IRR (after the analysis of the primary endpoint is performed, this will change to investigator-assessed radiographic progression, as IRR will be discontinued) must provide additional consent to receive rucaparib treatment, as well as sponsor (or designee) approval. Patients who are eligible to cross-over as described in Section 6.4 and receive approval should receive the first dose of rucaparib within 28-days following the scan date resulting in confirmation of radiographic progression. Ineligible patients will continue with a 28-day Safety Follow-up Visit and long-term follow-up as in Sections 9.6.2 and 9.6.3.

Additionally, patients participating in the optional tumor tissue biopsy at the time of radiographic disease progression/treatment discontinuation after cross-over to rucaparib must provide additional consent for this procedure.

# 9.8 Screening Prior to Cross-over to Rucaparib

Following written informed consent, and unless otherwise specified, the screening assessments equivalent to 28 days before study start through 14 days before study start (Section 9.4.1) will be performed prior to initiating treatment with rucaparib within the allowable windows of time as indicated. Assessments performed within the specified windows, but prior to patient signing informed consent, are acceptable only if confirmed to have been standard of care. Assessments performed at treatment discontinuation and/or at the 28-day Safety Follow-up Visit following discontinuation of comparator therapy may be utilized, provided they were within the allowable windows of time as indicated.

Screening procedures may be repeated if the findings/results are considered invalid or not representative of the patient's baseline medical status. When screening procedures are repeated, the rationale should be documented in the source file.

## 9.8.1 Ongoing Assessments for Cross-over Patients:

Patients will continue with all assessments required from and including XO-Study Day 1 of the first dose of rucaparib through to 28-day follow-up after study drug is stopped per schedule of assessments, as described in Sections 9.5.1.1 to 9.5.1.5 and Sections 9.6.1 and 9.6.2 of this protocol. Radiographic assessments performed during the Cross-over Phase will not be submitted

for IRR. As described in Section 9.6.3, these patients will have appropriate follow-up visits after discontinuation of cross-over rucaparib treatment.

## 9.9 Methods of Data Collection

## 9.9.1 Medical History and Demographic/ Baseline Characteristics

Basic demographic and baseline characteristics will be collected during screening. In addition to the evaluation of a patient's medical history in terms of study eligibility, all relevant medical conditions will be documented in the appropriate eCRF. Events that occur after signing of informed consent but prior to initiation of study drug, unless an SAE and due to a protocol-mandated procedure, should be recorded in the Medical History eCRF.

The patient's entire oncology history will be collected in the appropriate eCRF including date of diagnosis for mCRPC (and other malignancy, if applicable), prior surgeries/ treatments received for cancer, dates of treatment administration, best response achieved, date of progression and how assessed, and BRCA1/BRCA2/ATM/other HRR gene mutation status (if known).

## 9.10 Prior and Concomitant Medication/ Procedure Assessments

Medications being used by the patient and surgical/ medical procedures experienced by the patient will be recorded as prior/ concomitant medications/ procedures during screening and as concomitant medications/ procedures following receipt of the first dose of study drug through the completion of the 28-day Safety Follow-up Visit after discontinuation of randomized treatment or cross-over treatment discontinuation if the patient crosses over. Medication information will be entered in the appropriate eCRF after it is obtained at each study visit.

# 9.11 Efficacy Evaluations

## 9.11.1 Disease/ Tumor Assessments

Radiographic tumor assessments including CT scans of the chest, abdomen & pelvis (and other anatomical regions as indicated) that are contrast-enhanced and have < 5 mm slice thickness, as well as skeletal scintigraphy (whole body) using 99mTc-MDP or HDP. MRI or non-contrast CT may be utilized for patients intolerant to contrast. Where indicated for neurological symptoms, MRI of the spine and skull should be performed. Other studies, such as PET, may also be performed. If a site can document that the CT performed as part of a PET/CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast) then the CT portion of the PET/CT can be used for RECIST Version 1.1 measurements. Disease assessment by CT/MRI and bone scans will be performed during screening, every 8 calendar weeks ( $\pm$  7 days) from Study Day 1 up to 24 weeks and then every 12 calendar weeks (± 7 days) thereafter. If study drug was discontinued for reasons other than radiographic disease progression confirmed by IRR, tumor assessments (using the same methodology as was used at initial study screening [eg, CT scan]) will continue until radiographic disease progression is confirmed by IRR. Once the analysis of the primary endpoint has been performed, radiographic scans will continue to be performed by the investigator as per the protocol schedule of assessments until radiographic disease progression is determined by the investigator; scans will no longer be submitted to or

read by IRR. The sponsor will inform investigators when submission of scans for IRR should discontinue. If a CR or PR is noted, confirmatory scans should be performed at least 4 weeks after the initial response was first documented. Modified RECIST Version 1.1/PCWG3 criteria will be used (Appendix 1); up to five lesions in any metastatic site shall be recorded for extra-skeletal disease according to PCWG3. Criteria for progressive disease (PD) and confirmation thereof are summarized in Table 8.

Copies of all radiographic scans during the Treatment Phase, including baseline scans and any scans collected in follow-up after the Treatment Phase, must be submitted for IRR. After the primary endpoint analysis is performed, confirmation of radiographic progression by IRR will no longer occur; radiographic progression and confirmation of disease progression will be performed by the investigator, including to assess eligibility for cross-over or consideration to continue treatment. Scans collected during the Cross-over Phase will not be submitted for IRR.

Table 8. Requirements for Confirmation of Radiographic Disease Progression in Bone per Investigator's Assessment

| Date Progression<br>Detected (Visit) | Criteria for Initial<br>Progression | Timing for Confirmation of Progression | Criteria for Documentation of Disease Progression on Confirmatory Scan |
|---|---|---|---|
| Week 9<br>(1 <sup>st</sup> on-treatment<br>scan) | Bone lesions: Two or more new lesions compared to <b>baseline</b> bone scan by PCWG3 | At least 6 weeks after progression identified or at Week 17 Visit | Two or more new lesions identified at Week 9 must persist at Week 17 and two or more additional new lesions must be identified on Week 17 bone scan (compared to Week 9 scan). |
| Week 17<br>(2 <sup>nd</sup> on-treatment<br>scan) | Bone lesions: Two or more new lesions on bone scan compared to Week 9 bone scan | At least 6 weeks after progression identified or at Week 25 Visit | Two or more new lesions identified at Week 17 must persist at Week 25 bone scan. |
| Week 25 or later (3 <sup>rd</sup> on-treatment scan and after) | Bone lesions: Two or more<br>new lesions compared to<br>Week 9 bone scan | At least 6 weeks after progression identified or at next regularly scheduled radiographic assessment | Two or more new lesions identified at Week 25 (or later) bone scan must persist at scan obtained 6 weeks later. |

Abbreviation: PCWG3 = Prostate Cancer Working Group Guidelines Version 3.

# 9.12 Safety Evaluations

#### 9.12.1 Adverse Event Assessment

The investigator has the responsibility for assessing the safety of the patients and for compliance with the protocol to ensure study integrity. During the Pre-Screening Phase and Screening Phase,

unless otherwise required by local regulations, SAEs which are related to protocol-mandated assessments will be reported. Once enrolled to study drug, patients will be monitored for all AEs/SAEs/AESIs during study participation and until 28 days after the last dose of study drug. Any ongoing SAEs, AESIs, or treatment-related Grade 3/4 AEs will be followed until resolution or stabilization. After the 28-day window, only SAEs assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

After the 28-day Follow-up Visit, **AESIs of MDS and AML**, **irrespective of causality, should be reported** per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

• AESIs of pneumonitis or similar events (ie, interstitial lung disease, pulmonary fibrosis, acute interstitial pneumonitis, alveolitis necrotizing, alveolitis, hypersensitivity pneumonitis, and organizing pneumonia) should be reported up to, but not beyond, the 28-Day Follow-up Visit (28-days after the last dose of rucaparib). After the 28-day Follow-up Visit, only pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements.

AEs and laboratory abnormalities will be graded according to the NCI CTCAE grading system (Version 4.03 or higher) and recorded in the eCRF.

Complete details for monitoring AEs (inclusive of SAEs and AESIs), including the definition of drug-related AEs, are provided in Section 10.

## 9.12.2 Clinical Laboratory Investigations

Samples for hematology, serum chemistry, and urinalysis will be analyzed by a local laboratory. The panels of laboratory tests to be performed are shown below:

**Hematology:** red blood cells (RBC) and parameters (hemoglobin, hematocrit, mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], and mean corpuscular hemoglobin concentration [MCHC]) and reticulocyte count, white blood cells (WBC) and differential (with ANC), and platelet count will be assessed at screening, during treatment at study visits, and at the Treatment Discontinuation and 28-day Follow-up Visits (including those for cross-over) for all patients. Hematology results must be reviewed by the investigator before the start of treatment with study drug and ongoing at times testing occurs. Additional and more frequent tests may be performed at the investigator's discretion.

Serum Chemistry: total protein, albumin, creatinine for estimating GFR using the Cockcroft-Gault formula (Appendix 3), BUN or urea, total bilirubin, alkaline phosphatase (ALP), ALT, AST, lactate dehydrogenase (LDH), glucose, sodium, potassium, chloride, CO<sub>2</sub>, calcium, phosphorus, and lipid panel (total cholesterol, low density lipoprotein [LDL], high density lipoprotein [HDL], and triglycerides), at screening, during treatment at study visits, and at the Treatment Discontinuation and 28-day Follow-up Visits (including those for cross-over) for all patients. Fasting is not required before blood sampling. Serum chemistry results must be reviewed by the investigator before the start of treatment with study drug and ongoing at times

testing occurs. Additional and more frequent tests may be performed at the investigator's discretion.

**Urinalysis:** performed locally on a freshly voided clean sample by dipstick for protein, glucose, blood, pH, and ketones. If dipstick findings are abnormal based on the investigator's judgment, then a microscopic evaluation will be performed to assess the abnormal findings. Urinalysis will be performed at screening, during treatment at study visits, and at the Treatment Discontinuation and 28-day Follow-up Visits (including those for cross-over) for all patients, but may be conducted at other times as clinically indicated.

Laboratory reports will be reviewed by the investigator or delegated physician who will then comment on out-of-range parameters and assess clinical significance. Clinically significant abnormalities and associated panel results will be documented in the eCRF as an AE; any results of unscheduled tests will also be recorded in the eCRF. Refer to Section 10.5 for guidelines on reporting of abnormal laboratory values as AEs.

## 9.12.3 Vital Signs

Vital signs will include blood pressure, pulse, and body temperature and will be taken after the patient has been resting for at least 5 minutes during screening, at study visits during the Treatment Phase, and at the Treatment Discontinuation and 28-day Follow-up Visits (including those for cross-over).

## 9.12.4 12-lead Electrocardiogram

For all patients, 12-lead ECGs will be performed at the following times:

- Screening (within 28 days prior to randomization)
- Treatment Discontinuation Visit

The following will be measured or calculated: heart rate, pulse rate, QRS, QT, QTc, and rhythm. The investigator or qualified designee will review the ECGs locally and assess the results as normal or abnormal (clinically significant or not clinically significant).

If it is clinically indicated, ECGs can be performed at other times during the study.

# 9.12.5 Physical Examinations, Body Weight and Height

Physical examinations will include an assessment of all the major body systems. Complete physical examinations will be performed during screening and at the Treatment Discontinuation Visit. Physical examinations at study visits during the Treatment Phase and 28-day Follow-up Visit (including cross-over) will be limited as appropriate.

Height will be measured during the screening visit only. Weight will be measured per institutional guidelines during screening, at study visits prior to therapy administration, and at the Treatment Discontinuation and 28-day Follow-up Visits (including those for cross-over).

## 9.12.6 ECOG Performance Status

ECOG performance status (Appendix 2) will be assessed during screening, at study visits during the Treatment Phase, and at the Treatment Discontinuation and 28-day Follow-up Visits (including cross-over). The ECOG performance status should be assessed by the same study personnel at each visit, if possible. For eligibility purposes, patients with borderline ECOG performance status should be considered carefully to avoid enrolling patients who may have significant impairment.

## 9.13 Biomarker Analysis – FFPE Tumor Tissue

An optional tumor biopsy obtained between the time of disease progression/randomized treatment discontinuation and the start of the next treatment will be obtained from consenting patients. The molecular profile of the progression biopsy will be compared with that from matched pretreatment primary or metastatic tumor tissue to identify mechanisms of resistance to rucaparib. Patients must provide additional consent for the optional tumor tissue biopsy sample. New lesions or lesions that are growing should be prioritized for the optional biopsy. If possible, collect the lesion responsible for progression. Detailed sample handling instructions are located in the Pathology Charter.

# 9.14 Biomarker Analysis – ctDNA/genomic DNA from Blood

Blood samples will be collected during Pre-Screening (for deleterious BRCA1/2 or ATM gene mutation assessment), Screening, before dosing on Study Day 1 and at treatment discontinuation from all patients entered in the study for plasma ctDNA analysis.

Blood will be collected for pharmacogenomics analyses on Study Day 1 from all patients; this sample is not collected on Cross-over Study Day 1. Genomic DNA will be extracted from the cellular portion of this blood sample and may be analyzed to determine whether the deleterious BRCA1, BRCA2 or ATM gene mutation identified is germline or somatic prior to final data analysis. Because the germline analysis will be done near the end of the study, there are no plans to share these results with the investigator. However, if an actionable mutation, as defined by the American College of Medical Genetics and Genomics

(https://www.ncbi.nlm.nih.gov/clinvar/docs/acmg/), is revealed that was not detected in tumor or plasma, these incidental findings will be made available to the investigator provided the results are generated from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. Sample collection details will be provided in a Laboratory Manual.

## 9.15 Pharmacokinetics Evaluation

For patients receiving rucaparib (except those in the Cross-over Phase), plasma samples are to be collected for trough level PK analysis of rucaparib before the morning dose on Study Day 29, Day 57, Day 85, and Day 113 as close to 12 hours after the previous dose as possible. If the start of the next dose is delayed, the PK sample should still be collected during this visit instead of on the delayed start of the next dose. Samples are not to be collected in patients receiving comparator therapy or crossing over to rucaparib. Refer to the Laboratory Manual for sample collection details for PK samples.

# 9.16 Patient-reported Outcomes (Health and Quality of Life Questionnaires)

Patient-reported outcomes utilizing the BPI-SF (Appendix 5), FACT-P (Appendix 6), EQ-5D-5L (Appendix 7), and analgesic drug score (Appendix 8) instruments will be assessed during screening, at study treatment visits during the Treatment Phase, the Treatment Discontinuation Visit, and at the 28-day Safety Follow-up Visit. The analgesic drug score will be recorded according to the World Health Organization's (WHO's) analgesic ladder: 0 for no analgesic, 1 for non-opioids, 2 for opioids for moderate pain, and 3 for opioids for severe pain. <sup>47</sup> Patients must complete the instruments before any other scheduled study procedures are performed and dosing occurs (if applicable).

PRO assessments should be collected at every study visit for all patients through disease progression in association with the radiographic assessments for disease progression. For patients who discontinue treatment prior to radiologic disease progression, PRO assessments should be collected until confirmed radiologic disease progression is documented.

## 10 ADVERSE EVENT MANAGEMENT

## 10.1 Definition of an Adverse Event

An AE is defined as any untoward medical occurrence in a patient administered a medicinal product that does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational medicinal product. This includes an exacerbation of pre-existing conditions or events, intercurrent illnesses, or drug interaction that is not recorded elsewhere in the eCRF under specific efficacy assessments. Anticipated fluctuations of pre-existing conditions, including the disease under study, that do not represent a clinically significant exacerbation or worsening are not considered AEs.

It is the responsibility of the investigator to monitor all AEs that occur during the study. AEs should be elicited by asking the patient a non-leading question (eg, "Have you experienced any new or changed symptoms since we last asked/since your last visit?"). The existence of an AE may be concluded from a spontaneous report of the patient; from the physical examination; or from special tests such as the ECG, laboratory assessments, or other study-specified procedure (source of AE). Symptoms reported spontaneously by the patient during the physical examination would also qualify as an AE (and hence documented in the AE eCRF, not in the physical examination eCRF, which is reserved for physical signs or findings).

## 10.2 Definition of a Serious Adverse Event

An SAE is any untoward medical occurrence that occurs at any dose (including after informed consent is given and prior to dosing if the SAE is related to a study procedure) that:

• Results in death. Any event resulting in death during the reporting period (from date of first dose of investigational product through 28 days after last dose) must be treated as an SAE

and reported as such. An event related to a study procedure that occurs after informed consent, but prior to dosing, that results in death must also be reported as an SAE. This excludes death due to progression of patient's underlying cancer. (refer Section 10.4)

- Is life-threatening (patient is at <u>immediate</u> risk of death from the event as it occurred)
- Requires in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Results in a congenital anomaly or birth defect
- <u>Important medical events</u> that may not result in death, are not life-threatening, or do not require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such events include allergic bronchospasm requiring intensive treatment in an emergency room or at home or the development of drug dependency or drug abuse.

## 10.3 Definition of an Adverse Event of Special Interest

AESIs (serious or nonserious) are defined as AEs of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the study sponsor to other parties (eg, regulators) might also be warranted.

Details on the sponsor's currently agreed list of AESIs for rucaparib can be found in the current rucaparib IB. These AESIs are to be reported to the sponsor **within 24** hours of knowledge of the event (see Section 10.7 for reporting instructions).

# 10.4 Events or Outcomes Not Qualifying as Serious Adverse Events

The following are not considered SAEs for the purposes of this protocol, and therefore do not need to be reported as such:

- Preplanned or elective hospitalization including social and/ or convenience situations (eg, respite care)
- Hospital visits of less than 24 hours duration (eg, patient presents to the emergency room, but is not admitted to a ward)
- Overdose of study drug or concomitant medication unless associated with an SAE. However, the event should still be captured as a nonserious AE in the appropriate eCRF page
- Events of progression of the patient's underlying cancer as well as events clearly related to progression of the patient's cancer (signs and symptoms of progression) and progression of disease leading to death should not be reported as an AE or SAE. This section excludes other SAEs with fatal outcome

 Events that meet the SAE criteria (as outlined in Section 10.2) and occur after informed consent but before the first dose of study drug, which are considered unrelated to protocolmandated procedures

# 10.5 Clinical Laboratory Assessments as Adverse Events and Serious Adverse Events

It is the responsibility of the investigator to assess the clinical significance of all abnormal values as defined by the list of reference ranges from the local laboratory. In some cases, significant changes in lab values within the normal range will require similar judgment.

An abnormal laboratory value that is not already associated with an AE is to be recorded as an AE only if any one of the following criteria is met:

- an action on the study drug is made as a result of the abnormality
- intervention for management of the abnormality is required
- at the discretion of the investigator should the abnormality be deemed clinically significant

## 10.6 Pregnancy or Drug Exposure During Pregnancy

A pregnancy is not considered to be an AE or SAE; however, any pregnancy occurring in a partner of a study patient during study participation or within 3 months of last dosing must be reported to the sponsor using the Pregnancy Report Form within the same timelines as an SAE.

A pregnancy will be followed through to outcome. Once the outcome of the pregnancy is known, the Pregnancy Outcome Report Form is to be completed and reported to the Sponsor.

AEs, SAEs, or AESIs that occur during pregnancy will be assessed and processed according to the AE or SAE/AESI processes using the appropriate AE or SAE/AESI forms.

# 10.7 Recording of Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest

Events that occur after signing of informed consent but prior to initiation of study drug, unless due to a protocol-mandated procedure, are to be recorded in the Medical History eCRF; however, events are to be reported as SAEs if serious and related to a protocol-mandated procedure during the Pre-Screening Phase or Screening Phase.

Any AE that occurs after first dose of study drug through 28 days after receiving the last dose of study drug will be recorded in the AE eCRF.

After the 28-day Follow-up Visit, only SAEs assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

After the 28-day Follow-up Visit, **AESIs of MDS and AML**, **irrespective of causality, should be reported** per Clovis Oncology PV requirements and captured in the Clovis Oncology PV database.

• AESIs of pneumonitis or similar events (ie, interstitial lung disease, pulmonary fibrosis, acute interstitial pneumonitis, alveolitis necrotizing, alveolitis, hypersensitivity pneumonitis, and organizing pneumonia) should be reported up to, but not beyond, the 28-day Follow-up Visit (ie, 28-days after the last dose of rucaparib). After the 28-day Follow-up Visit, only pneumonitis or similar events meeting the criteria for an SAE and assessed as potentially related to study drug should be reported per Clovis Oncology PV requirements.

Information on the follow-up of AEs, SAEs, and AESIs is provided in Section 10.8.

In order to avoid vague, ambiguous, or colloquial expressions, the AE should be recorded in standard medical terminology rather than the patient's own words. Whenever possible, the investigator should combine signs and symptoms that constitute a single disease entity or syndrome into a final diagnosis, if appropriate. For example, fever, cough, and shortness of breath may be reported as pneumonia, if that is a reasonable diagnosis.

Each AE is to be evaluated for causal relationship to the investigational drug, severity, and seriousness. The action taken and the outcome must also be recorded.

SAEs and AESIs that occur during the study or within 28 days after receiving the last dose of study drug, whether or not related to study drug, must be reported immediately (ie, **within 24 hours** of knowledge of the event or additional information for a previously-reported event) to the sponsor/ SAE designee. The contact information for reporting of SAEs/ AESIs can be found on the SAE/ AESI Reporting Form.

## 10.7.1 Onset Date of Adverse Events

The onset date is the date that the event or the signs/symptoms attributed to the event started.

## 10.7.2 Resolution Date of Adverse Events

The resolution date is the date that the event or the signs/symptoms attributed to the event resolved or resolved with sequelae or it is the date when the patient has reached a new baseline if the event is not expected to resolve.

## 10.7.3 Intensity of Adverse Events

The severity of each AE will be graded using the NCI CTCAE, Version 4.03 or higher grading scale. 48

Severity is not the same as Serious.

For AEs not covered by NCI CTCAE, the severity will be characterized as mild, moderate, severe, life-threatening, or fatal according to the following definitions:

- Mild events are usually asymptomatic or have mild symptoms with clinical or diagnostic observations only; intervention is not indicated
- Moderate events introduce a low level of inconvenience or concern to the patient, local or noninvasive intervention may be indicated, and may interfere with age-appropriate daily activities
- Severe events are medically significant, but not immediately life-threatening; interrupt the patient's usual self-care daily activities, disabling, and hospitalization (or prolongation of hospitalization) is indicated
- Life-threatening events require urgent intervention to prevent death; or
- Fatal events are those events that lead to the patient's death

## 10.7.4 Causal Relationship of Adverse Events to Study Drug

Medical judgment should be used to determine the cause of the AE considering all relevant factors such as, but not limited to, the underlying study indication, coexisting disease, concomitant medication, relevant history, pattern of the AE, temporal relationship to the study medication, and dechallenge or rechallenge with the study drug.

| Not Related to<br>Study Drug | An AE that is clearly due to extraneous causes (eg, concurrent disease, concomitant medications, disease under study, etc.) |
|---|---|
| | • It does not follow a reasonable temporal sequence from administration of the study drug |
| | It does not follow a known pattern of response to study drug |
| | • It does not reappear or worsen when study drug is restarted, or |
| | An alternative explanation is likely, but not clearly identifiable. |
| Related to | An AE that is difficult to assign to alternative causes. |
| Study Drug | It follows a strong or reasonable temporal sequence from administration of study drug |
| | • It could not be reasonably explained by the patient's clinical state, concurrent disease, or other concomitant therapy administered to the patient |
| | It follows a known response pattern to study drug, or |
| | It is confirmed with a positive rechallenge or supporting laboratory data. |

## 10.7.5 Outcome and Action Taken

The investigator will record the action taken and outcome for each AE according to the following criteria:

## Action Taken With Study Drug (check all that apply)

- Dose not changed
- Dose reduced
- Study drug interrupted
- Study drug withdrawn
- Not applicable
- Other action taken (check all that apply)
  - None
  - Procedure intervention
  - Concomitant medication taken
  - Transfusion given
  - Hospitalization
  - Other, (specify)

#### **Outcome**

- Recovered/Resolved
- Recovered/Resolved with sequelae
- Recovering/Resolving
- Not Recovered/Resolved
- Fatal
- Unknown

# 10.8 Follow-up of Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest

All AEs (including SAEs and AESIs) occurring during the study are to be followed up in accordance with good medical practice until resolved; judged no longer clinically significant; or, if a chronic condition, until fully characterized through 28 days after the last dose of study drug. Any SAEs, AESIs, and treatment-related Grade 3/4 AEs must be followed until resolution or stabilization, death, or until lost to follow-up. After the 28-day window, only SAEs assessed as potentially related to study drug, and **AESIs of MDS and AML**, **irrespective of causality**, **should be reported**.

• AESIs of pneumonitis or similar events (ie, interstitial lung disease, pulmonary fibrosis, acute interstitial pneumonitis, alveolitis necrotizing, alveolitis, hypersensitivity pneumonitis, and organizing pneumonia) should be reported up to, <u>but not beyond</u>, the 28-day Follow-up Visit (ie, 28-days after the last dose of rucaparib). After the 28-day Follow-up Visit, <u>only</u> pneumonitis or similar events **meeting the criteria for an SAE and assessed as potentially related to study drug** should be reported per Clovis Oncology PV requirements.

# 10.9 Potential Drug-induced Liver Injury

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event. All occurrences of potential DILIs, meeting the defined criteria (see Section 7.5.1.1),<sup>46</sup> must be reported as SAEs (see Section 10.7 for reporting details).

# 10.10 Regulatory Aspects of Serious Adverse Event and Adverse Events of Special Interest Reporting

It is important that the investigator provide an assessment of relationship of the SAE or AESI to study treatment at the time of the initial report. For reporting SAEs/AESIs or pregnancies, use the applicable report forms. The contact information for reporting of SAEs/AESIs or pregnancies can be found on each of the forms.

The sponsor or its designee is responsible for submitting reports of AEs associated with the use of the drug that are both serious and unexpected to the US FDA, according to 21 Code of Federal Regulations (CFR) 312.32; to the European regulatory authorities according to the European Commission Clinical Trials Directive (2001/20/EC); and to other applicable regulatory authorities, according to national law and/or local regulations. All investigators participating in ongoing clinical studies with the study medication will receive copies of these reports for prompt submission to their IRB or IEC. In accordance with the European Commission Clinical Trials Directive (2001/20/EC), the sponsor or its designee will notify the relevant ethics committees in concerned member states of applicable suspected unexpected serious adverse reactions (SUSARs) as individual notifications or through periodic line listings.

The sponsor or its designee will submit all safety updates and periodic reports to the regulatory authorities as required by applicable regulatory requirements.

## 11 PLANNED STATISTICAL METHODS

## 11.1 General Considerations

All efficacy analyses will be done at a two-sided 0.05 significance level, including all data from the randomized portion of the study.

All safety analyses will be summarized for all patients who received at least one dose of protocol-specified treatment.

Quantitative variables will typically be summarized using frequencies and percentages for appropriate categorizations and may also be summarized using descriptive statistics. For variables summarized with descriptive statistics, the following will be presented: N, mean, standard deviation (StD), median, minimum, and maximum. Categorical variables will be presented using frequencies and percentages.

The Kaplan-Meier methodology will be used to summarize time-to-event variables. If estimable, the 25th, 50th (median), and 75th percentiles with the 95% CI will be summarized for each

randomized treatment group. The stratified HR from the Cox proportional hazards model will be used to estimate the HR between the randomized treatment groups for the primary endpoint.

The number of patients with events and the number of censored patients will also be presented. For stratified analyses, if one or more of the strata contain few patients (eg, < 5 patients) or only patients from a single treatment group, or if the convergence criteria in SAS are not met, strata will be combined to ensure a sufficient number of patients in each stratum by first removing the hepatic metastases variable (which is equivalent to combining the 2 categories) and then combining the BRCA1/2 categories, if necessary.

For secondary, exploratory, and subgroup analyses, statistical testing will not be stratified. Stratified analyses may be performed as sensitivity analyses. For time-to-event analyses the log-rank test will be used for treatment group comparisons.

The primary and key secondary endpoints will be tested among the patients with a deleterious BRCA1/2 mutation and the ITT Population, using an ordered step-down multiple comparisons procedure. The primary endpoint of rPFSirr in the subgroup of patients with a deleterious BRCA1/2 mutation will be tested first at a two-sided 0.05 significance level. If rPFSirr in the subgroup of patients with a deleterious BRCA1/2 mutation is statistically significant, then rPFSirr will be tested in the ITT Population (see Section 11.3). Continuing in an ordered step-down manner, the key secondary endpoints of OS and ORR (by IRR) will be tested at the two-sided 0.05 significance level. Once statistical significance is not achieved for one test, statistical significance will not be declared for all subsequent analyses in the ordered step-down procedure. See Section 11.6 for details about the ordered step-down procedure.

As a secondary endpoint of the study, trough concentrations ( $C_{min}$ ) of rucaparib will be summarized with descriptive statistics overall and by cycle in all patients with at least one PK sample collected.

Further details to describe handling of missing, unused, and spurious data will be in the Statistical Analysis Plan (SAP). Unless otherwise specified, baseline is defined as the last measurement on or prior to the first day of study drug administration or randomization date, if the patient was never treated.

All statistical analyses will be conducted with the SAS® System, Version 9.3 or higher. Further details around the statistical analyses planned in this study will be outlined in the SAP. Changes to or deviations from the SAP will be described in the clinical study report (CSR).

# 11.2 Determination of Sample Size

The total enrollment planned for this study is approximately 400 patients. A total of approximately 300 patients with a deleterious BRCA1/2 gene mutation will be randomized and approximately 100 patients with a deleterious ATM gene mutation may be randomized. This is a multicenter, multinational study. Patients will be enrolled across approximately 150 study sites worldwide.

The total enrollment planned is approximately 400 patients, with approximately 300 patients in the subgroup with a deleterious BRCA1/2 mutation and approximately 100 patients in the

subgroup with a deleterious ATM mutation. The median rPFS is assumed to be 6 months for the control arm and 10 months for rucaparib in the subgroup of patients with a deleterious BRCA1/2 mutation and 9 months for rucaparib in the total population. A sample size of approximately 300 patients in the subgroup with a deleterious BRCA1/2 mutation should result in approximately 200 events of rPFS, which will provide approximately 90% power to detect a HR of 0.6 at a one-sided 0.025 significance level. A sample size of approximately 400 total patients should result in approximately 270 events of rPFS, which will provide approximately 90% power to detect a HR of 0.67 at a one-sided 0.025 significance level.

## 11.3 Analysis Populations

The following analysis populations are defined for the study:

**Safety Population** – The safety population will consist of all patients who received at least one dose of protocol-specified treatment.

**Intent-to-Treat Population** – The ITT population will consist of all randomized patients (ie, patients with BRCA-mutated mCRPC and patients with ATM-mutated mCRPC).

**BRCA Subgroup** – The BRCA Subgroup will consist of patients in the ITT population with BRCA-mutated mCRPC.

**IRR Efficacy Population** – The IRR efficacy population will consist of all patients evaluable for response by RECIST Version 1.1/PCWG3 criteria (Appendix 1) per independent radiology review.

**Investigator Efficacy Population** – The investigator efficacy population will consist of all patients evaluable for response by RECIST Version 1.1/PCWG3 criteria (Appendix 1) per investigator.

## 11.4 Patient Disposition

Patient disposition will be summarized using frequency counts and the corresponding percentages. The number of patients in each analysis population, number of patients discontinued, and the primary reason for discontinuation will be summarized.

# 11.5 Demographics and Baseline Characteristics

All demographic (eg, age, race, and ethnicity as allowed by local regulations) and baseline characteristics will be summarized for the safety population.

The following BRCA/ATM gene mutation characteristics will also be summarized:

- BRCA1/2 or ATM gene mutation status (germline or somatic)
- HRR gene mutation (BRCA1, BRCA2, or ATM)

Descriptive statistics may also be used to summarize the continuous variables.

# 11.6 Step-down Procedure of Primary and Secondary Endpoints

The primary and key secondary endpoints will first be tested in the BRCA subgroup and then in the ITT Population (ie, BRCA + ATM) using an ordered step-down multiple comparisons procedure. The primary endpoint of rPFSirr in the BRCA subgroup will be tested first at a two-sided 0.05 significance level. If rPFSirr in the BRCA subgroup is statistically significant, then rPFSirr will be tested in the ITT Population. Continuing in an ordered step-down manner, the key secondary endpoints will be tested at the two-sided 0.05 significance level. To preserve the overall Type 1 error rate, statistical significance will only be declared for a secondary endpoint if the primary endpoints and previous secondary endpoints are also statistically significant. The ordered step-down procedure is illustrated in Figure 3.

Figure 3. Ordered Step-down Procedure

# Primary Endpoint PFSirr Secondary Endpoints OSa ORRirr ORRirr ORRirr

Abbreviations: BRCA = breast cancer gene; irr = central independent radiology review; ITT = Intent-to-treat; ORR = objective response rate; OS = overall survival; rPFSirr = radiographic progression-free survival by central independent radiology review.

As described in Section 11.7.2 and Section 11.9, OS will be analyzed at the time of the primary analysis (interim OS analysis) and again for a final OS analysis when maturity is reached. If the interim OS results are not statistically significant, p-values for all secondary endpoints will be considered descriptive until the final OS analysis has been performed as part of the step-down procedure.

## 11.7 Efficacy Analyses

## 11.7.1 Primary Efficacy Analysis

The primary efficacy endpoint for the study is rPFSirr, defined as the time from randomization to the first objective evidence of radiographic progression, or death due to any cause (whichever occurs first). Radiographic disease progression includes confirmed soft tissue disease progression and confirmed bone disease progression as per modified RECIST Version 1.1/PCWG3 criteria.

The primary endpoint of rPFSirr will be analyzed using Cox proportional hazard methodology. The stratified HR from the Cox proportional hazards model will be used to estimate the HR between the randomized treatment groups.

Assessment of rPFS by the investigator (rPFSinv) will also be conducted as a supportive analysis for rPFSirr.

## 11.7.2 Secondary Efficacy Analyses

Overall survival time will be calculated as the time from randomization to death (by any cause) +1 day. Patients who have not died will be censored on the date the patient was last known to be alive. OS will be analyzed using Cox proportional hazard methodology and a log-rank test. The HR from the Cox proportional hazards model will be used to estimate the HR between the randomized treatment groups. The log-rank test will be the official test used for the hierarchical testing outlined in Section 11.6. OS will be analyzed at the time of the primary analysis (interim OS analysis) and again for a final OS analysis when maturity is reached (see Section 11.9).

ORR is defined as the percentage of patients with a confirmed best response of CR or PR in patients with measurable disease at study entry. Modified RECIST Version 1.1 criteria will be used to determine ORR (ie, CR or PR by IRR assessment and no progression in bone per PCWG3 by IRR assessment). Per RECIST Version 1.1, to be assigned a best overall response of CR or PR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. The proportion of responders will be analyzed using a Cochran-Mantel-Haenszel (CMH) test. ORR will be analyzed separately for both IRR and investigator assessments. Only tumor scans included for the evaluation of the primary endpoint are considered for the ORR endpoint.

DOR is defined as the time from the first response (modified RECIST Version 1.1 in patients with visceral/nodal disease) until the first date that PD (using the same criteria) is documented. DOR will be summarized and analyzed for the responders using the same methodology as described for the primary endpoint. DOR will be analyzed separately for both IRR and investigator assessments.

Time to PSA progression is defined as the time from randomization to the date that a  $\geq$  25% increase and absolute increase of  $\geq$  2 ng/mL above the nadir (or baseline value for patients who did not have a decline in PSA) in PSA was measured. The increase must be confirmed by a second consecutive assessment conducted at least 3 weeks later. This endpoint will be analyzed in patients with both baseline and at least 1 post-baseline value using Cox proportional hazard

methodology. The HR from the Cox proportional hazards model will be used to estimate the HR between the randomized treatment groups.

Confirmed PSA response is defined as  $\geq 50\%$  (or  $\geq 90\%$ ) reduction in PSA from baseline on at least two assessments conducted at least 3 weeks apart. PSA response will be calculated for all patients with PSA values at baseline and at least one post-baseline assessment. PSA will be assessed by a local laboratory.

Patient-reported outcome endpoints by FACT-P and BPI-SF will be scored according to their respective scoring manuals.

Patient-reported Outcome EQ-5D-5L: Analyses of changes and/ or percent changes from baseline will be analyzed for each scheduled post-baseline visit and for the final visit for the EQ-5D-5L instrument and the EQ visual analog scale (VAS). Patients who do not have both a baseline measurement and at least one post-baseline measurement will not be included. At a given visit, the change and/or percent change from baseline will be compared between the randomized treatment groups using an analysis of covariance (ANCOVA) using the treatment as a categorical factor and baseline measurement for the parameter as a continuous covariate.

CBR is defined as the combination of CR, PR, and SD as defined by modified RECIST Version 1.1 with no progression in bone per PCWG3 criteria.

In all patients with at least one PK sample collected, the trough plasma rucaparib PK data (C<sub>min</sub>) and summary statistics (N, mean, StD, minimum, median, max, CV%) will be reported.

## 11.7.3 Exploratory Efficacy Analyses

The endpoints for exploratory analyses are:

- To assess concordance in BRCA1/BRCA2/ATM gene mutation status in matched Pre-Screening biopsy tissue, archival primary and metastatic tumor tissue and plasma ctDNA
- To assess changes in the molecular profile over time of matched pre and post-treatment tumor or plasma samples
- To evaluate LOH in metastatic disease site biopsy and archival primary and metastatic tumor tissue samples
- To evaluate mechanisms of response and resistance in ctDNA and progression tumor tissue samples
- 11.7.3.1 Concordance of HRR Gene Mutation Status between Metastatic Disease Site Biopsy, Archival Primary and Metastatic Tumor Tissue, and Plasma ctDNA

Pairwise comparisons will be performed for HRR genotyping results between centrally-assessed Pre-Screening biopsy tissue, archival primary and metastatic tumor tissue (where available), and plasma ctDNA in all combinations.
# 11.7.3.2 Changes in Tumor Samples and Changes in Circulating Tumor DNA

Changes in the molecular profile over time of matched pairs of pre and post-treatment tumor tissue (if available) and plasma will be evaluated. Additionally, analysis of plasma ctDNA from serially collected blood will be performed to assess early changes in ctDNA that may associate with response to rucaparib, and to identify and characterize the emergence of mechanisms of resistance.

# 11.7.3.3 Loss of Heterozygosity

Metastatic disease site biopsy and archival primary and metastatic tumor tissue samples, where available, will be analyzed and assigned a percentage loss of heterozygosity (% LOH) score. The concordance between % LOH in archival primary and metastatic tumor tissue and screening biopsy tissue will be evaluated, and the relationship between % LOH (treated as a binary variable) and response to rucaparib will be explored.

## 11.7.3.4 Circulating Tumor DNA in Plasma as a Molecular Marker of Efficacy

Analysis of ctDNA from serially collected blood will be performed to assess early changes in plasma ctDNA that may associate with response to rucaparib, to compare longitudinal ctDNA profiles between rucaparib and comparator arms, and to identify and characterize the emergence of mechanisms of resistance to rucaparib.

# 11.8 Safety Analyses

All safety analyses will be summarized by randomization treatment group. Data form the cross-over period will be summarized separately.

Safety endpoints are incidence of AEs, clinical laboratory abnormalities, and dose modifications.

Data from all patients who receive at least one dose of study drug will be included in the safety analyses. AEs, clinical laboratory results, vital signs, ECG results, ECOG performance status, body weight, and concomitant medications/ procedures will be tabulated and summarized.

#### 11.8.1 Adverse Events

AEs will be classified using the Medical Dictionary for Drug Regulatory Activities (MedDRA) classification system. The severity of the toxicities will be graded according to the NCI CTCAE v4.03 or later. Only TEAEs will be summarized: TEAEs are defined as AEs with onset date on or after the date of first dose of study drug until the date of the last study drug dose plus 28 days.

The number and percentage of patients who experienced TEAEs for each system organ class (SOC) and PT will be presented. Multiple instances of the TEAE in each SOC and multiple occurrences of the same PT are counted only once per patient. The number and percentage of patients with at least one TEAE will also be summarized.

Separate tables will be presented as follows:

- All TEAEs;
- TEAEs by CTCAE grade;
- Grade 3 or greater TEAEs;
- Treatment-related TEAEs;
- Serious TEAEs;
- TEAEs with an outcome of death;
- TEAEs leading to discontinuation of study medication;
- TEAEs resulting in interruption/delay of study medication; and
- TEAEs resulting in dose reduction of study medication.

The incidence of TEAEs will be summarized by relationship to study drug according to the following categories: "treatment-related," or "not treatment-related". If a patient experiences multiple occurrences of the same AE with different relationship categories, the patient will be counted once, as a relationship category of treatment-related.

If a patient experiences multiple occurrences of the same AE with different toxicity grades, the patient will be counted once for the maximum (most severe) toxicity grade. AEs with a missing toxicity grade will be presented in the summary table with a toxicity grade of "Missing." For each toxicity grade, the number and percentage of patients with at least one TEAE of the given grade will be summarized.

### 11.8.2 Clinical Laboratory Evaluations

Clinical laboratory evaluations include the continuous variables for hematology, serum chemistry, and urinalysis. The laboratory values will generally be presented in SI units. The on-treatment period will be defined as the time from the first dose of study drug to 28 days after the last dose of study drug. Laboratory values collected during the on-treatment period will be included in the summary tables. The laboratory values collected after the on-treatment period will only be presented in the data listings.

The summary of laboratory data will include shift tables based on CTCAE for shifts in grade from baseline to maximum, minimum and last value during the on-treatment period.

Supporting laboratory data including normal ranges and abnormal laboratory flags will be provided using by-patient listings. Separate listings will be produced for clinically significant laboratory abnormalities (ie, those that meet Grade 3 or 4 criteria according to CTCAE).

# 11.8.3 Vital Sign Measurements

The on-treatment period will be defined as the time from the first dose of study drug to 28 days after the last dose of study drug. Vital sign measurements collected during the on-treatment period will be included in the summary tables. The vital sign measurements collected after the on-treatment period will only be presented in the data listings.

The summary of vital sign data will include descriptive statistics (N, mean, StD, minimum, median, third quartile, and maximum) of the maximum, minimum and last value during the on-treatment period. Summaries using descriptive statistics (N, mean, StD, minimum, median and maximum) of the change from baseline to the maximum, minimum, and last value during the on-treatment period will also be given.

# 11.9 Interim Analysis

Other than the analysis of OS described below, no formal interim efficacy analyses are planned; however, ongoing review of data by the IDMC will occur.

OS will be analyzed at the time of the primary analysis (interim OS analysis) and again for a final analysis when maturity is reached. It is anticipated that the data for OS will be heavily censored at the time of the primary endpoint analysis. To adjust for multiple analyses of OS at a later stage, a stopping rule will be applied. The Haybittle-Peto<sup>49, 50</sup> stopping rule will be applied where any interim (early) OS with a p-value < 0.001 can be used to claim superiority. This means that a two-sided p-value very close to 0.05 can still be utilized at the final analysis which is projected to be once approximately 70% of the death events has been collected.

### 12 PATIENT DISPOSITION

# 12.1 Removal of Patients from the Study or Study Drug

A patient must be discontinued from protocol-prescribed therapy if <u>any</u> of the following apply:

- Consent withdrawal for any reason at the patient's own request or at the request of their legally authorized representative;
- Radiographic progression of patient's underlying cancer per modified RECIST Version 1.1/PCWG3 (unless, in the opinion of the investigator, the patient continues to derive clinical benefit);
- Unequivocal clinical progression of the patient's underlying cancer that in the opinion of the investigator requires immediate change in systemic anticancer therapy, or results in marked deterioration in ECOG performance status to Grade 3 or higher (adapted from Ryan et al, 2017);<sup>51</sup>
- Any event, adverse or otherwise, that, in the opinion of the investigator, would pose an unacceptable safety risk to the patient;
- An intercurrent illness that, in the opinion of the investigator, would affect assessments of the clinical status to a significant degree and requires discontinuation of therapy; or
- Noncompliance by the patient with protocol-mandated procedures

Discontinuation of treatment does not necessarily indicate study discontinuation for a patient. Samples collected for research will continue to be used unless the patient explicitly withdraws consent for their use. If the patient withdraws consent to continue in the study or discontinues the study for another reason it will be documented in the appropriate eCRF. A patient may withdraw

consent to participate in an additional part of a study that has an additional consent (ie, optional tumor biopsy) yet continue to participate and be treated/ followed in the main part of the study.

The sponsor may discontinue the study early for any of the reasons noted in Section 13.7.

## 13 STUDY ADMINISTRATION

# 13.1 Regulatory and Ethical Considerations

#### 13.1.1 Good Clinical Practice

This study will be conducted in accordance with the protocol and applicable standard operating procedures (SOPs); and in compliance with applicable regulations and guidelines including:

- International Council for Harmonisation (ICH) E6 (R2);
- The Code of Federal Regulations (21 CFR Parts 11, 50, 54, 56, and 312);
- European Union (EU) Directives 2001/20/EC, 2003/94/EC, 2005/28/EC, 536/2014 and
- All applicable local requirements, including the principles of the Declaration of Helsinki.

The investigator will assure that no amendments to the protocol will take place without prior agreement from the sponsor and documented approval from the IRB/IEC, and local health authority (where applicable), except where necessary to eliminate an immediate hazard(s) to the study participants.

Significant noncompliance with the protocol, SOPs, Good Clinical Practice (GCP), and/or applicable regulatory requirement(s) by an investigator/institution, or by member(s) of the sponsor staff or its representatives will lead to prompt action by the sponsor to secure compliance. If monitoring and/or auditing identifies serious noncompliance on the part of an investigator/institution, the sponsor will take steps to secure compliance or terminate the investigator's/institution's participation in the study. When an investigator's/institution's participation is terminated because of significant noncompliance, the sponsor will promptly notify the regulatory authority(ies) and other appropriate parties (eg, IEC/IRB).

All potential serious breaches of GCP must be reported to the sponsor or designee within 24 hours. A serious breach is a breach of the conditions and principles of GCP in connection with the study or the protocol, which is likely to affect, to a significant degree, the safety or physical or mental integrity of the participants of the study or the scientific value of the study.

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study site personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure or debarment).

# 13.1.2 Regulatory Authority Approvals

The sponsor or designee will submit the study protocol plus all relevant study documents to applicable regulatory agencies for approval prior to the study start. No patient will begin the study-specific pre-screening or screening until appropriate regulatory approval of the study protocol has been received.

Each investigator must complete a Form FDA 1572 (or equivalent, when participating in a US Investigational New Drug Application [IND] study). In addition, local statement of investigator documents must be provided where required. Each investigator must submit to the sponsor (or designee) financial disclosure information for studies under a US IND or if required by national law and/or local regulations.

The study will be registered on regionally-relevant registries, including www.clinicaltrials.gov, EudraCT, and other applicable clinical study registry systems as appropriate. Data generated from this study must be handled in accordance with any laws, rules, and regulations related to the privacy of personal data or personal health information applicable in the jurisdiction where the data are processed, including without limitation, the US Health Information Portability and Accountability Act of 1996 (HIPAA), and it implementing regulations, and the EU General Data Protection Regulation 2016/679 (GDPR).

### 13.1.3 Institutional Review Board or Independent Ethics Committee Approval

This protocol, all protocol amendments, and any material to be provided to the patient (such as the ICF, advertisements, patient information sheets (PIS), or descriptions of the study used to obtain informed consent) must be reviewed and approved by the IEC/ IRB before study start, according to national law and/or local regulations. There must be proof of submission of the IB to the IRB/IEC. The sponsor will supply relevant information to the investigator to submit the study protocol and additional study documents to the IEC/ IRB.

Verification of the IEC's/IRB's approval of the study protocol and the written ICF will be transmitted to the sponsor by the investigator or by other means as determined between the investigator and the sponsor.

No patient will begin the study-specific prescreening or screening until appropriate IEC/ IRB approval of the study protocol and ICF/PIS have been received and the investigator has obtained the patient's legally-effective ICF/PIS.

The investigator will submit appropriate reports on the progress of the study to the IEC/ IRB at least annually in accordance with applicable national law and/ or local regulations and in agreement with the policy established by the IEC/ IRB.

The IEC/ IRB must be informed by the investigator of all subsequent protocol amendments and of all SAEs or SUSARs occurring during the study that are likely to affect the safety of the patients or the conduct of the study, according to institutional policies.

#### 13.2 Patient Information and Consent

## 13.2.1 General Aspects of Informed Consent

All information about the clinical study, including the patient information and the ICF, is prepared and used for the protection of the human rights of the patient according to ICH GCP guidelines, the Declaration of Helsinki, and local requirements.

The ICF(s), prepared by the investigator with the assistance of the sponsor, must comply with all applicable regulations, be approved along with the study protocol by the IEC/IRB and be acceptable to the sponsor.

It is the responsibility of the investigator to obtain legally-effective informed consent from each patient participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study, answering all questions from the patients regarding the study, and prior to undertaking any study-related procedures.

#### 13.2.2 Informed Consent Process

The patient must be provided with the patient information, if applicable, and the most current IEC/IRB-approved ICF. The investigator or their designee shall discuss with each patient the nature of the study, its requirements, and that participation is voluntary and may be terminated at any time by the investigator or participant. To participate in the study, informed consent must be obtained from each prospective patient prior to any protocol-specific activities.

The ICF must be in language fully comprehensible to the prospective patient. Patients or legally-authorized representatives (where acceptable according to national law and/or local regulations) must be given sufficient time and opportunity to inquire about the details of the study and to discuss and decide on their participation in the study with the investigator. The patient and the person conducting the informed consent discussion for the study will personally sign and date the ICF in addition to any other required signature (if applicable). A copy of the signed ICF will be retained by the patient or legally-authorized representative and the original ICF will be filed in the investigator file. The process of obtaining informed consent will be documented in the patient's source documents. The date when a patient's informed consent was obtained will be captured in the patient's source documents and eCRF. The patient will need to re-consent if the ICF is updated during the study, such as after an amendment to the protocol, if mandated by the IEC/IRB.

The ICF will contain a separate section that addresses the use of remaining mandatory or optional samples for optional exploratory research. The investigator or authorized designee will explain to each study patient the objectives of the exploratory research. Patients will be told that they are free to refuse to participate and may withdraw their consent at any time and for any reason during the storage period. A separate consent will be required to document a patient's agreement to allow any remaining specimens to be used for exploratory research.

# 13.3 Patient Confidentiality

The investigator must assure that patients' anonymity is strictly maintained and that their identities are protected from unauthorized parties. Only identification codes (ie, no names or, in some regions, initials or date of birth) according to country regulations will be recorded on any form submitted to the sponsor and the IEC/IRB. The investigator must maintain a list with the identity of all study participants, but not intended for use by the sponsor.

The investigator further agrees to take all reasonable precautions to prevent the disclosure of confidential patient information to any unauthorized party or into the public domain. The investigator will notify Clovis Oncology within 24 hours of a security event that impacts or has the potential to impact the confidentiality, integrity, or availability of patient study data.

# 13.4 Study Monitoring

The sponsor, or contract research organization (CRO) or contract monitor acting on the sponsor's behalf, will contact or visit the investigator at the study center prior to the entry of the first patient (unless the sponsor or the CRO has worked with the center recently in the same or comparable indication, the site location and facilities have not changed significantly since after the last visit by the sponsor or CRO, and the potential investigator/site are currently in good standing with respect to regulatory compliance, in which case this initial visit maybe waived) and at appropriate intervals during the study until after the last patient is completed.

In accordance with ICH GCP guidelines, and local regulations, the clinical monitor will periodically review, via direct access, eCRFs, study documents, and medical records (office, clinic, or hospital) for patients enrolled in this study. Monitors will not share patient identifiers with the sponsor. Additionally, the clinical monitor will review and assess research facilities, and clinical laboratory facilities associated with the study. Clinical monitoring will be scheduled to occur at mutually convenient times until completion of the study. If these requirements are in conflict with local regulatory restrictions or institutional requirements, the investigator must inform the sponsor of these restrictions before initiation of the study.

Where applicable, if the sponsor or their representatives are not able to come to the study center, patient study data may be reviewed by them remotely, in conformity with the applicable institutional guidance and local regulations. The site staff may place relevant medical records, with personal identifiers removed, into a secure computer system for the sponsor or their representative to view, allow them to view these records during a video conference, and/or provide them direct access to patient's electronic medical records. This review would occur in a manner that protects the confidentiality of study patient data. Whether a patient's medical records are reviewed at the study center or remotely, their identity and medical records will be kept secure during this process. Remote review of patient study data should not be carried out if adequate data protection, including data security and protection of personal data even if pseudonymized, is not ensured. Further details will be provided in the study training materials and/or the clinical monitoring plan.

The investigator must ensure provision of sufficient time, reasonable space, and adequate qualified personnel for the monitoring visits. The purpose of these visits is to allow the clinical monitor an opportunity to verify adherence to the study protocol and assess the completeness, consistency, and accuracy of data entered in the eCRFs and other documents; however, the investigator retains ultimate responsibility for the quality and integrity of data generated by the site. The clinical monitor will confirm all aspects of the study that are essential for human patient protection and safety as well as those related to the validity and the reliability of study data.

The investigator will make all source data (ie, the various study records, laboratory test reports, other patient records, drug accountability forms, and other pertinent data) and eCRFs for the entire study period available for the monitor. Monitoring is done by comparing study patients' relevant source data that is maintained in site records with the information entered on the eCRFs (ie, source data verification and review).

By agreeing to participate in the study, the investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of the monitoring visits are resolved. Contact information for the study monitor is located in the investigator file. Representatives from the sponsor may also contact and visit the investigators and monitor data during the study.

# 13.5 Case Report Forms and Study Data

The data will be collected using an electronic data capture (EDC) system by remote data entry on eCRFs. Sites will receive training on the EDC system. All users will be supplied with unique login credentials.

Data collection is the responsibility of the clinical study staff at the site under the supervision of the site investigator. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. All source documents will be completed in a neat, legible manner, according to the principles of Attributable, Legible, Contemporaneous, Original or Certified Copy, Accurate, and 'Plus' (+) Complete, Consistent, Enduring, and Available (ALCOA+), to ensure accurate interpretation of data. Data recorded in the eCRF should be consistent with the data recorded on the source documents.

Prior to study start, the investigator will prepare a list showing the signature, handwritten initials, delegated tasks, and dates of delegations for all individuals delegated responsibility on this study. This "study site personnel and delegation list" must be kept current throughout the study.

Clinical data and clinical laboratory data will be entered into a 21 CFR Part 11-compliant EDC system. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. If a patient withdraws from the study, the reason must be noted in the source documents and eCRF. If a patient is withdrawn from the study because of a treatment-limiting AE, thorough efforts will be made to clearly document the outcome.

Laboratory data and investigator observations on the results and any other clinically significant test results are to be documented in the source documents and entered into applicable eCRFs.

Full information regarding EDC and completing eCRFs is included in the investigator files. All questions or comments related to EDC should be directed to the assigned monitor.

Clinical data will be entered directly into the eCRFs from the source documents for all participants who are enrolled.

# 13.6 Independent Data Monitoring Committee

An IDMC will be established to review safety and efficacy data in compliance with a prospective charter. The IDMC will be comprised of medical oncologists with experience in treating patients with the cancer being studied and a statistician, all of whom are not otherwise involved in the study as investigators. The IDMC responsibilities, authorities, and procedures for this study will be documented in the IDMC charter, which will be endorsed and signed by the IDMC members prior to the first data review meeting.

The IDMC will meet at least semi-annually after sufficient data has been collected. The IDMC chairperson may convene a formal IDMC meeting if there are safety concerns. The sponsor can also request an IDMC review of safety data. Details regarding the IDMC will be in the committee charter.

# 13.7 Study Termination and Site Closure

The sponsor, the investigator/institution, or IEC/IRB reserve the right to terminate the study at any time. Should this be necessary, the sponsor and investigator will arrange discontinuation procedures. In terminating the study, the sponsor and the investigator will assure that adequate consideration is given to the protection of the patients' interests. If the trial is terminated prematurely, the sponsor will promptly inform the investigators/institutions, and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension. The investigators will promptly inform their IRB/IEC, providing the reason(s) for the termination or suspension by the sponsor or by the investigator/institution, as specified by the applicable regulatory requirement(s).

The sponsor reserves the right to terminate the study at any time for medical or administrative reasons. When feasible, a 30-day written notification will be given.

The entire study will be stopped if:

- The protocol-specified treatment is considered too toxic to continue the study;
- Evidence has emerged that, in the opinion of the sponsor or the investigator(s), makes the continuation of the study unnecessary or unethical;
- The stated objectives of the study are achieved; or
- The sponsor discontinues the development of rucaparib.

Regardless of the reason for termination, all data available for the patient at the time of discontinuation of follow-up must be recorded in the source documents and on the eCRF. All reasons for discontinuation of treatment must be documented.

# 13.8 Study Protocol Amendments

Protocol amendments must be made only with the prior approval of the sponsor. Agreement from the investigator must be obtained for all protocol modifications and changes to the informed consent document. The IEC/ IRB must be informed of all amendments and give approval prior to their implementation. The sponsor will submit any study protocol amendments to the concerned regulatory authorities (as required) for approval and keep the investigator(s) updated as detailed in the ICH GCP guidelines. Managing protocol deviations is described in Section 13.10.1.

# 13.9 Retention of Study Documents

The study site will maintain a study file, which will contain all documents defined in the ICH E6(R2) Guideline for Good Clinical Practice. The investigator will have control of all essential documents generated by the site. Source documents must be maintained and ALCOA+ documentation practice used. Any changes to source data will be traceable, will not obscure the original entry, and will be explained if necessary (via an audit trail). The investigator must implement procedures to ensure the integrity of any data generated.

The sponsor and investigator will maintain a record of the location(s) of their respective essential documents including source documents. The storage systems used during the study and for archiving (irrespective of media used) must provide for documentation identification, version, history, search, and retrieval. The investigator agrees to keep records and those documents that include (but are not limited to) the identification of all participating patients, medical records, study-specific source documents, source worksheets, all original signed and dated informed consent forms, copies of all eCRFs, query responses, and detailed records of drug disposition to enable inspections or audits from regulatory authorities, the IEC/IRB, and the sponsor or its designees.

The investigator shall retain records and documents, including signed ICFs, pertaining to the conduct of the study for a period of 25 years after study completion or, if no application is to be filed or if the application is not approved for such indication, until at least 5 years after the investigation is discontinued. However, these documents will be retained for a longer period of time if required by the applicable regulatory requirement(s), institutional policies, or if needed by the sponsor. In addition, the investigator must make provision for the patients' medical records to be kept for the same period of time.

No data shall be destroyed without the agreement of the sponsor. Copies of original documents will fulfill the requirements for certified copies. Should the investigator wish to assign the study records to another party or move them to another location, the sponsor must be notified in writing of the new responsible person and/or the new location. The sponsor will inform the investigator, in writing, when the study-related records are no longer needed.

All clinical study information will be recorded, handled, and stored in a way that allows accurate reporting, interpretation, and verification, irrespective of the media used.

Patients' medical records and other original data will be archived in accordance with the archiving regulations or facilities of the investigational site; but at a minimum, for the period defined by the applicable regulatory requirements.

# 13.10 Quality Control and Assurance

The sponsor will implement and maintain quality control and quality assurance procedures with written SOPs to ensure that the study is conducted, and data are generated, documented, and reported in compliance with the protocol, GCP, and applicable regulatory requirements.

#### 13.10.1 Protocol Deviations

The investigator may not deviate from the protocol unless necessary to eliminate immediate hazards to the patient. A deviation may result in the subject having to be withdrawn from the study which could potentially render that patient's data nonevaluable. Any deviation must be documented in the source documents and reported to the sponsor.

## 13.10.2 Study Site Training

Each investigator and the site personnel for this study will be trained by the sponsor and/ or a designee (ie, a CRO) on GCP and on the design, conduct, procedures, and administrative aspects of this study. This training may include, but is not limited to, on-site training, Investigator Meeting(s), and/ or tele/ videoconferencing. Training may be ongoing as refresher, to address specific items, or to introduce changes in the study. When site staff join after study training has been conducted, the investigator is responsible for ensuring that the new staff member is trained.

## 13.10.3 Quality Assurance Audits and Inspections

An audit of a clinical center may be conducted by a quality assurance auditor appointed by the sponsor. The purpose of an audit, which is independent of and separate from routine monitoring or quality control functions, is to evaluate study conduct and compliance with the protocol, SOPs, ICH GCPs, and the applicable regulatory requirements. The investigator will be informed if an audit is to take place and advised as to the scope of the audit. IRB/IEC representatives may also conduct an audit of the study at any time.

Representatives of the FDA, European Medicines Agency (EMA), or other regulatory agencies may conduct an inspection of the study at any time. If informed of such an inspection, the investigator will notify the sponsor immediately.

## 13.10.4 Direct Access to Source Data/ Documents for Audits and Inspections

The investigator will ensure that the auditors or inspectors have access to the clinical supplies, study site facilities, and laboratory, and that all data (including original source documentation) and all study files and audit trails are available, if requested. It is important that the

investigator(s) and their staff cooperate with the quality assurance auditor or regulatory authority inspector during an audit or inspection.

# 13.11 Clinical Study Report

A clinical study report will be prepared under the responsibility and supervision of the sponsor and signed by the sponsor's Chief Medical Officer, Head of Biostatistics, and Head of Regulatory Affairs; thereby indicating their agreement with the analyses, results, and conclusions of the CSR. The CSR will be provided to the clinical investigator(s) and regulatory agency(ies) as required by the applicable regulatory requirements.

# 13.12 Publication and Disclosure Policy

All information for the study provided by the sponsor or designee to the investigator, including, but not limited to, the IB, this protocol, eCRFs, the protocol-specified treatment, and any other study information, will remain the sole and exclusive property of the sponsor during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without the prior written consent of the sponsor. The investigator further agrees to take all reasonable precautions to prevent the disclosure of this information by any employee or agent of the study center to any third party or into the public domain.

All data generated from this study will be maintained by the sponsor. All data generated from this study, and all information furnished by the sponsor, the investigators, and other participating study groups shall be held in strict confidence. Independent analysis and/or publication of study data by the investigator(s) or any member of their staff are not permitted without the prior written consent of the sponsor. Any collaborative publications will be authored in accordance with the applicable guidelines (eg, International Committee of Medical Journal Editors [ICMJE]).<sup>52</sup> Written permission to the investigator will be contingent on the review of the statistical analysis and manuscript/abstract by the sponsor and participating cooperative groups, and will provide for nondisclosure of the confidential or proprietary information.

In all cases, the parties agree to provide all manuscripts or abstracts to all other parties 60 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties.

# 13.13 Investigator Oversight

The investigator has full responsibility for supervising any individual or party to whom they delegate study-related duties and functions conducted at the study site, including satellite locations. The responsibility for supervision includes the services of any party or individual retained by the investigator for this purpose, regardless of location. All staff delegated study responsibilities must be documented on an approved Delegation of Authority log for the study and this filed with the essential documents. In addition, the investigator must ensure that delegated staff are qualified by training, experience and licensure (as applicable). The investigator should implement procedures to ensure integrity of the study and data generated.

# 14 REFERENCE LIST

- 1. Annunziata CM, O'Shaughnessy J. Poly (ADP-ribose) polymerase as a novel therapeutic target in cancer. Clin Cancer Res. 2010;16(18):4517-26.
- Bryant HE, Schultz N, Thomas HD, Parker KM, Flower D, Lopez E, et al. Specific killing of BRCA2-deficient tumours with inhibitors of poly(ADP-ribose) polymerase. Nature. 2005;434(7035):913-7.
- 3. Farmer H, McCabe N, Lord CJ, Tutt AN, Johnson DA, Richardson TB, et al. Targeting the DNA repair defect in BRCA mutant cells as a therapeutic strategy. Nature. 2005;434(7035):917-21.
- 4. Kohler BA, Sherman RL, Howlader N, Jemal A, Ryerson AB, Henry KA, et al. Annual Report to the Nation on the Status of Cancer, 1975-2011, Featuring Incidence of Breast Cancer Subtypes by Race/Ethnicity, Poverty, and State. J Natl Cancer Inst. 2015;107(6):djv048.
- 5. Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011;61(2):69-90.
- 6. Bancroft EK, Page EC, Castro E, Lilja H, Vickers A, Sjoberg D, et al. Targeted prostate cancer screening in BRCA1 and BRCA2 mutation carriers: results from the initial screening round of the IMPACT study. Eur Urol. 2014;66(3):489-99.
- 7. Castro E, Goh C, Olmos D, Saunders E, Leongamornlert D, Tymrakiewicz M, et al. Germline BRCA mutations are associated with higher risk of nodal involvement, distant metastasis, and poor survival outcomes in prostate cancer. J Clin Oncol. 2013;31(14):1748-57.
- 8. Robinson D, Van Allen EM, Wu YM, Schultz N, Lonigro RJ, Mosquera JM, et al. Integrative clinical genomics of advanced prostate cancer. Cell. 2015;161(5):1215-28.
- 9. Mateo J, Carreira S, Sandhu S, Miranda S, Mossop H, Perez-Lopez R, et al. DNA-Repair Defects and Olaparib in Metastatic Prostate Cancer. N Engl J Med. 2015;373(18):1697-708.
- 10. Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, et al. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014;371(5):424-33.
- 11. Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, et al. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010;363(5):411-22.
- 12. Parker C, Gillessen S, Heidenreich A, Horwich A, Committee EG. Cancer of the prostate: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015;26 Suppl 5:v69-77.
- 13. Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, et al. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013;368(2):138-48.

- 14. Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, et al. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004;351(15):1502-12.
- 15. Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, et al. Abiraterone plus Prednisone in Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2017;377(4):352-60.
- 16. Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, et al. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018;378(15):1408-18.
- 17. Hussain M, Fizazi K, Saad F, Rathenborg P, Shore ND, Demirhan E, et al. PROSPER: A phase 3, randomized, double-blind, placebo (PBO)-controlled study of enzalutamide (ENZA) in men with nonmetastatic castrationresistant prostate cancer (M0CRPC). J Clin Oncol. 20 February 2018;36, no. 6\_suppl:3-3.
- 18. Azad AA, Eigl BJ, Murray RN, Kollmannsberger C, Chi KN. Efficacy of enzalutamide following abiraterone acetate in chemotherapy-naive metastatic castration-resistant prostate cancer patients. Eur Urol. 2015;67(1):23-9.
- 19. Suzman DL, Luber B, Schweizer MT, Nadal R, Antonarakis ES. Clinical activity of enzalutamide versus docetaxel in men with castration-resistant prostate cancer progressing after abiraterone. Prostate. 2014;74(13):1278-85.
- 20. Loriot Y, Bianchini D, Ileana E, Sandhu S, Patrikidou A, Pezaro C, et al. Antitumour activity of abiraterone acetate against metastatic castration-resistant prostate cancer progressing after docetaxel and enzalutamide (MDV3100). Ann Oncol. 2013;24(7):1807-12.
- 21. Noonan KL, North S, Bitting RL, Armstrong AJ, Ellard SL, Chi KN. Clinical activity of abiraterone acetate in patients with metastatic castration-resistant prostate cancer progressing after enzalutamide. Ann Oncol. 2013;24(7):1802-7.
- 22. Otto H, Reche PA, Bazan F, Dittmar K, Haag F, Koch-Nolte F. In silico characterization of the family of PARP-like poly(ADP-ribosyl)transferases (pARTs). BMC Genomics. 2005;6:139.
- 23. de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, et al. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010;376(9747):1147-54.
- 24. Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fosså SD, et al. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013;369(3):213-23.
- 25. Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, et al. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016.
- 26. Mukhopadhyay A, Elattar A, Cerbinskaite A, Wilkinson SJ, Drew Y, Kyle S, et al. Development of a functional assay for homologous recombination status in primary cultures of epithelial ovarian tumor and correlation with sensitivity to poly(ADP-ribose) polymerase inhibitors. Clin Cancer Res. 2010;16(8):2344-51.

- 27. Goggins M, Schutte M, Lu J, Moskaluk CA, Weinstein CL, Petersen GM, et al. Germline BRCA2 gene mutations in patients with apparently sporadic pancreatic carcinomas. Cancer Res. 1996;56(23):5360-4.
- 28. Drew Y, Plummer R. The emerging potential of poly(ADP-ribose) polymerase inhibitors in the treatment of breast cancer. Curr Opin Obstet Gynecol. 2010;22(1):67-71.
- 29. Pellegata NS, Sessa F, Renault B, Bonato M, Leone BE, Solcia E, et al. K-ras and p53 gene mutations in pancreatic cancer: ductal and nonductal tumors progress through different genetic lesions. Cancer Res. 1994;54(6):1556-60.
- 30. Pritchard CC, Mateo J, Walsh MF, De Sarkar N, Abida W, Beltran H, et al. Inherited DNA-Repair Gene Mutations in Men with Metastatic Prostate Cancer. N Engl J Med. 2016.
- 31. McCabe N, Turner NC, Lord CJ, Kluzek K, Bialkowska A, Swift S, et al. Deficiency in the repair of DNA damage by homologous recombination and sensitivity to poly(ADP-ribose) polymerase inhibition. Cancer Res. 2006;66(16):8109-15.
- 32. Fong PC, Yap TA, Boss DS, Carden CP, Mergui-Roelvink M, Gourley C, et al. Poly(ADP)-ribose polymerase inhibition: frequent durable responses in BRCA carrier ovarian cancer correlating with platinum-free interval. J Clin Oncol. 2010;28(15):2512-9.
- 33. Audeh MW, Carmichael J, Penson RT, Friedlander M, Powell B, Bell-McGuinn KM, et al. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer: a proof-of-concept trial. Lancet. 2010;376(9737):245-51.
- 34. Tutt A, Robson M, Garber JE, Domchek SM, Audeh MW, Weitzel JN, et al. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and advanced breast cancer: a proof-of-concept trial. Lancet. 2010;376(9737):235-44.
- 35. Gelmon KA, Tischkowitz M, Mackay H, Swenerton K, Robidoux A, Tonkin K, et al. Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triple-negative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol. 2011;12(9):852-61.
- 36. Kaye SB, Lubinski J, Matulonis U, Ang JE, Gourley C, Karlan BY, et al. Phase II, Open-Label, Randomized, Multicenter Study Comparing the Efficacy and Safety of Olaparib, a Poly (ADP-Ribose) Polymerase Inhibitor, and Pegylated Liposomal Doxorubicin in Patients With BRCA1 or BRCA2 Mutations and Recurrent Ovarian Cancer. J Clin Oncol. 2012;30(4):372-9.
- 37. Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, et al. Olaparib Maintenance Therapy in Platinum-Sensitive Relapsed Ovarian Cancer. N Engl J Med. 2012.
- 38. Sandhu SK, Schelman WR, Wilding G, Moreno V, Baird RD, Miranda S, et al. The poly(ADP-ribose) polymerase inhibitor niraparib (MK4827) in BRCA mutation carriers and patients with sporadic cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2013;14(9):882-92.

- 39. De Bono JS, Mina LA, Gonzalez M, Curtin NJ, Wang E, Henshaw JW, et al. First-in-human trial of novel oral PARP inhibitor BMN 673 in patients with solid tumors. J Clin Oncol. 2013;31 (suppl; abstr 2580).
- 40. Kristeleit RS, Shapiro G, LoRusso P, Infante JR, Flynn M, Patel MR. A phase I dose-escalation and PK study of continuous oral rucaparib in patients with advanced solid tumors. J Clin Oncol. 2013;31(suppl):2585.
- 41. Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, et al. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009;361(2):123-34.
- 42. Sandhu SK, Schelman WR, Wilding G, Moreno V, Baird RD, Miranda S, et al. The poly(ADP-ribose) polymerase inhibitor niraparib (MK4827) in BRCA mutation carriers and patients with sporadic cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2013;14(9):882-92.
- 43. Kaufman B, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmaña J, et al. Olaparib monotherapy in patients with advanced cancer and a germline BRCA1/2 mutation. J Clin Oncol. 2015;33(3):244-50.
- 44. Halabi S, Lin CY, Kelly WK, Fizazi KS, Moul JW, Kaplan EB, et al. Updated prognostic model for predicting overall survival in first-line chemotherapy for patients with metastatic castration-resistant prostate cancer. J Clin Oncol. 2014;32(7):671-7.
- 45. Halabi S, Kelly WK, Ma H, Zhou H, Solomon NC, Fizazi K, et al. Meta-Analysis Evaluating the Impact of Site of Metastasis on Overall Survival in Men With Castration-Resistant Prostate Cancer. J Clin Oncol. 2016;34(14):1652-9.
- 46. US Department of Health and Human Services, Food and Drug Administration, CDER, CBER. Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation 2009 [Available from: http://www.fda.gov/downloads/Drugs/.../Guidances/UCM174090.pdf.
- 47. Sandblom G, Carlsson P, Sennfält K, Varenhorst E. A population-based study of pain and quality of life during the year before death in men with prostate cancer. Br J Cancer. 2004;90(6):1163-8.
- 48. National Cancer Institute. Common Terminology Criteria for Adverse Events, Version 4.03 14 June 2010 [Available from: http://www.eortc.be/services/doc/ctc/CTCAE\_4.03\_2010-06-14 QuickReference 5x7.pdf.
- 49. Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol. 1971;44(526):793-7.
- 50. Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, et al. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer. 1976;34(6):585-612.
- 51. Ryan CJ, Kheoh T, Scher HI, De Porre P, Yu MK, Morris MJ. Clinical versus radiographic progression and overall survival for patients (pts) with metastatic castration-resistant prostate cancer (mCRPC) from COU-AA-302. J Clin Oncol. 20 February 2017;35(no. 6\_suppl):193.

- 52. International Committee of Medical Journal Editors. Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals December 2017 [Available from: http://www.icmje.org/recommendations/.
- 53. Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-47.
- 54. US Department of Health and Human Services, Food and Drug Administration, CDER. Guidance for Industry: Clinical Drug Interaction Studies Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions January 2020 [Available from: https://www.fda.gov/media/134581/download.

# 15 APPENDICES

| Appendix I | Modified Response Evaluation Criteria in Solid Tumors Criteria (Version 1.1) and Prostate Cancer Working Group 3 Criteria |
|---|---|
| Appendix 2 | Eastern Cooperative Oncology Group (ECOG) Performance Status Scale |
| Appendix 3 | Cockcroft-Gault Formula |
| Appendix 4 | Examples of CYP Substrates with Narrow Therapeutic Range |
| Appendix 5 | Brief Pain Inventory – Short Form (BPI-SF) |
| Appendix 6 | Functional Assessment of Cancer Therapy – Prostate (FACT P) |
| Appendix 7 | Euro-Quality of Life 5D 5L (EQ-5D-5L) Patient Reported Outcome |
| Appendix 8 | Analgesic Use Questionnaire |

# 15.1 Appendix 1 - Modified Response Evaluation Criteria in Solid Tumors Criteria (Version 1.1) and Prostate Cancer Working Group 3 Criteria

The RECIST guidelines (Version 1.1) are described in Eisenhauer et al. 2009<sup>53</sup> at http://www.eortc.be/Recist/Default.htm and PCWG3 criteria as described by Scher, et al. 2016.<sup>25</sup>

A short summary is given below.

#### Measurable Disease:

<u>Tumor lesions</u>: measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) with the following:

- A minimum size of 10 mm by CT scan (CT scan slice thickness no greater than 5 mm)
- A minimum size of 10 mm caliper measurement by clinical exam (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable)
- A minimum size of 20 mm by chest X-ray

All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be  $\geq 15$  mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be not greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

#### Nonmeasurable Disease:

All other lesions (or sites of disease), including small lesions (longest diameter < 10 mm or pathological lymph nodes with  $\ge 10$  to < 15 mm short axis), as well as truly nonmeasurable lesions, are considered nonmeasurable disease. Lesions considered truly nonmeasurable include leptomeningeal disease, ascites, pleural/pericardial effusions, inflammatory breast disease, lymphangitic involvement of skin and lung, and abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

## **Bone Lesions**

For the purposes of this study, bone metastatic lesions should be recorded at baseline and followed during treatment using PCWG3 criteria. Bone lesions should not be recorded as target or nontarget lesions to be followed by RECIST Version 1.1 criteria; this includes bone lesions with a soft tissue component and soft tissue lesions extending from a bone lesion.

#### **Lesions with Prior Local Treatment**

Tumor lesions situated in a previous irradiated area or in an area subjected to other locoregional therapy are usually not considered measurable unless there has been demonstrated progression in the lesion.

#### **Target Lesions**

All measurable lesions up to a maximum of 5 lesions per organ (per PCWG3), representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. A maximum of 10 target lesions total should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor response.

Prostate and prostatic bed lesions should NOT be selected as target lesions, according to PCWG3 criteria.

### **Nontarget Lesions**

RECIST Version 1.1 criteria require unequivocal quantification of the changes in tumor size for adequate interpretation of the sum of target lesions. Consequently, when the boundaries of the primary are difficult to delineate, this tumor should not be considered a target lesion. A maximum of 10 target lesions total should be selected.

#### **Guidelines for Evaluation of Measurable Disease**

CT and MRI are the best currently available and reproducible methods to measure target lesions selected for response assessment. Conventional CT and MRI should be performed with cuts of 5 mm or less in slice thickness contiguously. Spiral CT should be performed using a  $\leq$  5 mm contiguous reconstruction algorithm. If a site can document that the CT performed as part of a PET/CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast) then the CT portion of the PET/CT can be used for RECIST Version 1.1 measurements.

Lesions on chest X-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.

Ultrasound, endoscopy and laparoscopy should not be used to measure tumor lesions.

Cytology and histology can be used to differentiate between PR and CR in rare cases (eg, after treatment to differentiate between residual benign lesions and residual malignant lesions.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination when both methods have been used to assess the antitumor effect of a treatment.

# **Evaluation of Target Lesions**

| Complete Response | Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm. |
|---|---|
| Partial Response | At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. |
| Stable Disease | Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. |
| Progressive Disease | At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new extra-skeletal lesions is also considered progression. For bone lesions, refer to PCWG3 criteria for determining progressive disease. |

## **Evaluation of Nontarget Lesions**

| Complete Response | Disappearance of all nontarget lesions. |
|---|---|
| Stable Disease/Incomplete Response | Persistence of one or more nontarget lesion(s). |
| Progressive Disease | Appearance of one or more new extra-skeletal lesions and/or unequivocal progression of existing nontarget lesions. For bone lesions, refer to PCWG3 criteria for determining progressive disease. |

# **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

## Evaluation of Best Overall Response: Patients with Target (+/- Non-Target) Disease

| Target Lesions | Nontarget Lesions | New Lesions <sup>a</sup> | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not evaluated | No | PR |
| SD | Non-PD or not evaluated | No | SD |
| Not Evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

New bone metastatic lesions should not be considered as a 'Yes' response; only new extra-skeletal lesions.

#### **Evaluation of Best Overall Response: Patients with Non-Target Disease Only**

| Nontarget Lesions | New Lesions | Overall Response |
|-------------------|-------------|----------------------------|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD <sup>a</sup> |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

<sup>&</sup>lt;sup>a</sup> 'Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as endpoint for assessment of efficacy in some studies so to assign this category when no lesions can be measured is not advised.

Patients with global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be classified as having symptomatic deterioration. Every effort should be made to document the objective progression, even after discontinuation of treatment.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When evaluation of CR depends on this determination, it is recommended that the residual lesion be investigated (fine needle aspiration/biopsy) prior to confirming the complete response status.

#### Confirmation

If an initial CR or PR is noted, confirmatory scans must be performed at least 4 weeks later.

## **Duration of Response (DOR)**

CT scans are required for this study at screening and every 8 calendar weeks (within 7 days before or after is permitted) thereafter. Patients who have been on study at least 24 weeks, may

decrease the frequency of disease/ tumor assessments to every 12 calendar weeks (within 7 days before or after is permitted).

## **Duration of Overall Response**

The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started), including progression in bone per PCWG3 criteria.

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

#### Duration of Stable Disease

SD is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.

#### PCWG3 Criteria for Assessment of Bone Disease

PCWG3 criteria will be used to document evidence of disease progression in bone lesions as described by Scher, et al. 2016.<sup>25</sup>

# Imaging of Baseline Bone Disease

The use of bone scan as the standard for bone imaging is retained in PCWG3, with the presence or absence of metastasis recorded first. A quantitative measure of disease burden, such as lesion number, the bone scan index, or lesion area, is also suggested, recognizing that these measures require further analytical and prospective clinical validation. Changes in lesions considered metastatic on bone scintigraphy should be followed and assessed serially using a bone scan assessment form. Areas/lesions on bone scintigraphy that are suggestive can be assessed further with CT or MRI and followed separately, but such supplemental imaging should not be used to establish indicator lesions for the purposes of a study.

Different modalities for imaging bone metastases can provide different information for the same patient. However, because of the lack of standards for reporting disease presence or changes after treatment, PET imaging with sodium fluoride, fluorodeoxyglucose, choline, or prostate-specific membrane antigen, bone marrow MRI (body MRI), and other modalities that are in use to image bone, should be approached as new biomarkers subject to independent validation.

Criteria for progression in bone at study entry

- Two new lesions observed on 99mTc-MDP or HDP radionuclide bone scintigraphy
- Confirm ambiguous results by other imaging modalities (eg, CT or MRI) however only positivity on the bone scan defines metastatic disease to bone

#### Documentation of baseline bone disease

- Presence or absence of metastasis recorded first
- A quantitative measure of disease burden, such as lesional number, the bone scan index, or lesion area, is required
- Changes in lesions considered metastatic on bone scintigraphy should be followed and assessed serially using a bone scan assessment form. Areas/lesions on bone scintigraphy that are suggestive can be assessed further with CT or MRI and followed separately, but such supplemental imaging should not be used to establish indicator lesions for the purposes of a study

## Following for bone progression during the study

- Exclude pseudoprogression in the absence of symptoms or other signs of progression
- At least two new lesions on scans during the 12-week flare window (ie, the first post-treatment scan), which are persistent and appear with at least two additional lesions on the next scan after the 12-week flare window (2+2 rule)
- If at least two additional new lesions are seen on the next (confirmatory) scan performed after the 12-week flare window, the date of progression is the date of the first post-treatment scan, when the first two new lesions were documented
- For scans after the 12-week flare window (ie, after the first post-treatment scan), at least two new lesions relative to the first post-treatment scan confirmed on a subsequent scan
- Date of progression is the date of the scan that first documents the second lesion
- Changes in intensity of uptake alone do not constitute either progression or regression

## Controlling for Flare by Applying the 2+2 Rule using the First Post-treatment Scan as Baseline



PCWG3 Criteria for Confirmation of Radiographic Progression in Bone by Investigator Assessment (to be used in conjunction with modified RECIST Version 1.1 criteria for visceral and nodal disease)

| Date Progression Detected (Visit) | Criteria for Progression in Bone | Criteria for Confirmation of Progression in<br>Bone |
|---|---|---|
| scan) | bone scan compared to baseline bone scan by PCWG3 | Two or more new bone lesions identified at Week 9 must persist at Week 17 and 2 or more additional new lesions must be identified on Week 17 bone scan (compared to Week 9 scan) |
| scan) | I wo or more new lesions on bone scan compared to Week 9 bone scan. | Two or more new lesions identified at Week 17 must persist at Week 25 bone scan |
| (3 <sup>rd</sup> on-<br>treatment scan | Two or more new lesions bone scan compared to <u>Week 9</u> bone scan | Two or more new lesions identified at Week 25 (or later) bone scan must persist at scan obtained 6 weeks later |

# 15.2 Appendix 2 - Eastern Cooperative Oncology Group (ECOG) Performance Status Scale

| ECC | OG Performance Status |
|---|---|
| 0 | Fully active, able to carry on all predisease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (eg, light house work or office work). |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | Capable of only limited self-care; confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |

In the event performance status is assessed by the Karnofsky Performance Status scale, the following conversion chart applies.

| Karnofsky Performan | ce Status | | ECOG<br>Performance<br>Status |
|---|---|---|---|
| <b>General Description</b> | Score | Specific Description | Score |
| Able to carry on normal activity and to | 100 | Normal; no complaints; no evidence of disease | 0 |
| work; no special care needed | 90 | Able to carry on normal activity; minor signs or symptoms of disease | 1 |
| | 80 | Normal activity with effort; some signs or symptoms of disease | _ |
| Unable to work; able to live at home and | 70 | Cares for self, unable to carry on normal activity or to do active work | 2 |
| care for most personal needs; varying amount | 60 | Requires occasional assistance, but is able to care for most of personal needs | |
| of assistance needed | 50 | Requires considerable assistance and frequent medical care | 3 |
| Unable to care for self; requires equivalent of | 40 | Disabled; requires special care and assistance | _ |
| institutional or hospital care; disease | 30 | Severely disabled; hospital admission is indicated although death not imminent | 4 |
| may be progressing rapidly | 20 | Very sick; hospital admission necessary; active supportive treatment necessary | |
| | 10 | Moribund; fatal processes progressing rapidly | |
| | 0 | Dead | 5 |

# 15.3 Appendix 3 - Cockcroft-Gault Formula

## **Estimated Glomerular Filtration Rate**

Estimated GFR using serum creatinine value is at Screening and each time clinical chemistry testing occurs.

Male 
$$CL_{cr} = \frac{(140 - age) \times Body Weight (kg)}{72 \times Serum Creatinine}$$

Female 
$$CL_{cr} = 140 - age) \times Body Weight (kg) \times 0.85$$
  
72 × Serum Creatinine

This formula expects weight to be measured in kilograms and creatinine to be measured in mg/dL; the calculated units are mL/min.

When serum creatinine is measured in µmol/L:

$$eC_{Cr} = rac{(140 ext{ - Age}) imes ext{Mass (in kilograms)} imes ext{Constant}}{ ext{Serum Creatinine (in $\mu$mol/L)}}$$

Where Constant is 1.23 for men and 1.04 for women.

# 15.4 Appendix 4 - Examples of Sensitive CYP Substrates (not an inclusive list)

| Examples of 0 | CYP Sensitive Substrates Drugs <sup>a</sup> |
|---|---|
| Enzyme or<br>Transporter | Sensitive Substrate Drugs |
| CYP1A2 | Tizanidine, theophylline, alosetron, caffeine, duloxetine, melatonin, ramelteon, tasimelteon |
| CYP2C9 | Celecoxib |
| CYP2C19 | S-mephenytoin, omeprazole |
| CYP3A | Alfentanil, sirolimus, tacrolimus, avanafil, buspirone, conivaptan, darifenacin, darunavir, ebastine, everolimus, ibrutinib, lomitapide, lovastatin, midazolam, naloxegol, nisoldipine, saquinavir, simvastatin, tipranavir, triazolam, vardenafil, budesonide, dasatinib, dronedarone, eletriptan, eplerenone, felodipine, indinavir, lurasidone, maraviroc, quetiapine, sildenafil, ticagrelor, tolvaptan |

Source: FDA Guidance on Clinical Drug Interaction Studies — Cytochrome P450 Enzyme- and Transporter-mediated Drug Interactions, January 2020<sup>54</sup>

Abbreviations: AUC = area under the concentration-time curve; CYP = cytochrome P450; FDA = Food and Drug Administration.

Sensitive substrates are drugs that demonstrate an increase in AUC of ≥ 5-fold with strong index inhibitors of a given metabolic pathway in clinical Drug-drug interaction studies. This table is prepared to provide examples of clinical sensitive or moderate sensitive index substrates and is not intended to be an exhaustive list.

# 15.5 Appendix 5 - Brief Pain Inventory - Short Form (BPI-SF)

A sample form for the BPI-SF is below and background for the questionnaire is available at https://www.mdanderson.org/research/departments-labs-institutes/departments-divisions/symptom-research/symptom-assessment-tools/brief-pain-inventory.html.



| Date: | / | | _/ | | | | | | | | Time: |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Name: | | | Last | | | | F | irst | 7996 | | Middle Initial |
| 7. W | hat tre | eatm | ents o | r med | cations | аге уоц | receiv | ing for | your pa | ain? | |
| | | | | | much r | | | | | | |
| | | | lease<br>ceived | | the one | percen | tage th | at most | shows | now | much relief |
| N | | )% | 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% | Complete<br>Relief |
| 9. C | ircle th | | | | at descr | ibes ho | w, duri | ing the | past 24 | hour | s, pain has |
| | | | th you | | | | | | | | |
| A. | . G | | al Acti | vity<br>3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| D | oes no<br>terfere | t | | _ | | | | | | | Completely<br>Interferes |
| B. | . M | ood | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Ď | oes no<br>terfere | t | 2 | 3 | - | 3 | 0 | | ۰ | | Completely<br>Interferes |
| | | | ng Abil | | | Ļ | | - | | | 40 |
| - T | 1<br>oes no<br>terfere | t | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>Completely<br>Interferes |
| D | | | | | | | | | | | sework) |
| | oes no<br>terfere | t | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>Completely<br>Interferes |
| E | | | | | er people | | | | | | |
| | 1<br>oes no<br>terfere | t | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>Completely<br>Interferes |
| | S | | _ | 200 | 1000 | | 2 | | - | 11110 | 700 |
| _ | oes no<br>terfere | t | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>Completely<br>Interferes |
| G | . Е | njoyr | nent o | f life | | | | | | | |
| | 1<br>oes no<br>terfere | ot | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>Completely<br>Interferes |

# 15.6 Appendix 6 - Functional Assessment of Cancer Therapy – Prostate (FACT-P)

A sample form for the FACT-P is below and background for the questionnaire is available at http://www.facit.org/facitorg/questionnaires.

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | PHYSICAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| GP1 | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| GP2 | I have nausea | 0 | 1 | 2 | 3 | 4 |
| GP3 | Because of my physical condition, I have trouble meeting the needs of my family | 0 | 1 | 2 | 3 | 4 |
| GP4 | I have pain | 0 | 1 | 2 | 3 | 4 |
| GP5 | I am bothered by side effects of treatment | 0 | 1 | 2 | 3 | 4 |
| GP6 | I feel ill | 0 | 1 | 2 | 3 | 4 |
| GP7 | I am forced to spend time in bed | 0 | 1 | 2 | 3 | 4 |
| | SOCIAL/FAMILY WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
| GS1 | I feel close to my friends | 0 | 1 | 2 | 3 | 4 |
| GS2 | I get emotional support from my family | 0 | 1 | 2 | 3 | 4 |
| GS3 | I get support from my friends | 0 | 1 | 2 | 3 | 4 |
| GS4 | My family has accepted my illness | 0 | 1 | 2 | 3 | 4 |
| GS5 | I am satisfied with family communication about my illness | 0 | 1 | 2 | 3 | 4 |
| GS6 | I feel close to my partner (or the person who is my main support) | 0 | 1 | 2 | 3 | 4 |
| Q1 | Regardless of your current level of sexual activity, please answer the following question. If you prefer not to answer it, please mark this box and go to the next section. | | | | | |
| GS7 | I am satisfied with my sex life | 0 | 1 | 2 | 3 | 4 |

Please circle or mark one number per line to indicate your response as it applies to the <u>past 7</u> days.

| | | EMOTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|---|
| | GE1 | I feel sad | 0 | 1 | 2 | 3 | 4 |
| | GE2 | I am satisfied with how I am coping with my illness | 0 | 1 | 2 | 3 | 4 |
| | GE3 | I am losing hope in the fight against my illness | 0 | 1 | 2 | 3 | 4 |
| | GE4 | I feel nervous | 0 | 1 | 2 | 3 | 4 |
| | GE5 | I worry about dying | 0 | 1 | 2 | 3 | 4 |
| | GE6 | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| Γ | | FUNCTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
| | GF1 | FUNCTIONAL WELL-BEING I am able to work (include work at home) | | | | - | • |
| | GF1 | | at all | bit | what | a bit | much |
| | | I am able to work (include work at home) | at all | <b>bit</b> | what | a bit | much 4 |
| | GF2 | I am able to work (include work at home) | 0<br>0<br>0 | <b>bit</b> 1 1 | <b>what</b> 2 2 | 3 3 3 | <b>much</b> 4 4 |
| | GF2<br>GF3 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 | what 2 2 2 | 3 3 3 | 4<br>4<br>4 |
| | GF2<br>GF3<br>GF4 | I am able to work (include work at home) | 0<br>0<br>0<br>0 | bit 1 1 1 1 | what 2 2 2 2 2 | 3 3 3 3 3 | 4 4 4 4 |

# Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | ADDITIONAL CONCERNS | Not at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| C2 | I am losing weight | . 0 | 1 | 2 | 3 | 4 |
| C6 | I have a good appetite | | 1 | 2 | 3 | 4 |
| P1 | I have aches and pains that bother me | . 0 | 1 | 2 | 3 | 4 |
| P2 | I have certain parts of my body where I experience pain | . 0 | 1 | 2 | 3 | 4 |
| Р3 | My pain keeps me from doing things I want to do | . 0 | 1 | 2 | 3 | 4 |
| P4 | I am satisfied with my present comfort level | . 0 | 1 | 2 | 3 | 4 |
| P5 | I am able to feel like a man | . 0 | 1 | 2 | 3 | 4 |
| Р6 | I have trouble moving my bowels | . 0 | 1 | 2 | 3 | 4 |
| P7 | I have difficulty urinating | . 0 | 1 | 2 | 3 | 4 |
| BL2 | I urinate more frequently than usual | . 0 | 1 | 2 | 3 | 4 |
| P8 | My problems with urinating limit my activities | . 0 | 1 | 2 | 3 | 4 |
| BL5 | I am able to have and maintain an erection | . 0 | 1 | 2 | 3 | 4 |

# 15.7 Appendix 7 - Euro-Quality of Life 5D 5L (EQ-5D-5L) Patient-reported Outcome

A sample form for the EQ-5D-5L is included on the next page. Background information for the questionnaire is available at http://www.euroqol.org/home.html.



## **Health Questionnaire**

English version for the USA

USA (English) © 2009 EuroQol Group EQ-5DTM is a trade mark of the EuroQol Group

| Under each heading, please check the ONE box that best describe | bes your nealth TODAY |
|---|---|
| MOBILITY | |
| I have no problems walking | |
| I have slight problems walking | |
| I have moderate problems walking | |
| I have severe problems walking | |
| I am unable to walk | |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | |
| I have extreme pain or discomfort | |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | |

2

USA (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

- We would like to know how good or bad your health is TODAY.
- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =



3

USA (English) © 2009 EuroQol Group EQ-5D $^{\mathrm{IM}}$  is a trade mark of the EuroQol Group

# 15.8 Appendix 8 - Analgesic Use Questionnaire

A sample form for the Analgesic Use Questionnaire is included on the next page.



# **Analgesic Use Questionnaire**

Please indicate the strongest pain medication you have taken within the past 24

| hours: |
|---|
| ☐ 0 = No pain medication |
| ☐ 1 = Non-opioid pain medication such as aspirin [salicylate], acetaminophen [paracetamol], other non-steroidal anti-inflammatory drug [NSAID], etc. |
| ☐ 2 = Mild opioid pain medication such as codeine, hydrocodone, tramadol, etc. |
| ☐ 3 = Strong opioid pain medication such as morphine, oxycodone, |

V1.0 18Oct2016 Page 1 of 1